## CLINICAL STUDY PROTOCOL

#### **KSL0117**

**Study title:** A multicenter, double blind, randomised, parallel groups study

to assess the efficacy and tolerability after single oral administration of Ketoprofen lysine salt 40 mg granules versus Placebo in male and female subjects with acute pain syndrome

after removal of molar teeth

**Study number:** KSL0117

**Phase of development:** III

**Study drug:** OKITASK<sup>®</sup> 40 mg granules for oral administration

**Study disease:** Acute pain syndrome after molar teeth removal

**Sponsor:** Dompé farmaceutici s.p.a.

Contact name and

address:

Mauro P. Ferrari

Via Santa Lucia, 6 20122 Milano, Italy

Tel. +39 02 58383271

Initial version and

date:

Final Version 1.0 - September 26 (As amended on January 25,

2018)

**Prevail Version:** In the event of any inconsistencies between Russian and English

version, the English version shall prevail

## **Confidentiality Statement**

You agree that this document is confidential information of Dompé farmaceutici s.p.a. You should not, directly or indirectly, publish, distribute or otherwise disclose its contents and make available to third parties any part of this document. You should also use this document with the only purpose for which it was provided to you. You may disclose the information only after a written permission of Dompé farmaceutici s.p.a, or to representatives of relevant regulatory authorities, or by the judiciary. The fact of any disclosure of information contained in this document, whether it is authorized or not, should be immediately reported to Dompé farmaceutici s.p.a.


## PROTOCOL APPROVAL PAGE

| SPONSOR: Dompé farmaceutici S.p.A. | |
|---|---|
| Signature: / Muff | Date: 28 - Jan - 2018 |
| Name and position: Marcello Allegretti, ChemD | |
| Chief Scientific Officer | |
| Signature: Mauro P. Ferrari, PharmD | Date: 25-JAH-2018 |
| Early Clinical Development Manager | |
| Signature: Name and position: Luigi Lanata, MD Medical Affairs Director | Date: 25-JAN-2018 |
| CRO: IPHARMA LLC Signature Name and position: Natalia Vostokova, PharmD Chief Operating Officer, IPHARMA LLC | Date |
| Signature Name and position: Julia Trakhtenberg, MD, PhD Medical Director, IPHARMA LLC | Date 30 Jan 2018 |


## INVESTIGATOR PROTOCOL AGREEMENT PAGE

## **FULL NAME:**

I, the undersigned, certify that I have read and understood this protocol. I agree to follow the protocol KSL0117 "A multicenter, double blind, randomised, parallel groups study to assess the efficacy and tolerability after single oral administration of Ketoprofen lysine salt 40 mg granules versus Placebo in male and female subjects with acute pain syndrome after removal of molar teeth".

I undertake to conduct the study in accordance with the requirements of Good Clinical Practice Guidelines of International Conference on Harmonization (ICH Topic E6 (R2) Guideline for Good Clinical Practice (EMA/CHMP/ICH/135/1995 – 1 December 2016)) and Eurasian Economic Union (EAEU), principles outlined in the Declaration of Helsinki, and applicable regulations of Russian Federation.

| Date: | Signature: |
|-------|------------|


## STUDY CONTACTS

| SPONSOR | Dompé farmaceutici s.p.a.<br>Via Santa Lucia, 20122 Milano, Italy |
|---|---|
| Mauro P. Ferrari | Early Clinical Development Manager Tel. +39 02 58383271 E-mail: mauro.ferrari@dompe.com |
| Luigi Lanata | Medical Affairs Director Tel. +39 02 58383473 E-mail: luigi.lanata@dompe.com |
| Laura Boga | Senior Safety Manager – Drug Safety Tel. +39 02 58383568 Fax +39 02 36026913 E-mail: laura.boga@dompe.com SAE reporting: farmacovigilanza@dompe.com |
| SAE/pregnancy reporting | Dompé Drug Safety Fax +39 02 36026913 E-mail: farmacovigilanza@dompe.com |
| CRO (MONITORING,<br>MEDICAL<br>MONITORING) | IPHARMA LLC 7 Nobel str. Skolkovo Innovation Center Moscow, 143026, Russia |
| Natalia Vostokova | Chief Operating Officer Tel. +7 (495) 276-11-43 Fax +7 (495) 276-11-47 E-mail: nv@ipharma.ru |
| Julia Trakhtenberg | Medical Director Tel. +7 (495) 276-11-43 Fax +7 (495) 276-11-47 E-mail: jat@ipharma.ru |
| Victoria Yavorskaya | Medical Advisor<br>Tel. +7 (495) 276-11-43<br>Fax +7 (495) 276-11-47<br>E-mail: yvv@ipharma.ru |
| Valeriy Poddubnyy | Project Manager Tel. +7 (495) 276-11-43 Fax +7 (495) 276-11-47 E-mail: vap@ipharma.ru |
| SAE/pregnancy reporting (available 24 hours a day) | Medical department of IPHARMA Fax +7 (495) 276-11-47 E-mail: SAE@ipharma.ru |


| DATA<br>MANAGEMENT,<br>BIOSTATISTICS | KeyStat LLC,<br>3, 2 <sup>nd</sup> line of Krasnoarmeyskoy svobody str.<br>Smolensk, 214000, Russia |
|---|---|
| Dmitry Khamtsov | Biostatistics and general management Tel. +7 (915) 644-47-13 E-mail: dmitry.khamtsov@keystatsolutions.com |
| CENTRAL<br>LABORATORY | Not applicable |
| LOCAL DEPOT | VORTEX CLINICAL SERVICES 3, Centralnaya str. Golyovo village, Krasnogorskiy district Moscow region, 143405, Russia |
| Vladimir Nesterin | Head of Quality Assurance Tel. + 7 (495) 785-65-78 Tel. + 7 (495) 783-76-53 E-mail: Vladimir.Nesterin@vortexcs.com |
| CLINICAL SITES | According to the approved list of sites available in TMF |


#### **SYNOPSIS**

**Sponsor:** Dompé farmaceutici s.p.a., Italy **Study drug:** OKITASK<sup>®</sup> 40 mg granules

Active substance: Ketoprofen Lysine Salt 40 mg

**Study title:** A multicenter, double blind, randomised, parallel groups study to assess the efficacy and tolerability after single oral administration of Ketoprofen lysine salt 40 mg granules versus Placebo in male and female subjects with acute pain syndrome after removal of molar teeth.

**Study number:** KSL0117 **Phase of development:** III

#### **Primary objective:**

To assess the efficacy of  $OKITASK^{®}$  40 mg granules versus Placebo in patients with acute pain syndrome after removal of one molar tooth by comparing  $AUC_{0-6h}$  of post-treatment pain profile measured by VAS.

## **Secondary objectives:**

To assess the following efficacy and safety parameters of OKITASK® 40 mg granules versus Placebo in patients with acute pain syndrome after removal of one molar tooth:

- Time profile of pain and time profile of pain relief using VAS scales
- Time to first perceptible pain relief (TFPR) and time to meaningful pain relief (TMPR)
- Proportion of patients requiring rescue medication (analgesia) and time to rescue analgesia
- Patient's overall assessment
- Rate of adverse events (AE)

#### **Background:**

Dompé farmaceutici s.p.a. plans to register OKITASK® 40 mg granules which is a new dosage form of Ketoprofen Lysine Salt in Russia.

Ketoprofen is a highly potent NSAID of the propionic acid derivative group. Introduced in 1973, ketoprofen has been, to date, one of the most widely used NSAIDs, accepted as an effective and well tolerated anti-inflammatory treatment. The salification of ketoprofen with the amino-acid lysine remarkably increases the solubility of ketoprofen in water, allowing the development of liquid oral dosage forms of ketoprofen and resulting in three main clinical advantages: 1) a faster absorption from the gastrointestinal (GI) tract compared to the parent compound; 2) a faster-acting anti-inflammatory and analgesic activity; 3) a shorter permanence of the active drug in the stomach and, therefore, a reduced potential for GI irritation and/or ulcerative effects [1].

Ketoprofen lysine salt in the form of granules for oral solution (OKi® 80 mg sachets containing 80 mg of Ketoprofen Lysine Salt in a bipartite sachet, each part containing 40 mg of Ketoprofen Lysine Salt) is already registered and commercialized by Dompé in Italy since 1994 and in Russia since 1998 for the short-term treatment of symptoms of inflammatory conditions with pain.


Dompé farmaceutici s.p.a. September 26, 2017 (As amended on January 25, 2018)

The current study will assess the efficacy and safety of OKITASK® 40 mg granules versus Placebo in patients with acute pain syndrome after extraction of one molar tooth.


## Study design:

This is a multicenter, double-blind, randomized, parallel groups, placebo-controlled study to assess the efficacy and safety of OKITASK® 40 mg granules in patients with acute pain syndrome after removal of molar teeth. The study will be conducted at 4-6 Russian sites. A total expected number of enrolled subjects is 70 (35 per each group). Patients' enrollment to the sites is competitive.

The study will consist of three periods: screening, study treatment and follow-up.

At Screening after signing the informed consent form, patient's demography, medical history and concomitant medications will be collected, oral cavity will be examined, weight and vital signs will be measured and pregnancy test will be performed for inclusion/exclusion criteria assessment. Screening procedures might take up to 4 days before the scheduled tooth extraction procedure including the actual day of extraction.

On Day 1 the patient will undergo extraction of a molar tooth as indicated for the patient's dental condition. The tooth extraction will be conducted using routine technics and anesthetics (recommended types of anesthesia are provided in section 5.9 Concomitant and rescue therapy of the protocol). After that the patient will stay at the site for treatment of pain syndrome according to the protocol.

Pain intensity will be assessed using VAS within 3 hours after the tooth extraction procedure. Patient's overall assessment will be also recorded. If pain intensity on VAS is above 30 mm and pain relief is required, the patient will be randomized in the study.

The patients will be assigned to one of two treatment group in 1:1 ratio:

Group 1. OKITASK® 40 mg – 35 patients

Group 2. Placebo – 35 patients

The patient will assess pain by VAS at 0' – immediately before study drug dosing.

Upon study drug administration the patients will immediately start two stopwatches. One of them will be stopped once the patient feels first perceptible pain relief; the second one will be stopped once the patient feels the meaningful pain relief.

The patient will stay at the site for 6 hours post-dose for pain and AE assessment. Pain intensity will be assessed by VAS at 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) post-dose. Pain relief will be assessed by VAS at 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) post-dose.

Patients should mark actual time points of VAS measurement. Deviations from planned time points will not be considered as protocol deviations. Only omitted values will be considered as protocol deviations.

Patients' overall assessment will be performed right before the discharge from the site.

Follow-up phone call to the patient to assess AEs will be performed on Day 3 (48 hours after the study drug dosing). Any SAE spontaneously reported by the patient within 30 days of dosing will be collected.

Should the patient require rescue medication at any time during 6 hours post-dose, the last VAS measurement and patient's overall assessment will be performed before the rescue medication dosing (see 7.3).


## **Patients population:**

Male and female adult patients scheduled for extraction of a molar tooth.

#### Inclusion and exclusion criteria:

#### **Inclusion criteria:**

- 1. Signed Informed Consent Form;
- 2. Male and female, from 18 years to 65 years (inclusively);
- 3. Subjects who undergo removal of a **non-impacted** molar tooth within 3 hours before randomization in the study;
- 4. Subjects in generally good health (based upon criteria for safe administration of outpatient conscious sedation);
- 5. Subjects requesting relief for postoperative pain within 3 h after the tooth extraction (VAS ≥30 mm);
- 6. Subjects willing to undergo observation period for up to 9 hours after the tooth extraction:
- 7. Ability to complete a 100 mm VAS and a category scale during the observation period (about 9 hours);
- 8. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study;
- 9. Contraception (for females): females of child-bearing potential must be using at least one reliable method of contraception, as follows:
  - a. hormonal oral, implantable, transdermal, or injectable contraceptives;
  - b. a non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide;

#### or should have:

- c. a male sexual partner who agrees to use a male condom with spermicide;
- d. a sterile sexual partner.

#### **Exclusion criteria:**

- 1. Subjects undergoing extraction of impacted and dystopic teeth, tooth preserving operations, apically positioning flap/vestibuloplasty with free gingival graft from the palate;
- 2. Subjects undergoing more than one tooth extraction in the same extraction procedure;
- 3. Subjects undergoing dental implantation simultaneously with tooth extraction;
- 4. Allergy: ascertained or presumptive hypersensitivity to the active substances (ketoprofen and paracetamol as rescue medication) and/or formulations' ingredients; history of hypersensitivity to drugs (in particular to NSAIDs) or allergic reactions in general, which the Investigator considers may affect the outcome of the study;
- 5. Diseases: relevant history of renal, hepatic, cardiovascular, respiratory (including asthma), skin, haematological, endocrine, gastro-enteric and genitourinary tract or


neurological and autoimmune diseases, that may interfere with the aim of the study;

- 6. Medications: non-steroidal anti-inflammatory drugs (NSAIDS) and other analgesics [in particular ketoprofen, paracetamol and acetylsalicylic acid (ASA)], antihistamines, sedating medications, including herbal and BASs, taken 48 h before surgery;
- 7. Investigational drug trials: participation in the evaluation of any drug within 3 months before screening (including the last study procedure);
- 8. Relevant history of drug and alcohol abuse.
- 9. Positive Pregnancy test in female patients of childbearing potential (including patients in post-menopausal status for less than 2 years).

## Investigational Product dosage and route of administration:

Active substance: Ketoprofen Lysine Salt (KLS)

Pharmacological class: Anti-inflammatory and Antirheumatic Products, Non-Steroids (ATC code: M01AE03).

Dosage form: 40 mg KLS granules (corresponding to 25 mg ketoprofen)

Dosing: 1 sachet – single dose

Storage conditions: Keep at temperature not higher than +25°C

Manufacturer: Dompé farmaceutici s.p.a. (Italy)

Re-packaging (primary and secondary): Monteresearch (Italy)

Batch control and release: Dompé farmaceutici s.p.a. (Italy)

**Control: Placebo** 

Dosage form: 0 mg KLS granules

Dosing: 1 sachet - – single dose

Storage conditions: Keep at temperature not higher than +25°C

Manufacturer: Monteresearch (Italy)

Batch control and release: Dompé farmaceutici s.p.a. (Italy)

## **Efficacy endpoints:**

## Primary efficacy endpoint:

-  $AUC_{0-6h}$  of pain profile between time 0 (baseline value of VAS) and 6 hours post-treatment

Pain will be assessed by a horizontal 100 mm Visual Analogue Scale (VAS): 0 no pain – 100 worst pain imaginable at: 0' (just before taking the first medication VAS should be >30 mm) and 5', 10', 15', 30', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) after the drug administration.

Patients should mark actual time points of VAS measurement. Deviations from planned time points will not be considered as protocol deviations. Only omitted values will be considered as protocol deviations.

The  $AUC_{0-6h}$  will be calculated using the trapezoidal rule. Should the patient require rescue medication at any time during 6 hours post-dose, the last VAS measurement


assessment will be performed. The last observation will be used for calculation of  $AUC_{0-6h}$  (LOCF).

## Secondary efficacy endpoints:

## - Time profile of pain and time profile of pain relief

Pain will be assessed by a horizontal 100 mm Visual Analogue Scale (VAS): 0 no pain – 100 worst pain imaginable at: 0' (just before taking the first medication VAS should be >30 mm) and 5', 10', 15', 30', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) after the drug administration.

Patients should mark actual time points of VAS measurement. Deviations from planned time points will not be considered as protocol deviations. Only omitted values will be considered as protocol deviations.

Pain relief will be assessed by a horizontal 100 mm VAS: 0 no relief – 100 maximum relief at: 5', 10', 15', 30', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) after the drug administration.

Should the patient require rescue medication at any time during 6 hours post-dose, the last VAS assessment will be performed. Further efficacy measurements (if any) will be discontinued from the analysis.

## - Time to first perceptible relief (TFPR) and time to meaningful pain relief (TMPR)

Time to first perceptible relief (TFPR) and time to meaningful pain relief (TMPR) will be measured by stopwatches. Upon study drug administration the patients will immediately start two stopwatches. One of them will be stopped once the patient feels first perceptible pain relief; the second one will be stopped once the patient feels the meaningful pain relief

# - Proportion of patients requiring rescue medication (analgesia) and time to rescue analgesia

In the event of poor pain control, the patient will receive a rescue medication for analgesia (i.e. paracetamol 500-1000 mg tablets). Time to rescue medication with an alternative analgesic, if it occurred, will be also recorded (NB: subjects will be encouraged to postpone the rescue medication until after 1 hour post-dose). If Paracetamol 500 mg-1000 mg is not effective, the patient will be allowed to take another dose of Paracetamol 500 mg-1000 mg. Interval between dose taking is not less than 4 hours; the maximum daily dose is 4000 mg.

## - Patient's overall assessment

Patient's overall assessment (5-point scale): 1 = very good, 2 = good, 3 = satisfactory, 4 = poor, 5 = very poor.

Assessment will be performed after VAS at Baseline and just before discharge from the site. If a patient takes rescue medication, the Patient's overall assessment will be performed after the last VAS assessment.

## Safety endpoints:

## - Adverse events (AE) rates

AEs will be collected according to the subject's complaints, oral cavity examination, and vital signs.


## **Statistical methods:**

All subjects data collected on the eCRF will be listed by subject, treatment group and center. Appropriate descriptive statistics will be produced, according to the variable. For continuous data, the mean, standard deviation (SD), median, range (minimum and maximum) and 95% confidence interval (CI) will be presented. For categorical data, frequencies and percentages will be presented. If appropriate, 95% CI for proportions will be presented. Unless otherwise specified, the significance level used for statistical testing will be 0.05 and two-sided tests will be used. A Statistical Analysis Plan will be issued describing details of all the statistical methods and analysis to be applied to trial results.

## Analysis of the primary efficacy endpoint:

Primary variable will be the  $AUC_{0-6h}$  of pain profile between time 0 (baseline value of VAS) and 6 hours post-treatment.

 $AUC_{0-6h}$  analysis will be based on actual rather than scheduled timings and will be calculated using the trapezoidal rule. If the actual time is not recorded, the scheduled time will be used instead.

Treatment AUCs will be compared by means of Student's t-test for independent data. Null hypothesis  $(H_0)$  that  $OKITASK^{@}$  is not different from Placebo will be rejected and alternative hypothesis  $(H_1)$  that  $OKITASK^{@}$  is superior to Placebo will be accepted if mean  $AUC_{0-6h}(OKITASK^{@})$  is less than mean  $AUC_{0-6h}(Placebo)$  and p < 0.05.

## Analysis of the safety endpoints:

All AEs recorded on eCRF during the study will be coded by System Organ Class (SOC) and Preferred Term (PT) using the Medical Dictionary for Drug Regulatory Affairs (MedDRA [5]). They will be tabulated and summarized by treatment, relation to study treatment and severity.


## Sample size:

Sample size calculation was based on the paper of Seymour 1996 [3] concerning a randomized, double-blind, placebo-controlled study of treatment with placebo, paracetamol (500 and 1000 mg) and ketoprofen (12.5 and 25 mg).

The unadjusted  $AUC_{0-6h}$  values for placebo and ketoprofen were about 263 and 173 mm h-1, respectively. The corresponding SD were 106 mm h-1 (about 40% of the mean value for placebo AUC) and 121 mm h-1 (about 70% of the mean value for ketoprofen 25 mg AUC).

The testing hypothesis for this trial is the superiority of ketroprofen versus placebo that in statistical term is:

H0: mean of placebo  $\geq$  mean of ketoprofen (no difference between treatments)

H1: mean of placebo < mean of ketoprofen (clinically and statistically significant difference between the groups)

A total of 58 subjects (29 subjects per group) will be necessary to assess a difference of 90 mm h-1 between the groups with a power of 80%,  $\alpha = 0.05$ , SD = 121 mm h-1, and randomization rate of 1:1. Sample size calculation was performed using SAS 9.2 [4].

Assuming a drop-out rate of 15%, 70 subjects in total (35 subjects per group) should be enrolled. Considering the screen-failure rate of about 30%, up to 100 patients will be screened in the study. Patients' enrollment to the sites is competitive.

#### Randomization:

Subjects will be randomly assigned one of the two equal groups at 1:1 ratio. Randomization will be conducted with the use of interactive web response system (IWRS).

#### **Protocol version and date:**

KSL0117 Final version 1.0 dated September 26, 2017 (As amended on January 25, 2018).


| TABLE OF CONTENT | |
|------------------------------------------------|----|
| STUDY CONTACTS | 4 |
| SYNOPSIS | 6 |
| LIST OF ABBREVIATIONS | 17 |
| 1. INTRODUCTION | 19 |
| 2. STUDY OBJECTIVES | 21 |
| 2.1. Primary objective | 21 |
| 2.2. Secondary objectives | 21 |
| 3. STUDY DESIGN | 22 |
| 3.1. General design and study plan | 22 |
| 3.1.1. Study design | 22 |
| 3.2. Rationale of the study design | 25 |
| 3.3. Study duration | 25 |
| 3.4. Previous experience with OKITASK® | 26 |
| 3.4.1. Preclinical Data | 27 |
| 3.4.2. Clinical Data | 28 |
| 3.5. Dose Rationale and Risk/Benefits | 35 |
| 4. STUDY POPULATION | 37 |
| 4.1. Study population | 37 |
| 4.2. Inclusion Criteria | 37 |
| 4.3. Exclusion Criteria | 37 |
| 4.4. Re-screening procedures | 38 |
| 5. STUDY DRUG | 39 |
| 5.1. Description | 39 |
| 5.2. Treatment Regimen | 40 |
| 5.3. Randomization and blinding | 40 |
| 5.4. Unblinding procedure | 40 |
| 5.5. Study treatment compliance | 40 |
| 5.6. Packaging and labelling | 40 |
| 5.7. Study drug accountability | 41 |
| 5.8. Study drug storage | 41 |
| 5.9. Concomitant and rescue therapy | 41 |
| 5.10. Prohibited prior and concomitant therapy | 42 |
| 6. STUDY PROCEDURES | 43 |
| 6.1. Informed Consent | 43 |
| 6.2. Patients registration | 43 |
| 6.3. Demographic data and medical history | 43 |
| 6.4. Oral cavity examination | 43 |
| 6.5. Vital signs, weight and height | 43 |


58

10.5. Record keeping

| | rug OKITASK <sup>®</sup><br>rotocol KSL0117 Final version 1.0 | Dompé farmaceutici s. <sub>1</sub><br>September 26, 2017 (As amended on January 25, 20 | |
|---|---|---|---|
| 10.6. | Ethical aspects | | 58 |
| 10.6 | 5.1. Independent Ethics Committee | | 58 |
| 10.6 | 5.2. Ethical considerations | | 58 |
| 10.6 | 5.3. Informed Consent | | 58 |
| 10.7. | Financing | | 59 |
| 10.8. | Publication Policy | | 59 |
| 11. | REFERENCES | | 60 |
| 12. | APPENDIX | | 63 |
| 12.1. | Visual analogue scale "Pain intensity" | | 63 |
| 12.2. | Visual analogue scale "Pain relief" | | 63 |
| 12.3. | Patient's overall assessment (5-point so | eale) | 63 |
| LIST | OF TABLES | | |
| Table | 1 Schedule of visits and procedures | | 24 |
| Table | 2. Study KSL0112 Summary Pharmacok | kinetic Data and 90% Confidence Intervals | 30 |
| LIST | OF FIGURES | | |
| _ | | on (μg/mL) vs. time profiles after administration | |
| _ | | anules (T) (• solid line) and 40 mg of ketoprofen | |
| • | | ted line) in semilogarithmic scale | |
| _ | <u> </u> | chet. | |
| Figure | 3 Labeling of the sachet | | 41 |


## LIST OF ABBREVIATIONS

| AA | Arachidonic acid |
|----------|-----------------------------------------------------|
| ADME | Absorption, Distribution, Metabolism, Excretion |
| ADR | Adverse drug reaction |
| AE | Adverse events |
| ALT | Alanine transaminase |
| AUC | Area under the concentration-time curve |
| ASA | Acetylsalicylic acid |
| BAS | Biologically Active Suppliments |
| BMI | Body mass index |
| BP | Blood pressure |
| CI | Confidence Interval |
| CFS | Cell-free supernatant |
| CNS | Central nervous system |
| COX | Cyclo-oxygenase |
| СРК | Creatine phosphokinase |
| CRF | Case report form |
| CVS | Cardiovascular system |
| DNA | Desoxyribonucleic acid |
| ECG | Electrocardiogram/electrocardiography |
| eCRF | Electronic Case Report Form |
| ED | Early discontinuation (early discontinuation visit) |
| ET | End of treatment |
| ETV | Early Termination Visit |
| EU | European Union |
| FS | Food Supplement |
| FVC | Forced vital capacity |
| GI tract | Gastro-intestinal tract |
| GLP | Good Laboratory Practice |
| Н | Hour |
| HR | Heart rate |
| IASP | International Association for the Study of Pain |
| ICD | International Classification of Diseases |
| ICSRs | Individual case safety reports |


| I.V. | Intravenous |
|--------|----------------------------------------------|
| IEC | Independent Ethics Committee (local) |
| IMP | Investigational medicinal product |
| KA | Ketoprofen acid |
| KLS | Ketoprofen lysine salt |
| KP | Ketoprofen |
| MeDRA | Medical Dictionary for Regulatory Activities |
| МоН | Ministry of Health |
| NSAIDs | Non-steroid anti-inflammatory drugs |
| NZW | New Zealand White |
| OA | Osteoarthritis |
| OTC | Over-the-Counter |
| PID | Pain intensity different |
| PD | Pharmacodynamic(s) |
| PK | Pharmacokinetic(s) |
| PG | Prostaglandins |
| POM | Prescribtion only medications |
| RA | Rheumatoid arthritis |
| REMD | Rescue medication |
| SADR | Serious adverse drug reaction |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SDV | Source Data Verification |
| SmPC | Summary of Product Characteristics |
| SOC | System Organ Class |
| SOP | Standard Operation Procedures |
| TEAEs | Treatment-Emergent Adverse Events |
| TFPR | Time to first perceptible relief |
| TMPR | Time to meaningful pain relief |
| TC | Telephone contact |
| TK | Toxicokinetic |
| VAS | Visual Analogue Scale |


#### 1. INTRODUCTION

Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) are a chemically heterogeneous group of compounds, often chemically unrelated, which share some therapeutic effects and adverse reactions. The principal therapeutic effects of NSAIDs derive from their ability to inhibit prostaglandin production through the inhibition of an important enzyme in the prostaglandin synthetic pathway, cyclo-oxygenase or COX. All NSAIDs have antipyretic, antalgic and anti-inflammatory properties, and are commonly used for the treatment of inflammatory diseases, especially musculoskeletal disorders, characterized by pain and inflammation. The most common adverse reactions of NSAIDs are gastrointestinal and cardiovascular effects [1].

Ketoprofen lysine salt (KLS), introduced in Italy in 1980 has proved to exert antiinflammatory, analgesic and antipyretic activities comparable to those of ketoprofen with the advantage, due to its better solubility, of allowing a wide range of formulations, high dosage flexibility and a reliable tolerance profile [3].

The salification of ketoprofen with the amino-acid lysine remarkably increases the solubility of ketoprofen in water, allowing the development of liquid oral dosage forms of ketoprofen and resulting in three main clinical advantages: 1) a faster absorption from the gastrointestinal (GI) tract compared to the parent compound; 2) a faster-acting anti-inflammatory and analgesic activity; 3) a shorter permanence of the active drug in the stomach and, therefore, a reduced potential for GI irritation and/or ulcerative effects.

In comparative studies, ketoprofen appears to be at least as effective as other anti-inflammatory and antalgic agents [3]. The side effects of ketoprofen are similar to those of all NSAIDs, gastrointestinal disturbances being the most frequent: nausea, vomiting, diarrhea, flatulence, constipation, dyspepsia, abdominal pain, more rarely peptic ulcerations, perforation, gastritis or gastrointestinal bleeding [3]. Approximately 30% of subjects experience mild gastrointestinal side effects with ketoprofen, which are decreased if the drug is taken with food or antacids [3. Other less frequent undesirable effects of ketoprofen are cutaneous events (urticaria, erythema, cutaneous rash), general events (allergic and anaphylactoid reactions), nervous events (dizziness and vertigo), cardiovascular events (palpitations, tachycardia, hypotension and hypertension), respiratory events (bronchospasm, dyspnea), renal events (retention of water) and disorders of haematic crisis and of the urinary tract. In most of the cases, symptoms are transient and resolve with the suspension of the therapy and with a specific pharmacological treatment.

Ketoprofen Lysine salt in the form of granules for oral solution (OKi<sup>®</sup> 80 mg sachets containing 80 mg of KLS in a bipartite sachet, each part containing 40 mg of KLS) has been registered and commercialized by Dompé in Italy since 1994 and in Russia since 1998 for the short-term treatment of symptoms of inflammatory conditions with pain.

KLS 40 mg granules in sachets was registered in Italy since 2001 for the treatment of pain of various nature and origin (headache, toothache, neuralgia, menstrual pain, muscular and osteoarticular pain) but was not commercialized.

Ketoprofen at the lower dose of 25 mg (corresponding to 40 mg of KLS granules) has been studied in humans as an analgesic. Different presentations of ketoprofen 25 mg oral formulations are marketed in the EU by different MAH and under different trademarks (e.g.: Toprec® by Sanofi-Aventis, France; Toprek® by Sanofi-Aventis, Italy, Fastum® by Menarini, Italy).

The new formulation of ketoprofen Lysine salt 40 mg granules for oral administration (corresponding to 25 mg as ketoprofen) is similar in terms of content of active ingredient to the marketed ketoprofen 25 mg formulations for oral administration. OKITASK® 40 mg granules (ketoprofen Lysine salt 40 mg, corresponding to 25 mg of ketoprofen) has been commercialized in


Italy since 2012 for the following therapeutic indications: pain of various kinds and origins, in particular headache, toothache, neuralgia and menstrual, muscular and osteoarticular pain. OKITASK® 40 mg granules has been also commercialized in Albania since May 2015 and Kosovo since July 2016; a new formulation of OKITASK® 40 mg in tablets was authorized in Italy in February 2017.

The safety of KLS has been reported to be comparable to that of ketoprofen in preclinical toxicological studies; moreover, because of the faster GI absorption the permanence of the drug in the GI tract is thought to be reduced and, therefore, a lower potential for GI irritation is expected in humans.

The safety evaluation of OKi® granules for oral solution and OKi® drops in humans has been carried out within clinical studies performed with the KLS oral formulations (both pharmacokinetic and clinical efficacy studies) by careful monitoring of all adverse events (AEs) and adverse drug reactions (ADRs) occurring in the studies. In addition, a specific safety trial has been performed to investigate the potential of KLS to induce GI irritation and/or ulceration.

The extremely low frequency of the AEs after treatment with KLS and their occurrence also in subjects treated with placebo suggest a very good safety profile for both  $OKi^{®}$  granules and  $OKi^{®}$  drops [3].

The post-marketing experience with oral formulations of OKi<sup>®</sup> shows that AEs are quite rare. Nonetheless, the adverse effects could be minimized by using the lowest effective dose of the new KLS 40 mg orodispersible granules for oral administration. In fact the corresponding dose of ketoprofen acid is 25 mg instead of 50 mg contained in one sachet of OKi<sup>®</sup> 80 mg granulates for oral solution.

This proposed study has been designed to demonstrate the efficacy of OKITASK® 40 mg granules for oral administration in a model of mild and moderate pain with the proposal its further registration in Russia.


## 2. STUDY OBJECTIVES

## 2.1. Primary objective

The primary objective of this study is to assess the efficacy of  $OKITASK^{\otimes}$  40 mg granules versus Placebo in patients with acute pain syndrome after removal of one molar tooth by comparing  $AUC_{0-6h}$  of post-treatment pain profile measured by VAS.

## 2.2. Secondary objectives

Secondary objectives of this study are to assess the following efficacy and safety parameters of OKITASK® 40 mg granules versus Placebo in patients with acute pain syndrome after removal of one molar tooth:

- Time profile of pain and time profile of pain relief using VAS scales
- Time to first perceptible pain relief (TFPR) and time to meaningful pain relief (TMPR)
- Proportion of patients requiring rescue medication and time to rescue medication
- Patient's overall assessment
- Rate of adverse events (AE)


#### 3. STUDY DESIGN

## 3.1. General design and study plan

This is a multicenter, double blind, randomised, parallel groups study to assess the efficacy and tolerability after single oral administration of Ketoprofen lysine salt 40 mg granules versus Placebo in male and female subjects with acute pain syndrome after removal of a molar tooth.

The study will be conducted at 4-6 Russian sites. A total expected number of enrolled subjects is 70 (35 per each group). Patients' enrollment to the sites is competitive.

## 3.1.1. Study design

The study will consist of three periods: screening, study treatment and follow-up.

## 3.1.1.1. Screening

At Screening after signing the informed consent form, patient's demography, medical history and concomitant medications will be collected, oral cavity will be examined, weight and vital signs will be measured and pregnancy test will be performed for inclusion/exclusion criteria assessment. Screening procedures might take up to 4 days before the scheduled tooth extraction procedure including the actual day of extraction.

On Day 1 the patient will undergo extraction of a molar tooth as indicated for the patient's dental condition. The tooth extraction will be conducted using routine technics and anesthetics (recommended types of anesthesia are provided in section 5.9 Concomitant and rescue therapy of the protocol). After that the patient will stay at the site for treatment of pain syndrome according to the protocol.

Pain intensity will be assessed using VAS within 3 hours after the tooth extraction procedure. Patient's overall assessment will be also recorded. If pain intensity on VAS is above 30 mm and pain relief is required, the patient will be randomized in the study.

#### 3.1.1.2. Study treatment

The patients will be assigned to one of two-treatment group in 1:1 ratio:

Group 1. OKITASK® 40 mg – 35 patients

Group 2. Placebo – 35 patients

The patient will assess pain by VAS at 0' – immediately before study drug dosing.

Upon study drug administration the patients will immediately start two stopwatches. One of them will be stopped once the patient feels first perceptible pain relief; the second one will be stopped once the patient feels the meaningful pain relief.

The patient will stay at the site for 6 hours post-dose for pain and AE assessment. Pain intensity will be assessed by VAS at 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) post-dose.

Pain relief will be assessed by VAS at 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) post-dose.

Patients should mark actual time points of VAS measurement. Deviations from planned time points will not be considered as protocol deviations. Only omitted values will be considered as protocol deviations.

Patients' overall assessment will be performed right before the discharge from the site.


Dompé farmaceutici s.p.a. September 26, 2017 (As amended on January 25, 2018)

Should the patient require rescue medication at any time during 6 hours post-dose, the last VAS measurement and patient's overall assessment will be performed before the rescue medication dosing.

## 3.1.1.3. Follow-up

Follow-up phone call to the patient to assess AEs will be performed on Day  $3\pm1$  (48 hours after the study drug dosing). Any SAE spontaneously reported by the patient within 30 days of dosing will be collected.

The study procedures schedule is summarized in Table 1.


## Table 1 Schedule of visits and procedures

| | | Study treatments | | | | | | | | Study treatments | | | | | | ED <sup>3</sup> | Follow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Test/Examination | Screening | Baseline <sup>1</sup><br>(Pre-dose) | | | | | | | | | Phone call | | | | | | |
| Day | Day-4Day 1 | Day 1 | | | | | | | Da | y 1 | | | | | | Day 1 | Day 3±1 |
| Hours | | 0 | | 0.08 | 0.17 | 0.25 | 0.5 | 0.75 | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | > 1 | 48 |
| Minutes | | 0 | | 5 | 10 | 15 | 30 | 45 | 60 | 90 | 120 | 180 | 240 | 300 | 360 | > 60 | |
| Informed consent & screening n° assignment | X | | | | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | | | |
| Medical history and underlying disease | X | | S | | | | | | | | | | | | | | |
| Oral cavity examination | X | | Study | | | | | | | | | | | | | | |
| Height <sup>6</sup> | X | | | | | | | | | | | | | | | | |
| Weight | X | | drug/placebo | | | | | | | | | | | | | | |
| Vital signs | X | | g/F | | | | | | | | | | | | | | |
| Pregnancy test | X | | lac | | | | | | | | | | | | | | |
| Extraction of a molar tooth | X (Day 1) | | ceb | | | | | | | | | | | | | | |
| Pain Intensity Assessment VAS (0-100 mm) <sup>7</sup> | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Inclusion/exclusion criteria <sup>2</sup> | X | | dm | | | | | | | | | | | | | | |
| Randomization number assignment | | X | administration | | | | | | | | | | | | | | |
| Patient's overall assessment (5-point scale) <sup>7</sup> | | X | tra | | | | | | | | | | | | X | X | |
| Pain Relief Assessment VAS (0-100 mm) | | | l tio | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Time to first perceptible relief (TFPR) | | | ם | | | | | | , | X | | | | | | | |
| measured by stopwatch <sup>4</sup> | | | | | | | | | | | | | | | | | |
| Time to meaningful pain relief (TMPR) | | | | | | | | | , | X | | | | | | | |
| measured by stopwatch <sup>4</sup> | | | | | | | | | | | | | | | | | |
| Rescue medication (if applicable) <sup>6</sup> | | | | | | | | | | | | | | | | X <sup>5</sup> | |
| Concomitant medications | X | X | ] | | | | | | 2 | K | | | | | | X | X |
| Previous therapy(ies) | X | X | 1 | | | | | | | | | | | | | | |
| Adverse events | X | X | X X | | | | | X | X | | | | | | | | |

- 1. After surgery, before the study drug administration
- 2. Confirmation of the Inclusion/Exclusion criteria prior to randomization
- 3. Should the patient require rescue medication at any time during 6 hours post-dose, the last VAS measurement and patient's overall assessment will be performed before the rescue medication dosing. Subjects will be encouraged to postpone the rescue medication until after 1 hour post-dose. The ED assessments will be performed before rescue treatment; actual time of VAS will be captured.
- 4. The time of stopwatch will be recorded on eCRF
- 5. In the event of poor pain control, subjects will be allowed access to rescue medication for analgesia (Paracetamol 500-1000 mg). Time to REMD (rescue) with an alternative analgesic, if it occurred, will be recorded. Subject will be encouraged to postpone the rescue medication until after 1 h post dose. If Paracetamol 500-1000 mg is not effective, the patient will be allowed to take another dose of Paracetamol 500-1000 mg every 6-8 hours; maximum daily dose is 4000 mg.
- 6. Height will be registered as reported by the patient.
- 7. Patients should mark actual time points of VAS measurement. Deviations from planned time points will not be considered as protocol deviations. Only omitted values will be considered as protocol deviations.


## 3.2. Rationale of the study design

This is a multicenter, double blind, randomised, parallel groups study to assess the efficacy and tolerability after single oral administration of Ketoprofen lysine salt 40 mg granules versus Placebo in male and female subjects with acute pain syndrome after removal of a molar tooth.

This proposed study has been designed to demonstrate the efficacy and safety of OKITASK® 40 mg granules for oral administration in a model of mild and moderate pain. Extraction of molar tooth is an acute surgical pain model that allows collecting the data for the pain profile at a clinical site within a specific timeline [2]. Demonstration of superiority of the study drug vs. placebo serves as a confirmation of the sensitivity of the pain model.

Demonstration of efficacy and safety of OKITASK<sup>®</sup> 40 mg granules as part of the clinical dossier for registration of the new formulation of KLS in Russia was chosen as the most relevant study design. Bioequivalence data for the drug is available from the study of OKITASK<sup>®</sup> 40 mg granules vs OKi® granules for oral solution conducted in 2015 in Switzerland [9].

The multicenter, double-blind, randomized, parallel groups, placebo-controlled study design is a standard design of adequate and well-controlled studies.

OKITASK® is ketoprofen Lysine salt; OKITASK® 40 mg corresponds to ketoprofen 25 mg which is a recommended initial dose for analgesia in OTC indications.

The use of placebo in this model is acceptable and ethically justified since 1) there is no risk to safety and well-being of the patients; 2) rescue treatment will be provided to patients if the study drug or placebo does not provide the sufficient pain relief. Subjects will be encouraged to postpone the rescue medication until after 1 hour post-dose. Paracetamol 500-1000 mg is chosen as a rescue medication as it belongs to a different pharmaceutical group of analgesics to avoid any drug interactions. If not effective, the patient will be allowed to take another dose of Paracetamol 500-1000 mg every 6-8 hours; interval between dose taking is not less than 4 hours; the maximum daily dose is 4000 mg.

The pain relief after the molar tooth extraction will be assessed in this study. As pain is always subjective, self-assessment scales provide the most valid measure of the experience. At present no validated objective measures are available that would be feasible in clinical trials. Pain intensity (PI) is still the key measure of efficacy of an analgesic drug and will be reported in this study. Visual analogue scale (VAS) will be used in this study to assess the pain intensity and pain relief. Primary endpoint will be the  $AUC_{0-6h}$  of pain profile between time 0 (baseline value of VAS) and 6 hours post-treatment. The 6-hour assessment timeline corresponds to PK profile of KLS with  $T_{max}$  within 0.75-1 hour and  $T_{1/2}$  of 1.5-2 hours.

Time profile of pain and time profile of pain relief using VAS, time to first perceptible relief (TFPR) and time to meaningful pain relief (TMPR), proportion of patients requiring rescue medication, time to rescue medication, and patient's overall assessment will be assessed in this study as secondary endpoints. TFPR and TMPR will be measured by two stopwatches.

KLS is supposed to be safe. Patients will be followed for 48 hours post-dose which exceeds 7 half-lives of KLS. Any SAE spontaneously reported by the patient within 30 days of dosing will be collected.

The study hypothesis and sample size are based on data from a placebo-controlled study of ketoprofen (difference between the groups in mean AUC of 90 mm h<sup>-1</sup> and SD of 121 mm h<sup>-1</sup>),  $\alpha = 0.05$  and power of 80% [3].

#### 3.3. Study duration

The duration of participation of each subject in the study will be up  $7\pm1$  days and will include: screening (up to 4 days), tooth extraction, randomization and study treatment (1 day), and follow-up (2 days).


Start of subjects' enrollment in the study is scheduled for October 2017. It is planned that all subjects will complete all study visits before March 2018.

The End of Study is defined as the date of the last visit of the last patient. The Clinical Study Report will be completed in June 2018.

## 3.4. Previous experience with OKITASK®

Pain is the most common symptom for which subjects seek medical attention. Although there is no exact definition of pain it can be defined as an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage (IASP). Acute and chronic pain are different clinical entities. Acute pain is provoked by a specific disease or injury, serves a useful biologic purpose, is associated with skeletal muscle spasm and sympathetic nervous system activation, and is self-limited [6].

NSAIDs have an established role in the relief of mild to moderate pain, minor febrile conditions, and for acute and chronic inflammatory disorders such as osteoarthritis, rheumatoid arthritis, juvenile idiopathic arthritis and ankylosing spondylitis. Acetylsalicylic acid, diclofenac, ibuprofen and naproxen are well known NSAIDs and proven medications in the self-management of conditions with mild to moderate pain and fever. The fastest acting of these active moieties, in an oral OTC formulation, reaches its peak plasma concentrations ( $T_{max}$ ) 20 – 60 minutes (diclofenac potassium tablets), the  $T_{max}$  values, along with the onset of pain relief, vary considerably with the  $T_{max}$  for naproxen being 2 to 4 hours. The current formulations and presentations are limited, with most requiring water in order to administer. There is a need for an OTC analgesic which is fast acting with a unique "on-the-go" formulation.

Ketoprofen, a derivative of propionic acid, is a well-known and established NSAID with proven analgesic, anti-inflammatory and antipyretic actions. It was first approved for clinical use in France and the United Kingdom in 1973. It is currently marketed throughout the world in a variety of forms such as capsules, granules, injectable solutions, suppositories, and topical gel [7].

It is frequently prescribed for the treatment of musculoskeletal and joint disorders such as ankylosing spondylitis, osteoarthritis, and rheumatoid arthritis, and in peri-articular disorders such as bursitis and tendinitis. It is also used in dysmenorrhea, postoperative pain, in painful and inflammatory conditions such as acute gout or soft-tissue disorders, and to reduce fever.

As an 'over the counter' medicine, ketoprofen is approved for the treatment of a range of mild to moderate pain conditions and relief of fever [8].

The chemical name of ketoprofen is 2-(3-benzoylphenyl)-propionic acid and the molecular formula is  $C_{16}H_{14}O_3$ . The assigned ATC Code for ketoprofen is M01AE03. There are pharmacopoeial preparations of ketoprofen products such as BP 2014: Ketoprofen Capsules; Ketoprofen Gel; USP 36: Ketoprofen Extended-Release Capsules.

Ketoprofen lysine salt (KLS) is a salt of ketoprofen, proven to exert the same anti-inflammatory, analgesic, and the antipyretic activities of the parent compound, ketoprofen. The salification of ketoprofen with the amino-acid lysine significantly increases the solubility of ketoprofen in water; improving both the rate and extent of absorption (T<sub>max</sub> 15 minutes) compared with conventional acid ketoprofen, as well as current OTC NSAIDs; studies have reported that the lysination of the compound promotes a gastroprotective effect, and this is supported by KLS post-marketing data whereby there have been fewer GI reactions reported than ibuprofen and, therefore this has provided the basis for the development of orodispersible granules for oral administration [10].


KLS is formulated as 40 mg granules is equivalent to 25 mg of ketoprofen which has been documented to be the dose demonstrating efficacy with a positive benefit:risk profile for an OTC ketoprofen formulation. The content of the sachet is placed directly on to the tongue.

The granules dissolve in saliva and can therefore conveniently be used without water, offering a palatable alternative to people who have difficulty swallowing conventional tablets and capsules. The KLS 40 mg granules formulation has been shown to be effective in controlling mild to moderate pain, with onset of pain relief in 5 minutes.

The indications approved in Italy as per SmPC [50] for KLS 40 mg granules are: pain of various types and origins, in particular: headache, toothache, neuralgia, menstrual pain, rheumatic pain and muscle aches.

KLS is indicated in adults and adolescent aged 15 years or above.

The proposed dosage is 40 mg of KLS (equivalent to 25 mg of ketoprofen) up to 3 times per day in adult and adolescent over 15 years.

All the proposed indications are characterized by a short duration, acute pain and can be self-diagnosed.

#### 3.4.1. Preclinical Data

KLS in terms of acute exposure resulted in a significant high dosage in rats and mice when treated orally or by intraperitoneal route (mean LD50 > 100 mg/kg rat, and > 400 mg/kg mice) [11], [12], [13], [14], [15].

The pharmacology studies and literature demonstrate that KLS possesses the antiinflammatory, analgesic and antipyretic activities described previously for the parent compound, KA, and support the therapeutic indications of the product under application (KLS 40 mg orodispersible granules).

In a study in the model of carrageenan-induced edema of the rat's paw, KLS administered either topically as foam formulation on the skin or given by oral route at the doses of 0.5, 1 and 2 mg/kg (one hour before the carrageenan injection) statistically significantly reduced the edema formation with the highest effect obtained with the 2 mg/kg KLS oral administration.

In a further study (assessing the anti-pyretic activity in the rat), KLS given orally at doses up to 3 mg/kg determined a dose-related inhibition of pyresis induced by yeasts (the highest antipyreticactivity was obtained with 3 mg/kg). In an in vitro model of ethanol-injured gastric mucosa of human cultured cells, Lysine and KLS but not KA clearly protected the cells viability affected by ethanol as well as both Lysine and KLS reduced the levels of malonyldialdehyde (MDA) induced by ethanol as well as the up regulation of NFkB and IL-8. MDA was not reduced by KA which only at a lesser extent it reduced the up regulation of NFkB and IL-8. These in vitro results clearly demonstrated the protective role of Lysine and the better tolerability profile of KLS compared to KA [18].

The pharmacological effects obtained in the different animal models as well as the in vitro data clearly support the intended clinical use and proposed dosing of KLS by orodispersible granules.

The absorption of KLS has been investigated in animals after oral (dog) and topical (cutaneous) application of a foam formulation. In the dog, the bioavailabily and pharmacokinetics of ketoprofen lysine salt, S-ketoprofen, R-ketoprofen and ketoprofen were compared in a 2-week oral study. At equimolar doses of the active principles, ketoprofen lysine salt and ketoprofen disclosed a similar drug disposition profile in a 2 h time but, the mean plasma levels at the first two sampling points was substantially higher for KLS compared to KA thus clearly suggesting that the onset of the pharmacological activity of KLS might well be earlier.


The topical application of KLS induced negligible plasma concentrations of ketoprofen (ng/ml) when compared with those obtained after intravenous administration ( $\mu$ g/ml); often, these concentrations were lower than the LOQ (i.e. below 0.05  $\mu$ g/ml). It was therefore concluded that after cutaneous application no significant systemic absorption of KLS occurs.

Cardiovascular effects of KLS have been studied in the dog. The compound was well tolerated after intramuscular or intravenous administration up to the doses of 10 mg/kg. Higher doses given by the intravenous route (25 - 50 mg/kg) induced a transient hypertensive effect followed, at the highest dose, by a mild hypotension. In rabbits, KLS, administered by intramuscular route up to the dose of 100 mg/kg, did not produce relevant effects on the cardiovascular system. This safety dose in rabbits when compared to the 120 mg/daily dose of ketoprofen Lysine salt orodispersible in human patients provides a safety factor of 16 fold.

The toxicology of KLS has been thoroughly investigated by single and repeated dose toxicity studies covering up to 13-week treatment duration. Genotoxicity, reproductive toxicity and local tolerance studies were also performed. Different administration routes (including the oral route) have been studied in animals in both rodent and non-rodent species. All the studies have been carried out by recognized Life Science Research Organizations (Ricerche Biomediche RBM, in Italy and Life Science Research in Israel), and all performed in compliance with the GLP procedures [11], [13], [14], [15], [16], [17], [18], [19], [20], [22], [21], [23], [24], [25], [26], [27], [28], [48].

The main target organs in all tested species were the GI tract and the kidneys as expected for a NSAID. The doses of 2.5 mg/kg/day and 7.5 mg/kg/day in the rat and marmoset, respectively, were the doses which proved to be devoid of toxic effects. These results are similar to those reported in published toxicological studies conducted with KA in rats and in non-rodent species.

The mutagenic and genotoxic potential of KLS was evaluated according to a standard package of in vitro and in vivo studies. No genotoxic and mutagenic activity was found for KLS.

No teratogenic effects or effects on the fertility or reproduction performances were observed in rabbits at the oral doses of 15, 30, 60 mg/kg/day. Some deaths occurred, possibly accounted for by gastrolesive effect of the compound.

Based on the pharmacological and toxicological data obtained, the non-clinical data of KLS confirms the similar preclinical profile of the compound to that of KA, and is fully supportive of the proposed strength and indications in humans. The potentially enhanced tolerability profile (as well evidenced in an in vitro study with human gastric mucosa cells), faster onset of action and optimized product format make it particularly suited to use in an OTC setting.

#### 3.4.2. Clinical Data

#### **Absorption and Distribution**

As summarised by Sarzi-Puttini, KLS has a higher solubility when compared to acid ketoprofen. This leads to a more rapid absorption of the active substance with a higher peak concentration, which is reached after 15 minutes compared to 60 minutes after ketoprofen administration. This rapid increase in peak plasma concentration of the KLS consequently results in a more rapid pharmacological activity; this is important considering that the speed of onset of analgesia is one of the most important factors for consumers in obtaining pain relief [29].

An analgesic effect-concentration relationship for ketoprofen was established in an oral surgery pain study with ketoprofen. The concentration of ketoprofen that produced 50% the maximum pain intensity difference (PID) (Ce50) was  $0.3 \mu g/ml$  (95% confidence limits: 0.1 to 0.5) [10]. The second biopharmaceutic study conducted on OKITASK 40 mg granules on 69 subjects demonstrated ketoprofen plasma levels measured at 5 minutes were 0.15  $\mu g/ml$  (standard deviation 0.19  $\mu g/ml$ ). Taking into consideration the confidence limits for the Ce50


 $(0.1 - 0.5 \mu g/ml)$ , KLS 40 mg granules can start exerting a clinically relevant analgesic effecting 5 minutes after first oral administration.

Linearity in the absorption kinetic has been demonstrated in the range of doses of ketoprofen between 12.5 mg and 200 mg [30].

When ketoprofen is given with food, the bioavailability (AUC) is not altered, but  $C_{max}$  is lower and  $T_{max}$  is slowed. The size of meal taken appears to have only a slight effect on the extent of ketoprofen absorption [31]. Ketoprofen is 99% bound to plasma proteins and substantial concentrations of drug are found in the synovial fluid [32].

KLS is rapidly and readily distributed into the central nervous system and can be detected in cerebrospinal fluid 15 minutes after administration of a 100 mg intramuscular injection of ketoprofen. The rapid diffusion can be explained by the high level of liposolubility of the KLS quickly passing the blood brain barrier [33].

#### Metabolism

Ketoprofen is rapidly and extensively metabolised in the liver, largely by conjugation. The drug also undergoes hydroxylation and subsequent conjugation with glucuronic acid. The glucuronide conjugate of ketoprofen and the hydroxylated metabolites are pharmacologically inactive, and no active metabolites have been identified.

#### **Excretion and Half-life**

The elimination half-life in plasma is about 1.5 hours. Ketoprofen is metabolised mainly by conjugation with glucuronic acid, and is excreted mainly in the urine [32].

Following a single oral dose of ketoprofen in healthy adults, about 60 - 80% of the dose is excreted in urine; most urinary excretion occurs within 24 h [38]. Elimination of the drug is reduced in the elderly [34], an important point to note when considering the safety of KLS 40 mg granules in this patient population. Age-related accumulation of ketoprofen in the elderly due to reduced clearance was also reported by Skeith and colleagues [35]. Therefore, the SmPC advises that caution should be applied for use in the elderly subjects.

Renal and eventually hepatic impairment reduces renal clearance of ketoprofen acylglucuronide conjugates (CLrconj) in a stereoselective fashion, and this appears to be the rate limiting step for clearance of ketoprofen, which leads to an increased concentration of the drug in the plasma [37], [35], [36]. KLS 40 mg granules is, therefore contraindicated in patients with severe renal or hepatic insufficiency.

#### **Bioequivalence study**

An open-label single-dose crossover study under fasting conditions to determine the comparative pharmacokinetic profile of ketoprofen lysine salt as orodispersible granules (40 mg administered without water) versus ketoprofen lysine salt as granules for oral solution (80 mg bipartite sachet, half sachet, Oki<sup>®</sup> 80 mg) after oral administration in healthy volunteers was performed [9].

Seventy-one (34 female and 37 male) subjects received at least one dose of study treatment (Okitask 40 mg granulates formulation in absence of water and OKi 80 mg granules for solution half sachet with water [240 mL]). After the first treatment administration, one subject withdrew consent to study participation for personal reasons, and one subject was discontinued by the Investigator due to intake of disallowed concomitant treatments during the washout period. So for the pharmacokinetic analysis, 69 subjects were eligible for data contribution (Study population: 34 females and 35 males [mean  $\pm$  SD age 33.6  $\pm$  9.0]).

The healthy volunteers were randomly assigned to receive:


**Test (T)** = **OKITASK® 40 mg granulates** (corresponding to 25 mg ketoprofen): the content of an entire sachet of the test formulation was placed on the tongue and dissolved in mouth during about 3 min in absence of water. The mouth was wet by drinking 20 mL of mineral water directly before placing the granules on the tongue. Afterwards, no fluid intake was permitted for 2 hours.

<u>Reference (R)</u> = OKi® 80 mg granules for solution bipartite sachet: half sachet = 40 mg of ketoprofen lysine salt (corresponding to 25 mg ketoprofen): the content of half sachet of the reference formulation was dissolved in 190 mL of mineral water. The subject drank the entire solution immediately. Then, 50 mL of mineral water were used to rinse the glass and the rinse was drunk immediately. Afterwards, no fluid intake was permitted for 2 hours.

The treatments were administered as a single dose in the morning to fasting subjects (overnight), and after 4 hours post-dose a standardised lunch was provided.

In each study period, blood samples were collected from the volunteers for assay of ketoprofen at the following times: (pre dose, 0) and at 0.08 (5 min), 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0, and 8.0 hours after dose.

Ketoprofen plasma concentrations were determined by means of a validated HPLC-UV method.

In line with the current European Guidelines, the pharmacokinetic (PK) parameters:  $AUC_{0-t}$ ,  $AUC_{0-\infty}$  and  $C_{max}$  were measured and analysed using analysis of variance (ANOVA). The data were transformed prior to analysis using a napierian logarithmic transformation. The statistical method for testing for bioequivalence (BE) was based upon the 90% confidence intervals (CIs) for the ratio of the population means (test/reference) for the PK parameters under consideration. This method is equivalent to the corresponding two one-sided test procedure, with the null hypothesis of bioequivalence at the 5% significance level (Schuirmann's two one-sided t-tests were used). The acceptance criterion for BE was that the 90% CIs of the ratio of geometric means was within the range 80.00-125.00%.

The statistical analysis took into account treatment, period, sequence, and subject within sequence, as fixed effects. Tmax was analysed using the non-parametric Friedman test.

The emergent pharmacokinetic profiles of the test product (OKITASK<sup>®</sup> 40 mg granulates) and reference (OKi 80 mg granules for solution, half sachet) indicated that both formulations are rapidly adsorbed, with a  $t_{max}$  of about 0.5 hour, and both produced a similar ketoprofen exposure.

With respect to the 90% confidence interval of the ratio (test/reference) of geometric means, all the values for each PK parameter were contained within the accepted range (80-125%) for bioequivalence. It can, therefore be concluded that OKITASK® 40 mg granulates, administered without water, are bioequivalent to OKi 80 mg granules for solution (half sachet: 40 mg) administered with 240 mL of water, in terms of both the rate ( $C_{max}$ ) and extent (AUC) of systemic ketoprofen absorption.

The summary pharmacokinetic and bioequivalence assessment data from the study KSL0112 are presented below.

Table 2. Study KSL0112 Summary Pharmacokinetic Data and 90% Confidence Intervals

| Treatment | Cmax (μg/ml) | Tmax (h) | AUC0-t<br>(μg.ml/h) | AUC0 <sub>-∞</sub> (μg<br><sub>"</sub> mL/h) | t½<br>(h) |
|---|---|---|---|---|---|
| T | $2.77 \pm 0.82$ | $0.46 \pm 0.19$ | $4.82 \pm 1.02$ | $4.93 \pm 1.07$ | $1.66 \pm 0.23$ |
| R | $3.16 \pm 0.75$ | $0.30 \pm 0.13$ | $4.62 \pm 1.08$ | $4.77 \pm 1.13$ | $1.87 \pm 0.31$ |
| Statistical Analysis | | | | | |


| 90% confidence interval ratio of geor | Estimate | Lower | Upper | |
|---------------------------------------|----------|--------|--------|--------|
| Treatment T vs R | AUC0-t | 104.71 | 102.63 | 106.84 |
| | AUC0₋∞ | 104.61 | 102.46 | 106.80 |
| | Cmax | 86.28 | 82.24 | 90.52 |

The graph below clearly shows that the ketoprofen plasma concentration versus time profiles for the two treatments evaluated in study KSL0112 are virtually superimposable.



Figure 1. Mean plasma ketoprofen concentration ( $\mu g/mL$ ) vs. time profiles after administration of 40 mg ketoprofen lysine salt orodispersible granules (T) ( $\bullet$  solid line) and 40 mg of ketoprofen lysine salt granules for oral solution (R) ( $\Box$  dotted line) in semilogarithmic scale.

The secondary endpoint of the study was the evaluation of the safety. No deaths or severe treatment emergent adverse events or serious adverse events occurred during the study period. Both test and reference formulations were well tolerated by study subjects. Ten (10) out of 71 subjects (14%) experienced one adverse event (AE) each. Specifically, 8 subjects (11.3%) experienced one AE after the test treatment and 2 subjects (2.9%) after the reference treatment administration. The Investigator judged 5 of the 10 reported AEs were related to treatment. Specifically, 4 subjects (5.6%) experienced one AE after test and one subject (1.4%) after reference administration. The most frequently reported AE was headache, which was experienced by 3 subjects (4.2%) receiving the test treatment. Other reported AEs occurred at a frequency not higher than one subject. No clinically meaningful effect of ketoprofen on vital signs, body weight, ECGs, or standard laboratory test parameters was observed.

In conclusion, OKITASK® 40 mg granulates, administered without water, are bioequivalent to OKi 80 mg granules for solution (half sachet: 40 mg), when administered with 240 mL of water, in terms of both the rate (Cmax) and extent (AUC) of systemic ketoprofen absorption in healthy male and female volunteers.


## **Pregnancy and Lactation**

The use of NSAIDs may reduce female fertility and it is not recommended in women planning pregnancy as with any medication inhibiting cyclo-oxygenase/prostaglandin synthesis. The administration of NSAIDs should be discontinued in women with fertility disorders or who are undergoing investigations of infertility.

NSAIDs can cross the placenta; exposure to NSAIDs in early pregnancy increases the risk of miscarriage and malformation of the foetus, and is believed to increase with dose and duration of therapy. The inhibition of the prostaglandin synthesis [39], [40], [41], [42] by all prostaglandin synthesis inhibitors may affect the unborn child, with exposure during the third trimester of pregnancy increasing incidence of premature closure of the foetal ductus arteriosus in utero, renal dysfunction that may progress to renal failure with oligo-hydroamniosis, prolonged gestation, dystocia and delayed parturition [43], [44], [45], [46]. Therefore, as with all NSAIDs and in accordance with guidance document EMEA/12148/04 [49], the use of KLS 40 mg granules is contra-indicated in the third trimester of pregnancy; the use of KLS 40 mg granules is not recommended during the first two trimesters of pregnancy, it is advised that during this period, KLS 40 mg granules should only be used if strictly necessary.

Ketoprofen can be detected in breast milk after administration. In a three day post-partum study, nursing mothers received 100 mg ketoprofen, as an IV bolus, every 12 hours. Milk samples were collected between the third and fourth doses. Analysis of these samples and extrapolation of the results indicate that a breast-fed infant would receive a mean dose  $8.5 \pm 5.5$  µg/kg/day, and a maximum dose of  $13.6 \pm 7.6$  µg/kg/day. The relative infant dose is  $0.31 \pm 0.17\%$  of the weight-adjusted maternal dose. In this study the relative infant dose of ketoprofen was less than that of the other drug studied, nalbuphine  $(0.59 \pm 0.27\%)$ .

The authors concluded that breast-feeding is permissible when nursing mothers are taking ketoprofen to treat post-partum pain. Nevertheless the use of KLS 40 mg granules is contraindicated during lactation as reported in the SmPC.

#### **Patient Exposure to KLS**

KLS products are authorised and marketed by Dompé farmaceutici S.p.A. with four different brand names: "Artrosilene, OKi, OKi Infiammazione e Dolore and OKITASK".

Dompé farmaceutici S.p.A. received the first marketing authorisation for products containing KLS (systemic formulation) under the brand name **Artrosilene** in Italy, on 13 June 1979 for the pharmaceutical form suppository. Artrosilene is currently authorized and marketed in different countries, in a number of pharmaceutical forms and dosages, by different administration routes for systemic administration, as follows:

- Oral (320 mg prolonged-release capsule, hard),
- Parenteral (160 mg/2 ml solution for injection),
- Rectal (160 mg suppositories).

The above mentioned product presentations were subsequently authorised and marketed in Albania, Kosovo and Russia under the same brand name, by Dompé farmaceutici S.p.A., as Marketing Authorisation Holder (MAH).

Dompé farmaceutici S.p.A. is also MAH of formulations for topical cutaneous use, authorized under the brand name Artrosilene (5 g/100 g cutaneous gel and 15 g/100 ml foam) and marketed in Italy and abroad.

KLS under the OKi<sup>®</sup> brand name was registered by Dompé farmaceutici S.p.A. (formerly Dompé S.p.A.) in Italy on 15 November 1994 and subsequently authorised and marketed in several countries worldwide under different trade names. KLS products under the OKi<sup>®</sup> or


related trade-marks are authorised in a number of pharmaceutical forms and dosages by different administration routes as follows:

- Oral: 80 mg granules for solution, 80 mg/mL drops solution;
- Parenteral: 160 mg/2 ml solution for injection;
- Rectal: 160-60-30 mg suppositories.

Two topical formulations are authorized under the brand  $OKi^{\mathbb{R}}$  Infiammazione e Dolore (1.6% mouthwash; 0.16% oromucosal spray), and are marketed in Italy. The mouthwash is marketed also in Albania, Kosovo, Malta, Russia (with Dompé as MAH) and in Greece and South Korea (with business partners as MAHs).

OKITASK<sup>®</sup> 40mg/sachet granules formulation received the first marketing authorisation in Italy on 17 September 2012; subsequently, almost 3 years later, the same product was authorised in Albania and later in Kosovo. The 40 mg film coated tablet formulation was authorised in Italy in February 2017.

As reported in the Addendum to Clinical Overview of OKITASK® (Data lock point on 16 September 2016) submitted to the Italian Regulatory Agency with the marketing authorization renewal request in December 2016, since first marketing (September 2012) up to 31 August 2016, a total number of 13.067.368 packages of OKITASK® granules has been sold by Dompé in the countries where the product is currently marketed. On the basis of sale data available and of the approved posology, it is assumed that one package is used by one patient, therefore the number of packages sold corresponds to the number of subjects treated. The estimated number of subjects treated cumulatively, up to 31 August 2016, exceeds 13 million.

#### **Adverse Events**

There are long-standing and well-recognised gastrointestinal (GI) and renal safety concerns with all NSAIDs (NICE 2015). In 2006 the European Medicines Agency (EMA 2006) stated that the overall benefit-risk balance for non-selective NSAIDs remains favourable when used in accordance with the product information, namely on the basis of the overall safety profile of the respective non-selective NSAID, and taking into account the patient's individual risk factors (e.g. GI, cardiovascular and renal).

Standard medical textbooks such as Martindale (2015) [32] and Dollery (1999) [47] note that acute interstitial nephritis has been associated with the administration of many NSAIDs including ketoprofen. GI disturbance with ketoprofen is described as common, and comparable in incidence to that produced by other propionic acid derivatives such as naproxen. Non-selective inhibition of prostaglandin synthesis by NSAIDs, including gastro-protective prostaglandins in the GI tract, is the principal reason for GI adverse events [47].

The most common AEs that occurred with KLS in the above presented studies for KLS products (OKITASK® and OKi® 80 mg) involved the GI tract. Typically, these were characterized by short-lasting episodes of gastric pirosis (heartburn) and pain of light severity with a safe profile even though taken on an empty stomach (BE studies). The causality relationship with orally administered OKi® 80 mg granules for solution, which is double the dose of KLS 40 mg granules, was considered possible for all the reported AEs concerning the GI tract. This experience is reflected in published clinical studies where GI adverse events are most commonly reported following oral administration of ketoprofen. GI adverse events with NSAIDs and, therefore with ketoprofen, can manifest as: nausea, vomiting, diarrhoea, flatulence, constipation, dyspepsia, abdominal pain, melaena, haematemesis, ulcerative stomatitis, exacerbation of Crohn's disease and gastritis.


To help reduce the risk of GI adverse effects the lowest effective dose of KLS, 40 mg, was chosen for the product KLS 40 mg granules, moreover the following contraindications and precautions are included in the proposed SmPC for KLS 40 mg granules:

The medicinal product should not be used in the following cases:

- In subjects with an active peptic ulcer, or any history of gastrointestinal bleeding, ulceration or perforation;
- In subjects with gastric or duodenal ulcer, chronic dyspepsia and gastritis. The following precautions must be considered before using the medicinal product;
- The use of KLS 40 mg granules with concomitant NSAIDs, including cyclooxygenase-2 selective inhibitors, should be avoided.
- Undesirable effects may be minimized by using the minimum effective dose for the shortest duration necessary to control symptoms.
- Caution should be advised in subjects receiving concomitant medications that could increase the risk of ulceration or bleeding, such as oral corticosteroids, anticoagulants such as warfarin, selective serotonin-reuptake inhibitors or anti-platelet agents such as aspirin.

## **Post-marketing Safety Data**

Ketoprofen was first approved for clinical use in France and the United Kingdom in 1973. It is currently marketed throughout the world in a variety of forms such as capsules, injectable solutions, suppositories, and topical gel.

Cumulative safety data on OKITASK® granules are taken from the Addendum to Clinical Overview submitted the Italian Regulatory Agency for the marketing authorization renewal request. Cumulatively, up to September 2016, a total of 59 Individual Case Safety Reports (ICSRs) including 119 ADRs, have been reported in subjects treated with KLS 40mg granules during post-marketing use. Among the reported cases, 22 ICSRs (37.3%) were assessed as having at least one serious ADR: cumulatively, the Company received 53 serious ADRs (44.5%) and 66 non-serious ADRs (55.5%). All cases were spontaneously reported in Italy and received either from Regulatory Authority (through the Italian National Pharmacovigilance Network) or from healthcare professional/subjects.

Considering the number of estimated subjects exposed to the drug, the frequency of ADRs (serious and non-serious) is very rare (<1/10,000).

The SOCs most frequently involved in adverse reactions were:

- "Skin and subcutaneous tissue disorders": 35 ADRs were reported under this SOC, of which 15 serious and expected (no unexpected ADR) and 20 non serious reactions.
- "Gastrointestinal disorders": 25 ADRs were reported under this SOC, of which 7 serious and expected (no unexpected ADR) and 18 non serious reactions.
- "Respiratory, thoracic and mediastinal disorders": 18 ADRs were reported under this SOC, of which 13 serious (11 expected/2 unexpected) and 5 non serious reactions.

The majority of the ADRs received were listed allergic reactions, consisting of cutaneous manifestations and/or respiratory or gastrointestinal symptoms, as described in the current version of the SmPC.

Cumulatively, no specific risk was highlighted for the medicinal product: no case with fatal outcome in patients treated was reported. No case of drug-drug interaction, overdose, misuse, off label use was received by the Company. No case report concerning exposure during pregnancy or breastfeeding was collected by the Company. One case of drug abuse (intentional) and one


case of medication error (non-intentional use) were reported, as described above: in both cases no sequelae were mentioned.

## **Safety Conclusions**

The clinical studies show that KLS, and other ketoprofen treatments, are effective and well tolerated in the treatment of the proposed indications for KLS 40 mg granules. The safety profile for ketoprofen (and its lysine salt) is well characterised in clinical studies in over 40 years of use as a POM medicine and subsequently as a non-prescription medicine (OTC). Serious adverse events with short-term oral use of low dose (25 mg) ketoprofen (equivalent to 40 mg KLS) are rare. Adverse reaction data provided for KLS 40 mg granules (OKITASK®) show that the most commonly reported adverse reactions affect the skin and subcutaneous tissue, with the most frequently reported ADR being urticaria.

The most commonly reported adverse events associated with short-term low dose (25 mg) ketoprofen occur in the GI tract, these are well characterised, easily recognised, are mild or moderate in intensity and resolve on cessation of treatment. However, data indicates that short term oral use of low dose KLS (40 mg) has fewer GI tract adverse events than other NSAIDs, this is considered to be due to the optimised rate of absorption. Studies indicate that the salification of ketoprofen with the lysine confers a degree of gastro-protection. Consumption of KLS with food to minimise GI adverse events is not necessary in short-term KLS use.

This clinical experience is adequately reflected in the corresponding SmPC and product labelling for KLS 40 mg granules. The available safety data for KLS, and other ketoprofen treatments, support short-term self-medication with orally administered KLS 40 mg up to 3 times a day, in adults over the age of 18 years.

In summary, the symptomatic benefits of KLS 40 mg granules, for an adult consumer of this medicine, far exceed the known risks.

#### 3.5. Dose Rationale and Risk/Benefits

The proposed dosage of KLS granules in this study is a single dose of 40 mg of KLS (equivalent to 25 mg of ketoprofen). This dose is one third of the daily dose authorized in Italy (adults and adolescents over 15 years: 1 sachet as a single dose or repeated 2 to 3 times a day, for more intense pain) and in the European countries (i.e. up to 3 times per day in adults above 18 years), 1 sachet as a single dose repeated 2 to 3 times a day as needed.

KLS has been widely used in clinical practice for over 35 years and as such, there is extensive experience with the drug.

No particular safety risks are foreseen with respect to the safety profile of the marketed  $OKITASK^{®}$  40 mg granules.

The presentation of OKITASK<sup>®</sup> granules in a single sachet delivers easy compliance for subjects due to the formulation, which can be conveniently swallowed without water and also by subjects who usually experience difficulties in swallowing tablets or capsules. Adequate warnings are provided in the product labelling for KLS 40 mg granules to ensure this product is self-administered correctly and safely.

Considering that planned KLS dose is 40 mg in single, no concern for the safety of study participants is expected.

The use of placebo in the study is acceptable and ethically justified since 1) there is no risk to safety and well-being of the patients; 2) rescue treatment will be provided to patients if the study drug or placebo does not provide the sufficient pain relief. Subjects will be encouraged to postpone the rescue medication until after 1 hour post-dose. Paracetamol 500-1000 mg is chosen as a rescue medication as it belongs to a different pharmaceutical group of analgesics to avoid any drug interactions. If Paracetamol 500-1000 mg is not effective, the patient will be allowed to


Dompé farmaceutici s.p.a. September 26, 2017 (As amended on January 25, 2018)

take another dose of Paracetamol 500-1000 mg every 6-8 hours; interval between dose taking is not less than 4 hours; the maximum daily dose is 4000 mg.

This study is considered as a low risk interventional trial considering that it is conducted with an authorized medicinal product tested in accordance with its marketing authorization in some European countries.


#### 4. STUDY POPULATION

### 4.1. Study population

Up to 100 male and female adult patients scheduled for extraction of a molar tooth will be screened in the study. 70 eligible patients will be randomized into one of two study groups at 1:1 ratio:

Group 1. OKITASK® 40 mg – 35 patients

Group 2. Placebo – 35 patients

#### 4.2. Inclusion Criteria

Eligible patients must meet the following inclusion criteria:

- 1. Signed Informed Consent Form;
- 2. Male and female, from 18 years to 65 years (inclusively);
- 3. Subjects who undergo removal of a non-impacted molar tooth within 3 hours before randomization in the study;
- 4. Subjects in generally good health (based upon criteria for safe administration of outpatient conscious sedation);
- 5. Subjects requesting relief for postoperative pain within 3 h after the tooth extraction  $(VAS \ge 30 \text{ mm})$ ;
- 6. Subjects willing to undergo observation period for up to 9 hours after the tooth extraction;
- 7. Ability to complete a 100 mm VAS and a category scale during the observation period (about 9 hours);
- 8. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study;
- 9. Contraception (for females): females of child-bearing potential must be using at least one reliable method of contraception during the study, as follows:
  - a. hormonal oral, implantable, transdermal, or injectable contraceptives;
  - b. a non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide;

### or should have:

- c. a male sexual partner who agrees to use a male condom with spermicide;
- d. a sterile sexual partner.

### 4.3. Exclusion Criteria

Patients will not be enrolled in the study if they have any of the exclusion criteria listed below:

- 1. Subjects undergoing extraction of impacted and dystopic teeth, tooth preserving operations, apically positioning flap/vestibuloplasty with free gingival graft from the palate;
- 2. Subjects undergoing more than one tooth extraction in the same extraction procedure;
- 3. Subjects undergoing dental implantation simultaneously with tooth extraction;


- 4. Allergy: ascertained or presumptive hypersensitivity to the active substances (ketoprofen and paracetamol as rescue medication) and/or formulations' ingredients; history of hypersensitivity to drugs (in particular to NSAIDs) or allergic reactions in general, which the Investigator considers may affect the outcome of the study;
- 5. Diseases: relevant history of renal, hepatic, cardiovascular, respiratory (including asthma), skin, haematological, endocrine, gastro-enteric and genitourinary tract or neurological and autoimmune diseases, that may interfere with the aim of the study;
- 6. Medications: non-steroidal anti-inflammatory drugs (NSAIDS) and other analgesics [in particular ketoprofen, paracetamol and acetylsalicylic acid (ASA)], antihistamines, sedating medications, including herbal and BASs, taken 48 h before surgery;
- 7. Investigational drug trials: participation in the evaluation of any drug within 3 months before screening (including the last study procedure);
- 8. Relevant history of drug and alcohol abuse.
- 9. Positive Pregnancy test in female patients of childbearing potential (including patients in post-menopausal status for less than 2 years).

### 4.4. Re-screening procedures

Patients may be rescreened if the extraction procedure is postponed or cancelled outside from the window Day -4 – Day 1. In this case the subject should sign new Informed consent form, new patient's number should be assigned and all the screening procedures will be repeated.

Patients may not be rescreened for the second extraction of molar tooth or participate in the study twice.


### 5. STUDY DRUG

## 5.1. Description

| Study Drug: | OKITASK® 40 mg granules |
|---|---|
| Active substance: | Ketoprofen Lysine Salt |
| | Ketoprofen: 2-(3-benzoylphenyl)-propionic acid; |
| | C <sub>16</sub> H <sub>14</sub> O <sub>3</sub> ; CAS 56105-81-8; MW 254.29 |
| | Lysine: 2,6-diaminohexanoic acid; |
| | C <sub>6</sub> H <sub>14</sub> N <sub>2</sub> O <sub>2</sub> ; CAS 70-54-2; MW 146.19 |
| Pharmacotherapeutic group: | Non-steroidal anti-inflammatory drug, propionic acid derivatives. |
| | ATC code: M01AE03 |
| Pharmaceutical form and | Granules for oral administration. |
| composition: | Composition Ketoprofen Lysine Salt, Povidone K-25, Silica (colloidal anhydrous), Hypromellose, Basic Butylated Methacrylate Copolymer (Eudragit EPO), Sodium laurilsulfate, Stearic Acid, Magnesium Stearate, Lime Flavor, Lemon Flavor, Frescofort Flavor, Aspartame, Mannitol, Xylitol, Talc |
| Presentation: | Granules in sachet. |
| | Sachet: opaque, PE/aluminum/PET sachets containing 700 mg of granules (40 mg ketoprofen lysine salt) |
| Daily dose KLS | 40 mg |
| Dosing regimen: | Single dose - 1 sachet |
| Storage conditions: | Keep at temperature not higher than +25°C |
| | Keep in a place, out of reach of children |
| Manufacturer: | Dompé farmaceutici S.p.A. (Italy) |
| Re-packaging (primary, secondary including labeling) | Monteresearch (Italy) |
| Batch control and release | Dompé farmaceutici S.p.A. (Italy) |

| Comparator product: | Placebo of OKITASK® 40 mg granules |
|---|---|
| Active substance: | None |
| Pharmacological Group: | Placebo |
| Pharmaceutical form and composition: | Granules for oral administration Placebo: Silica (colloidal anhydrous), Magnesium stearate, Lime flavor, Lemon flavor, Frescofort flavor, Aspartame, Mannitol, Xylitol, Talc. |
| Presentation: | Granules in sachet. Sachet: opaque, PE/aluminum/PET sachets containing 700 mg |


| Comparator product: | Placebo of OKITASK® 40 mg granules |
|---|---|
| | of granules |
| Daily dose KLS | 0 mg |
| Dosing regimen: | Single dose (1 sachet) |
| Storage conditions: | Keep at temperature not higher than +25 °C |
| | Keep in a place, out of reach of children |
| Manufacturer (primary, secondary including labeling): | Monteresearch (Italy) |
| Batch control and release | Dompé farmaceutici S.p.A. (Italy) |

### 5.2. Treatment Regimen

A single oral dose of OKITASK® 40 mg or Placebo will be administered to patients within 3 hours after extraction of a molar tooth (VAS  $\geq$  30 mm). Each patient will receive one sachet that contains KLS 40 mg (equivalent to 25 mg of ketoprofen) or Placebo. The content of the entire sachet will be placed on the patient's tongue and swallowed. The study drug dissolves in saliva, thus water may be not required.

#### 5.3. Randomization and blinding

This is a double-blind placebo-controlled study. Patients will be assigned to one of two treatment groups by the IWRS system in 1:1 ratio:

Group 1. OKITASK® 40 mg – 35 patients

Group 2. Placebo – 35 patients

Randomization will be performed after the surgery upon confirmation of the inclusion/exclusion criteria (VAS  $\geq$ 30 mm).

The double-blinding is provided by Placebo that is identical to OKITASK® 40 mg granules. The drug will be packaged and labeled in a manner that will exclude unblinding. IWRS will assign the study drug kit number that should be administrated by the subject. Randomization and IWRS manual will be provided to the Investigator before the beginning of the study.

#### 5.4. Unblinding procedure

The code of a particular subject may be broken in a medical emergency if knowing the identity of the treatment allocation would influence the treatment of the subject. Administration of rescue therapy does not require code break.

Unblinding of a patient's treatment may be performed in IWRS. The reason for breaking the code must be documented in the source documentation. If possible, Medical Monitor should be contacted before the code is broken; otherwise the Medical Monitor should be notified within 24 hours of breaking the code.

### 5.5. Study treatment compliance

The patients will take the study drug once in front of the Investigator. No specific drug compliance assessment is proposed in the study.

### 5.6. Packaging and labelling

The study drug will be provided by the Sponsor. The study drug will be packed and labeled according to the current Russian legislation and applicable requirements.


Labeling of the box containing the sachet is shown in Figure 2.

### Figure 2 Labeling of the box containing the sachet.

Labeling of the sachet is shown in Figure 3.

Figure 3 Labeling of the sachet

For clinical trial only - Clinical trial N° KSL0117

KIT # XXX\* OKITASK® 40mg granules or Placebo

Dosage: 1 sachet 40 mg or 0 mg of ketoprofen lysine salt

CRO: IPHARMA LLC Russia, tel. + 7 (495) 276-1143

Batch: XXXXXX Expired date: XXXXXX

Keep out of reach of children

\*Kits numbers will be prepared, according to the randomization drug list, and numbered from 001-150.

#### 5.7. Study drug accountability

The Investigator will be responsible for keeping records on study drug accountability to ensure the proper receipt, storage, distribution and return of the study drug. Used sachets will be stored at the site for accountability, monitoring and confirmation of administration to patients. In case of a sachet damage during administration that prevents the subject from study drug dosing, the appropriate entry must be made in the source documents and the accountability log, and the sachet must be replaced by IWRS.

### **5.8.** Study drug storage

Investigator will be responsible for ensuring adequate acceptance, storage, distribution and return of the study drug, as well as keeping inventory records and registration in IWRS.

Limited access and applicable temperature regimen should be ensured by the Investigator. The study drug should be stored at room temperature not exceeding +25°C. Temperature control should be performed using thermometers, registering minimum and maximum temperature within the reporting period. Information of temperature monitoring should be regularly entered into the temperature monitoring log (i.e. every day excluding weekends and holidays).

### 5.9. Concomitant and rescue therapy

All concomitant medications, including herbal therapy and biologically active supplements (BAS) must be registered in the source documentation and on the eCRF. This includes all pharmaceutical products and BAS

The concomitant therapy also includes anesthesia and rescue therapy allowed by the protocol which is applied to relief pain (if applicable).

Ultracain D (articaine 40 mg), Ultracain DS forte (articaine+epinephrine 40 mg+0.01 mg/ml), Ultracain DS (articaine+epinephrine 40 mg+0.005 mg/ml) 1-2 capules can be used for anesthesia. The Investigator can choose anesthesia taking into consideration the patient's condition, medical history and other reasons. Number of used capules and type of anesthesia for each patient will be recorded in the source documentation and on the eCRF.

In the event of poor pain control, the patient will receive a rescue medication for analgesia (i.e. Paracetamol 500-1000 mg tablets). Subjects will be encouraged to postpone the rescue medication until after 1 hour post-dose. If Paracetamol 500-1000 mg is not effective, the patient will be allowed to take another dose of Paracetamol 500-1000 mg every 6-8 hours; interval between dose taking is not less than 4 hours; the maximum daily dose is 4000 mg.

The drug name (preferably the name of the active substance), dosage, frequency of administration, route of administration, indication for use (including the underlying disease,


comorbid conditions, adverse event, or prevention), the date of beginning and ending of a concomitant drug administration should be registered in the source documentation and on the electronic Case Report Form.

If by the time of the study completion the concomitant therapy continues, a corresponding mark shall be entered on the electronic Case Report Form.

### 5.10. Prohibited prior and concomitant therapy

Prohibited medicines which should not be taken within 48 hours before screening and during Day 1:

- Antihistamines;
- Sedating medication (including herbal therapy and BAS).

Prohibited drugs should not be taken during Day 1:

- Medicines for anesthesia other than indicated by the protocol (e.g. procaine, lidocaine);
- NSAIDs and combinations which contain NSAIDs (except for the study drug);
- Analgesics: opioids, acetylsalicylic acid and its derivate, pyrazolones, other analgesics-antipyretics (except for the rescue therapy indicated by the protocol, if applicable);
- Antithrombotic medicines;
- Hemostatic sponge.

Participation in the evaluation of any investigational product within 3 months before screening and during the study is also prohibited.


#### 6. STUDY PROCEDURES

All study procedures will be performed according to the requirements and recommendations of the Good Clinical Practice guidelines of International Conference for Harmonization (ICH Topic E6 (R2) Guideline for Good Clinical Practice (EMA/CHMP/ICH/135/1995 – 1 December 2016)) and Eurasian Economic Union (EAEU), principals outlined in the Declaration of Helsinki, as well as according to the current legislation and applicable regulations of Russian Federation. The Investigator must consent to accept monitoring, audits and inspections at the clinical site and provide direct access to the study materials to the Sponsor and its representatives, Independent Ethics Committee and regulatory authorities.

### 6.1. Informed Consent

Informed consent will be obtained at screening before any study-related procedure. One copy of the signed informed consent form will be provided to the patient, the second signed copy will remain at the site with the patient's study records.

### **6.2. Patients registration**

| Each patient signed the Informed Consent Form will be assigned the individual registration |
|---|
| number that consists to four digits: \[ \] \[ \] - \[ \] - the first two digits correspond to the site |
| number, the second two digits correspond to the patient's order number at this site (01, 02, 03, |
| etc.). Then the randomistion number will be assigned by the IWRS. It consists in R and two |
| digits (R \( \sum \sum).\) The investigator will report this number on the label of the kit assigned to the |
| patient (see section 5.6). |

The instruction for registration of patients in IWRS will be provided to the Investigator before beginning of the study.

### 6.3. Demographic data and medical history

To assess the patient's compliance with the inclusion/exclusion criteria, the patient's demographic data (sex, date of birth/age, race) and full medical history, including significant acute and chronic disorders and conditions (e.g. post-menopause), surgical interventions and allergic reactions should be collected. Besides, patient should be asked about hospitalizations and/or surgical interventions scheduled within the study period (if applicable). All new diagnoses and conditions detected at screening should be attributed to the patient's medical history.

### 6.4. Oral cavity examination

Oral cavity examination includes assessment of general appearance, condition of mucous membranes, teeth, and throat.

Changes from baseline characteristics which are considered AEs, should be reported in the source documentation and in the eCRF.

### 6.5. Vital signs, weight and height

The examination includes measurement of blood pressure, pulse and respiratory rate after 10 minutes rest in a sitting position. Changes from baseline characteristics which are considered AEs, should be reported in the source documentation and in the eCRF.

Weight will be measured without shoes. Height will be captured as reported by the patient.

#### 6.6. Assessment scales

Assessment scales are presented in Appendix (Section 12).

### 1) Pain intensity

Pain intensity will be assessed by Visual Analogue Scale (VAS), consisting of a 100 mm long scale ranging from 0 mm (no pain) to 100 mm (worst pain imaginable) [Section 12.1]. The


patient will be asked to put a mark on his/her scale based on the current intensity of pain symptoms.

The Investigator should measure the distance from 0 to the mark on the scale with a standardized ruler and capture the result in the source documentation and on the electronic Case Report Form.

### 2) Pain relief

Pain relief will be assessed by Visual Analogue Scale (VAS), consisting of a 100 mm long scale ranging from 0 mm (no relief) to 100 mm (maximum relief) [Section 12.2]. The patient will be asked to put a mark on the scale based on his/her current intensity of pain relief.

The Investigator should measure the distance from 0 to the mark on the scale with a standardized ruler and capture the result in the source documentation and on the electronic Case Report Form.

### 3) Patient's overall assessment

The patient will be asked to provide his/her current overall assessment answering the question «Considering all the ways that the pain affects you, how well are you doing?». The patient will mark the answer on the 5-point scale: 1 = very good, 2 = good, 3 = satisfactory, 4 = poor, 5 = very poor [Section 12.3].

Patient overall assessment will be performed after VAS measurement at baseline and at 6 h. If a patient takes rescue medication, the Patient's overall assessment will be performed after the last VAS measurement (before rescue medication).

The Investigator should capture the score in the source documentation and on the electronic Case Report Form.

# 6.7. Determination of the Time to first perceptible relief (TFPR) and Time to meaningful pain relief (TMPR)

Upon study drug administration the patients will immediately start two stopwatches. One of them will be stopped once the patient feels first perceptible pain relief; the second one will be stopped once the patient feels the meaningful pain relief. Time to first perceptible relief (TFPR) and time to meaningful pain relief (TMPR) will be captured in the source documentation and on the eCRF.

### 6.8. Safety and Adverse Events

#### 6.8.1. Definitions

Adverse Event (AE) - Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, complaint or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. In this study AEs will be reported from the moment of signing the Informed Consent Form (prior to administration of the first dose of the study drug) to the follow-up (Day 3±1) after the last visit of the patient or last procedure per protocol.

#### Post-operative pain will not be considered as AE at the study.

**Adverse Drug Reaction (ADR)** - Any adverse event for which there is a reasonable possibility that the drug caused the adverse event. "Reasonable possibility" means there is evidence to suggest a causal relationship between the drug (at any dose) and the adverse event.

**Serious Adverse Event -** Any untoward medical occurrence that at any dose:


- results in death is life-threatening (i.e. the patient was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it were more severe)
- requires or prolongs hospitalization
- results in significant, persistent or permanent impairment or disability is a congenital anomaly or birth defect
- is an important medical event

Important medical events are those that may not be immediately life threatening, but are clearly of major clinical significance. They may jeopardize the subject, and may require intervention to prevent one of the other serious outcomes noted above. For example, drug overdose or abuse, a seizure that did not result in in-patient hospitalization or intensive treatment of bronchospasm in an emergency department would typically be considered serious.

NOTE: Hospitalization for social reasons, visits to day patient facility, hospitalization or operation preplanned prior to patient enrollment into the study for treatment of underlying condition, are not to be considered SAEs.

Unexpected Adverse Drug Reaction - An adverse reaction, the nature or severity of which is not consistent with the applicable product information (e.g., Investigator's Brochure for an unapproved investigational product or package insert/summary of product characteristics for an approved product) The group also includes ADRs specified in the investigator's brochure as characteristic for the class of products or expected as related to the pharmacological properties of the study product, but which had not been observed earlier.

**Suspected Unexpected Serious Adverse Reaction:** Any suspected adverse reaction that is both serious and unexpected (SUSAR). The determination of expectedness should be made on the basis of the IB.

### 6.8.2. Pregnancy

Women of childbearing potential are not excluded from the study as long as adequate birth control methods are being utilized. Women of childbearing potential are defined as all women physiologically capable of becoming pregnant including women in post-menopausal status for less than 2 years.

To participate to the study, subjects must agree to use adequate contraception measures. Adequate birth control measures include:

- a. hormonal oral, implantable, transdermal, or injectable contraceptives;
- b. a non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide;

or should have:

- c. a male sexual partner who agrees to use a male condom with spermicide;
- d. a sterile sexual partner.

Female participants of non-child-bearing potential or in post-menopausal status for at least 2 year will be admitted. For all female subjects, pregnancy test result must be negative.

Pregnancy is not a SAE, but refers to events that require an urgent reporting to the Sponsor. In case of pregnancy detected up to 30 days after study dosing, either occurring in a female patient or in a male patient's partner, the pregnancy status should immediately be reported to the Sponsor. Female patient will be monitored throughout pregnancy and up to 30 days after its


outcome. Health conditions of any newborn will also be followed up to 30 days after birth (including pregnancy of patient's partner). Relevant information will be recorded in source documents, eCRF and Pregnancy Report Form. Pregnancy reports should be completed and e-mailed/faxed following the procedure described in Paragraph 6.8.7 SAE and Pregnancy reporting.

### 6.8.3. **AE and SAE reporting**

During the study and at follow up visit subjects should report any AEs, in particular responding to open, non-probing questions from the Investigator. The investigators should also collect any SAE spontaneously reported by the patient within 30 days of dosing. For each AE/SAE reported by a patient, the Investigator should collect and document in source documents and eCRF all the needed information, including diagnosis and symptoms, date of onset and date of resolution, outcome, severity, criteria of seriousness, circumstances, that may denote possible relatedness to the study drug and concomitant therapy, underlying diseases or concomitant conditions, study procedures or other causes, actions related to the study drug, pharmaceutical treatment, medical interventions, results of laboratory and instrumental tests for AE, other circumstances, which may add to comprehensive description of the event.

The date of onset of SAE is the date of onset of the seriousness criterion. The preceding condition, if applicable, should be reported as a non-serious AE.

If an AE is serious, Investigator should also promptly submit a SAE report (specifying the seriousness criteria), within 24 hours from first knowledge to the IPHARMA Medical Monitor. Besides, the Sponsor should be provided with certified copies of source documents for that SAE (hospital discharge summary, autopsy report, death certificate, etc.). Data in source document and SAE form shall be duly anonymized.

Whenever more than one SAE is observed, the Investigator should identify which is the primary adverse event, i.e. the most relevant one. If other events are listed in the same report, the Investigator, along with their relatedness to the Investigational Product, should identify which adverse events are serious and which are non-serious. In any case, the Investigator is requested to record his/her opinion about the relatedness of the observed event(s) with the investigational medication.

AEs should be followed up and reported from the date of signing informed consent to the last visit or study related procedure (teleconference at follow-up).

Spontaneously reported SAE will be collected within 30 days after dosing: these events will be reported and assessed in the same way as SAEs occurring during the study.

In line with ICH E2A provisions on Post-Study events, although such information is not routinely sought or collected by the Sponsor, serious adverse events that occurred after the patient had completed a clinical study will possibly be reported by the Investigator to the Sponsor directly. Such "post-study cases" should be regarded for expedited reporting purposes as though they were study reports. Therefore, a causality assessment and determination of expectedness are needed for a decision on whether or not expedited reporting is required.

Monitor is responsible for verifying consistency of eCRF and SAE reports to the source documentation.

It is the Investigator's responsibility to assure that the subjects experiencing an AE receive definite treatment for any AE, if required.


### 6.8.4. Assessment of severity

For each AE the Investigator should assess its severity. For this purpose, the following gradation of the severity will be used:

| 1. Mild | Grade 1 - does not interfere with patient's usual function (awareness of symptoms or signs, but easily tolerated [acceptable]). |
|---|---|
| 2. Moderate | Grade 2 - interferes to some extent with patient's usual function (enough discomfort to interfere with usual activity [disturbing]). |
| 3. Severe | Grade 3 - interferes significantly with patient's usual function (incapacity to work or to do usual activities [unacceptable]) |

For each episode, the highest severity grade attained should be reported.

Note that severe adverse events do not always meet the criteria of seriousness, and, conversely, SAE does not have to be severe AE. Urgency of SAEs reporting does not depend of the severity of the event.

### 6.8.5. Relationship to the Study Drug

For each AE the Investigator should evaluate its possible relationship to the study drug according to the categories shown in the Table below.

| AE Category | Definition |
|---|---|
| 1. None<br>(Intercurrent<br>Event) | An event that is not and cannot be related to the Investigational Product, e.g. patient is a passenger in a road traffic accident. |
| 2. Unlikely (remote) | Relationship is not likely e.g. a clinical event including laboratory test abnormality with temporal relationship to drug administration which makes a causal relationship improbable and in which other drugs, chemicals or underlying disease provide more plausible explanations |
| 3. Possible | Relationship may exist, but could have been produced by the patient's condition or treatment or other cause |
| 4. Probable | Relationship is likely, the AE abates upon discontinuation of Investigational Product and cannot be due to the patient's condition |
| 5. Highly<br>Probable | Strong relationship, the event abates upon discontinuation of Investigational Product and, if applicable, re-appears upon repeat exposure |

#### **6.8.6.** Assessment of Expectedness

Expectedness will be determined based on the contents of the Investigators' Brochure.

| Expected | An adverse reaction, the nature or severity of which is consistent with the applicable product information (e.g. Investigators' Brochure) |
|---|---|
| Unexpected | An adverse reaction, the nature or severity of which is not consistent with information in the relevant source document (e.g. Investigators' Brochure) |

### 6.8.7. SAE and Pregnancy reporting

All SAE irrespective of severity and relatedness to the study drug, as well as pregnancy cases should be reported in English to IPHARMA Medical Monitor and the Dompé Drug Safety, by fax or e-mail, **within 24 hours** from the moment of first knowledge by the Investigator. Information about SAE should be sent in the form of SAE report. Information about pregnancy should be sent in the form of pregnancy report. In case of need, the Investigator may contact the Medical Monitor for consultation or explanations.


Reporting SAE/pregnancy

Company: IPHARMA LLC

Medical Monitor: Victoria Yavorskaya

Tel. +7 (925) 400-01-34

Fax: +7 (495) 276-1147

E-mail: SAE@ipharma.ru

Dompé Drug Safety:

Laura Boga, Safety Manager

Direct line: +39 02 58383462;

Fax: +39 02 36026913

E-mail: farmacovigilanza@dompe.com

IPHARMA Medical Monitor will be then responsible for verifying consistence of information reported and data included in SAE/Pregnancy Report Form, obtaining and reporting any additional information received from the Investigators, and forwarding fully completed SAE/Pregnancy Report Forms to Dompé Drug Safety, by e-mail immediately and anyway within 24 hours of knowledge of event.

Investigator should instruct each patient to report SAE or pregnancy during study and 30 days after the last visit to the study site. Investigator should provide in the SAE/pregnancy report form all information about the event. Each SAE report form should include at least the following information: patient details, event title, seriousness criterion, relatedness to the study drug, and outcome at the time of report.

For primary report the Investigator makes the following remark to the SAE report – "Primary report". If additional information about SAE (for example, new information about patient condition or results of laboratory tests) occurs Investigator should fill in a new form of SAE report with "Additional report" mark. Original of SAE report form should be kept in Investigator File.

The Investigator (or an authorized staff member) will be responsible for reporting any SAEs/SUSARs to the Local Ethics Committee and local institutions in accordance with local regulations and requirements.

The Sponsor shall be responsible to prepare and approve Periodic safety reports and SUSAR report and to forward them the IPHARMA for submission. IPHARMA will be responsible for Periodic safety reporting to the Regulatory Authorities in the Russian Territory and Investigators, and expedited reporting of SUSARs to the local Regulatory Authorities, in accordance with local regulations and requirements. The Sponsor will be responsible for regulatory reporting outside the Russian Territory, as applicable.

### 6.8.8. Overdose

Cases of overdose (accidental or intentional) which may or may not result in serious adverse reactions are to be reported by Investigator to IPHARMA and Dompé Drug Safety, following the same procedure for SAE, within 24 hours from the Investigator's knowledge of its occurrence. This includes reports related to drug intake with suicidal intentions and consequent drug overdose.

An overdose of  $OKITASK^{\circledR}$  is defined as the administration of more than 3 sachets on the given treatment day.


The Investigator shall provide in the SAE form information about symptoms, corrective treatment and outcome of overdose.

### 6.9. Early Withdrawal of Subjects

The patient has the right to withdraw from the study at any stage without giving reasons. The patient should be withdrawn from the clinical study if:

- Patient requires rescue medication (as anticipated by the protocol)
- Patient requires prohibited medications
- Investigator considers it important from the medical point of view
- Patient withdraws his consent
- Patient does not comply with the study related procedures
- AE or SAE which may impact safety or well-being of patient
- Patient is included into the study with violation of inclusion/exclusion criteria or significant protocol deviations that may impact patient's safety and integrity of the study data

If possible, the Investigator should discuss the need to withdraw the subject with the Medical Monitor or inform about subject withdrawal from the study (except discontinuation due to rescue therapy that is anticipated by the protocol). The reason for subject withdrawal (including date and time) should be specified in the source documents and on the eCRF. If a subject withdraws from the study for more than one reason, only the main reason should be specified. If a subject withdraws consent due to AE or SAE, the AE or SAE should be specified as the reason for subject withdrawal.

Besides, the Sponsor may terminate the study at any time. The Investigator has the right to terminate the study at any time for medical or regulatory reasons. Study may only be terminated after mutual consultations between the Investigator and the Sponsor.

SAEs and pregnancy ongoing at the time of study termination should be followed-up per protocol if not agreed otherwise between the Investigator and the Sponsor.

No subjects that will take the study medication and withdrawn from the study will be replaced.


#### 7. STUDY VISITS

### 7.1. Screening (Day -4 to Day 1)

- Procedure for obtaining informed consent
- Assignment of the screening number to the patient
- Collection of demographic data, medical history and underlying disease
- Evaluation of previous and concomitant therapy
- Oral cavity examination
- Vital signs and body weight and height (according to the patient's report)
- Pregnancy test
- Extraction of the molar tooth
- Pain intensity assessment (within 3 hours of the surgery)
- Assessment of adverse events
- Evaluation of inclusion/ exclusion criteria

Screening and surgery may occur in the same day considering that the day of extraction of the molar tooth will be Day 1. Patients may be rescreened if the extraction procedure is postponed or cancelled outside from the window Day -4 – Day 1. In this case the subject should sign new Informed consent form, new patient's number should be assigned and all screening procedures will be repeated.

Patients may not be rescreened for the second extraction of molar tooth or participate in the study twice.

### 7.2. Study treatment (Day 1)

#### Pre-dose

- Assessment of adverse events and concomitant medication
- Randomization and assignment of study drug kit number
- Evaluation of pain intensity by VAS (0 100 mm) at 0' (immediately before dosing).
- Patient's overall assessment (5-point scale)
- Study drug dosing.

Upon study drug administration the patients will immediately start two stopwatches. One of them will be stopped once the patient feels first perceptible pain relief; the second one will be stopped once the patient feels the meaningful pain relief.


#### Post-dose

- Evaluation of pain intensity by VAS (0 100 mm) at 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) post-dose<sup>1</sup>
- Evaluation of pain relief by VAS (0 100 mm) at 5', 10', 15', 30', 45', 60' (1 hour), 90' (1.5 hours), 120' (2 hours), 180' (3 hours), 240' (4 hours), 300' (5 hours), and 360' (6 hours) post-dose<sup>2</sup>
- Patient's overall assessment (5-point scale) after the last VAS assessment
- Assessment of Adverse events and concomitant medications

The patient will be discharged from the clinical site upon completion of all visit procedures.

### 7.3. Early termination (Day 1)

In case of early withdrawal of the patient, the following procedures will be performed (if applicable):

- Evaluation of pain intensity by VAS (0 100 mm)
- Evaluation of pain relief by VAS (0 100 mm)
- Patient's overall assessment (5-point scale) after the last VAS assessment
- Assessment of Adverse events and concomitant medications

The patient will be discharged from the clinical site upon completion of all visit procedures.

In the event of poor pain control, the patient will receive a rescue medication for analgesia (i.e. Paracetamol 500-1000 mg tablets). Subjects will be encouraged to postpone the rescue medication until after 1 hour post-dose. **NB:** If the patient will take the rescue medication the above procedure will be performed prior to administration of rescue therapy.

If Paracetamol 500-1000 mg is not effective, the patient will be recommended to take another dose of Paracetamol 500-1000 mg every 6-8 hours; interval between doses taking is not less than 4 hours; the maximum daily dose is 4000 mg.

### 7.4. Follow-up (Day $3 \pm 1$ day)

• Assessment of adverse events (telephone contact)

### 7.5. Unscheduled visits

At the Investigator's discretion subjects may be invited to an unscheduled visit at any time during the clinical trial for safety reasons, should repeated examination or procedure be required. At unscheduled visits the Investigator may perform the required procedures. Unscheduled visits should be documented in the source documentation and eCRF. Unscheduled visits should not modify the preplanned visit schedule per protocol.


\_

<sup>&</sup>lt;sup>1</sup> Patients should mark actual time points of VAS measurement. Deviations from planned time points will not be considered as protocol deviations. Only omitted values will be considered as protocol deviations.

### 8. QUALITY ASSURANCE

This study is to be conducted according SOPs of IPHARMA LLC, ICH Topic E6 (R2) Guideline for Good Clinical Practice and EAEU, principles outlined in the Declaration of Helsinki, and applicable regulations of Russian Federation. The compliance will be assured by auditing the clinical sites and study data.

The Investigator will enter all applicable study data as described in the protocol into eCRF provided by the Sponsor or its representative. CRAs will visit each clinical sites at a frequency described in the monitoring plan to review eCRFs for completeness and accuracy. For any inconsistency between source documents and completed eCRF queried should be raised, and the Investigator should reply the queries and/or resolve the inconsistencies. Upon completion of eCRFs and resolving all queries, the Investigator should electronically sign and date the eCRF of each patient. Completed eCRF pages will be reviewed during monitoring visits and transferred to the study database. Upon completion of the study, electronic copies of eCRFs (PDF file) will be stored at the Sponsor's archive and at study sites. Remote monitoring is not foreseen in the study. 100% Source Data Verification (SDV) will be performed at study sites.


### 9. STATISTICAL PLAN

#### 9.1. General consideration

All subjects data collected on the eCRF will be listed by subject, treatment group and center. Appropriate descriptive statistics will be produced, according to the variable. For continuous data, the mean, standard deviation (SD), median, range (minimum and maximum) and 95% confidence interval (CI) will be presented. For categorical data, frequencies and percentages will be presented. If appropriate, 95% CI for proportions will be presented. Unless otherwise specified, the significance level used for statistical testing will be 0.05 and two-sided tests will be used. A Statistical Analysis Plan will be issued describing details of all the statistical methods and analysis to be applied to trial results.

#### 9.2. Sample Size Determination

Sample size calculation was based on the paper of Seymour 1996 [3] concerning a randomized, double-blind, placebo-controlled study of treatment with placebo, paracetamol (500 and 1000 mg) and ketoprofen (12.5 and 25 mg).

The unadjusted AUC<sub>0-6h</sub> values for placebo and ketoprofen were about 263 and 173mmh<sup>-1</sup>, respectively. The corresponding SD were 106 mm h<sup>-1</sup> (about 40% of the mean value for placebo AUC) and 121 mmh<sup>-1</sup> (about 70% of the mean value for ketoprofen 25 mg AUC).

The testing hypothesis for this trial is the superiority of ketroprofen versus placebo that in statistical term is:

 $H_0$ : mean of placebo  $\geq$  mean of ketoprofen (no difference between treatments)

 $H_1$ : mean of placebo < mean of ketoprofen (clinically and statistically significant difference between the groups)  $\Delta$ =90 mm  $h^{-1}$ 

A total of 58 subjects (29 subjects per group) will be necessary to assess a difference of 90 mm h<sup>-1</sup> between the groups with a power of 80%,  $\alpha = 0.05$ , SD=121 mmh<sup>-1</sup>, and randomization rate of 1:1. Sample size calculation was performed using SAS 9.2 [4].

Assuming a drop-out rate of 15%, 70 subjects in total (35 subjects per group) should be enrolled. Considering the screen-failure rate of about 30%, up to 100 patients will be screened in the study.

#### 9.3. Randomization

Subjects will be randomly assigned into one of the two equal groups at 1:1 ratio. Randomization will be conducted with the use of interactive web response system (IWRS). IWRS will assign the study drug kit number that should be dispensed to the patient. Unblinding of the study for the statistical analysis will be performed after the database lock.

Patients' enrollment to the study is competitive between clinical sites.

#### 9.4. Subject Population(s) for Analysis

Disposition of all subjects will be determined prior to database lock and breaking the code.

#### 9.4.1. Intent-to-treat population

The Intent-to-treat (ITT) population will include all randomized patients who receive at least one dose of study medication and have at least one post-baseline efficacy measurement; it will be based on the treatment randomized, regardless of the treatment actually received. The ITT will be used for all efficacy analyses. Subject will be summarized according to the treatment to which they were randomized.


### 9.4.2. Safety population

The Safety population is defined as all randomized subject who received at least one dose of study medication. The Safety population will therefore be identical to the ITT population if all randomized subject receive at least one dose of study medication. The Safety population will be used to present all safety summaries, by actual treatment received.

### 9.4.3. Per-protocol population

ITT population patients comply with the per-protocol population if they complete the study treatment period, have all assessments for the primary efficacy analysis and considered compliant. The patients are compliant if they do not have any major protocol violations in the course of the study. Major protocol violations will be described in details in the Statistical Analysis Plan and identified prior to data-base lock.

### 9.4.4. Handling of missing data

Considering that the primary variable AUC<sub>0-6h</sub> is derived from pain intensity VAS measurements, analyses on primary and secondary variables with substitution of missing data, using the last observation carry forward (LOCF) methodology, has been considered in order to avoid bias in the inferential testing of treatment effect.

The sensitivity analysis will be done using the multiple imputation method for missing data. According to ICH-E9, definition of methods will be refined in the Statistical Analysis plan during the masked data review.

Substitution of missing data will be applied only on all patients that have at least one VAS value post-baseline (patient compliant with ITT population definition). In the SAP will be reported the details concerning the methodology that will be applied.

### 9.5. Demographics and baseline characteristics

Demographics and baseline characteristics will be presented for all subjects in the safety population, by treatment group and summarized using descriptive statistics.

#### 9.6. Efficacy analyses

#### 9.6.1. Analysis of the primary efficacy endpoints

Primary variable will be the  $AUC_{0-6h}$  of pain intensity profile between time 0 (baseline value of VAS) and 6 hours post-treatment.

AUC<sub>0-6h</sub> analysis will be based on actual rather than scheduled timings and will be calculated using the trapezoidal rule. If the actual time is not recorded, the scheduled time will be used instead. LOCF approach will be applied as described in Section 9.4.4.

Treatment AUCs will be compared by means of Student's t-test for independent data. Null hypothesis  $(H_0)$  that  $OKITASK^{\circledR}$  is no different from Placebo will be rejected and alternative hypothesis  $(H_1)$  that  $OKITASK^{\circledR}$  is superior to Placebo will be accepted if mean  $AUC_{0-6h}$   $(OKITASK^{\circledR})$  is less than mean  $AUC_{0-6h}$  (Placebo) and p < 0.05.

### 9.6.2. Analyses of the secondary efficacy endpoints

**Pain profile** – Pain intensity profile will be analyzed using Analysis of Variance (ANOVA) for repeated measurements. The model will include fixed effect terms for clinical site, time point and treatment. Time point will be specified as a repeated measurement. In order to select an appropriate matrix for the observations within each subject, 3 models will be fitted using the compound symmetry, Huynh-Feldt and unstructured structures. The matrix for the final model will be selected using Akaike's Information Criterion where the lowest value indicates the best fit. The importance of the treatment-by-site interaction will be investigated but if the term is not significant at the 10% level, it will be excluded from the final model. The adjusted least squares


means will be estimated for each combination of time point and treatment. The estimated treatment difference between OKITASK® and placebo at each time point will be presented together with the corresponding 95% confidence interval.

**Pain relief** – Pain relief will be analyzed using Analysis of Variance (ANOVA) for repeated measurements. The model will include fixed effect terms for site, time point and treatment. Time point will be specified as a repeated measurement. In order to select an appropriate matrix for the observations within each subject, 3 models will be fitted using the compound symmetry, Huynh-Feldt and unstructured structures. The matrix for the final model will be selected using Akaike's Information Criterion where the lowest value indicates the best fit. The importance of the treatment-by-site interaction will be investigated but if the term is not significant at the 10% level, it will be excluded from the final model. The adjusted least squares means will be estimated for each combination of time point and treatment. The estimated treatment difference between OKITASK® and placebo at each time point will be presented together with the corresponding 95% confidence interval.

Time to first perceptible relief (TFPR) – Kaplan-Meier curve and Log rank test will be used to describe and test treatment profile differences.

**Time to meaningful pain relief (TMPR)** – Kaplan-Meier curve and Log rank test will be used to describe and test treatment profile differences.

**Time to REMD** – Time to rescue medication will be calculated for each subject and presented using only median value. If the number of subjects will be adequate Kaplan-Meier curve and Log rank test will be used to describe and test treatment profile differences.

**Patient's overall assessment** – Cochran-Mantel-Haenzel test will be applied in order to test differences between treatments response.

#### 9.7. Safety analyses

**Oral cavity examination** – Data will be presented with the appropriate descriptive statistics at each time point by treatment group.

**Vital signs** – Vital signs (sitting blood pressure, pulse, and respiratory rate) will be presented with the appropriate descriptive statistics at each time point by treatment group.

Weight and height will be presented with the appropriate descriptive statistics by treatment groups.

#### **Adverse Events**

A summary of treatment-emergent AEs (TEAEs) reported after dosing, including the total number of AEs reported, the number and percentage of subjects reporting at least one AE, the number and percentage of subjects withdrawing prematurely due to an AE, the number and percentage of subjects with at least one SAE and the number and percentage of deaths, will be presented by treatment. In addition, a summary of the event by each category of drug relationship will be presented for AEs and also for SAE.

A breakdown of the number and percentage of subjects reporting each AE, categorized by System Organ Class (SOC) and preferred term (PT) coded according to the MedDRA dictionary (most updated version, available at the end of the study), will be presented. Note that counting will be of subjects not events and subjects are only counted once within each PT.

A further tabulation of these data, broken down by relationship to study drug, will be presented by SOC and PT. Relationship to study drug is categorized as recorded on the eCRF.

A summary of events reported, broken down by severity (mild, moderate, severe), will also be provided by SOC and PT.


A summary of AE leading to early discontinuation will be provided, grouped by SOC and PT.

All adverse events recorded on the eCRF will be listed.

#### **Serious Adverse Events**

A breakdown of the number and percentage of subjects reporting each SAE after dosing, categorized by SOC and PT coded according to the MedDRA dictionary, will be presented.

A further tabulation of these data, broken down by relationship to study drug, will be presented by SOC and PT.

A summary of SAEs reported, broken down by severity (mild, moderate, severe), will also be provided by SOC and PT.

A summary of SAEs leading to early discontinuation will be provided, grouped by SOC and PT.


#### 10. ADMINISTRATIVE PROCEDURES

### 10.1. Legal Aspects

The names of all subjects should be kept in strict confidence. Subject identification is carried out using the assigned number and the birth date. Subjects should be informed that any information held by the study site, the Sponsor or its representatives will be stored in strict confidentiality in accordance with regulatory requirements.

### 10.2. Investigator Responsibilities

The Investigator should conduct the clinical trial in accordance with the protocol, Guidances on Good Clinical Practice of the International Conference on Harmonization (ICH GCP E6 (R2)) and Eurasian Economic Union (EAEU), the principles laid down in the Declaration of Helsinki, and in accordance with applicable laws and regulations.

The Investigator should permit monitoring, auditing and inspections at the study site, and provide the direct access to all study-related materials to the Sponsor or its representatives, Independent Ethics Committee and regulatory authorities at any time.

The Investigator should perform supervision of any individual and/or third party involved in clinical trial and implement procedures to ensure integrity of trial related duties and functions performed and data generated.

The Investigator should keep all signed informed consent forms in original, as well as the complete list of trial participants including full names, addresses and telephone numbers, so that they could be identified later, if necessary. These documents shall not be copied for transmission to the Sponsor or its representatives. The Investigator is obliged to ensure the integrity of study materials, including source documentation, electronic copies of the eCase Report Form (as PDF file) and the Investigator's File for at least 15 years after the study completion or until specified by the Sponsor. The Investigator is obliged to ensure the source data are attributable, legible, contemporaneous, original, accurate and complete.

In any case written authorization by Dompé is necessary before documentation destruction by Investigator/Institution.

### **10.3.** Monitoring procedures

The Principal Investigator should provide the direct access to all source documents, eCRF and Investigator's File to the Sponsor's delegates, as well as IEC and regulatory authorities representatives. The source documentation includes the original documents, data and records (e.g., hospital records, clinical charts, notes, diaries, questionnaires, IP accountability logs, recorded data from automatic devices, verified and certified copies or discharge records, photographic negatives, microfilms or magnetic media, x-rays, and any other records related to the subject and used in the clinical trial).

Monitoring will be conducted by IPHARMA as per delegation in accordance with the IPHARMA SOPs and a study-specific Monitoring Plan. Besides the routine monitoring visits, the sponsor could decide to conduct co-monitoring visits at sites in agreement with IPHARMA.

#### 10.4. eCRFs for data recording

The Investigator should transfer the clinical study data from the source documents to the eCRF in the amount required. The guidelines on eCRF completion are to be learned at the Investigator's meeting and/or the initiation visit. If the Principal Investigator delegates the e-CRF completion to other employees of the study site, their names, positions, initials and signatures must be filled in the Delegation list and provided to the Sponsor or its representative.

All changes made to eCRF must have an audit trail, which means storing the data both with and without corrections, along with the reason for correction, the date and identification of the


person that made corrections. The completed eCRF must be signed by the Principal Investigator electronically.

### 10.5. Record keeping

The source documentation as well as electronic copies of e-CRF and the Investigator's File should be kept at the study site or at a special repository with restricted access for at least 15 years after the study completion or until specified by the Sponsor. The Sponsor shall be informed in case of handing the documents over to another person or institution. In any case written authorization by Dompé is necessary before documentation destruction by Investigator/Institution.

The study-related materials are to be stored by the Sponsor and its representatives in accordance with regulatory requirements.

### 10.6. Ethical aspects

### 10.6.1. Independent Ethics Committee

Prior to the clinical study initiation, all study sites should obtain the written approvals from Independent Ethics Committees (IEC) in accordance with the Guidelines on Good Clinical Practice of the International Conference on Harmonization (ICH GCP E6 (R2)) and Eurasian Economic Union (EAEU), the principles laid down in the Declaration of Helsinki, and in accordance with applicable laws and regulations of the Russian Federation. The following documents are be provided to the IEC: the Protocol with amendments, the patient information leaflet and the informed consent form, written materials to be provided to the patients, the Investigator's Brochure, information on the study drug safety, the information on payments and compensations to be received by the subjects, Investigator CVs and other documents upon request.

The list of IEC members and the statement of compliance with the principles of Good Clinical Practice and regulatory requirements shall be provided to the Sponsor.

### 10.6.2. Ethical considerations

The procedures described in the clinical study Protocol related to its implementation, evaluation and results documentation are designed to ensure that the Sponsor and the Investigator comply with the Guidelines on Good Clinical Practice of the International Conference on Harmonization (ICH GCP E6 (R2)) and Eurasian Economic Union (EAEU). This clinical study will also be conducted in accordance with applicable laws and regulations. This includes the possibility of auditing by the Sponsor representatives and/or regulatory authorities. The Investigator should permit monitoring, auditing and inspections at the study site, and provide the direct access to all study-related materials to the Sponsor or its representatives, Independent Ethics Committee and regulatory authorities at any time.

#### **10.6.3. Informed Consent**

Prior to the clinical study initiation, the Investigator must obtain the written approval of the IEC for the Patient Information Leaflet and the Informed Consent Form and any other written materials to be provided to the patients. The written approval of the IEC and the approved documents should be kept in the Investigator's File.

In obtaining the informed consent, the Investigator should comply with the Guidelines on Good Clinical Practice of the International Conference on Harmonization (ICH GCP E6 (R2)) and Eurasian Economic Union (EAEU), the principles laid down in the Declaration of Helsinki, and in accordance with applicable laws and regulations of the Russian Federation. The informed consent form must be dated and personally signed by the subject prior to the start of any study procedures.


The process of obtaining the informed consent should be described in details in the source documentation, including the subject's consent to participate in this clinical study and the date of signing the informed consent form.

### 10.7. Financing

The study is conducted and fully sponsored by Dompé farmaceutici s.p.a. (Italy). All expenses associated with the study conduct, including state fees, insurance and payments to the study sites, Investigators and third parties involved in the study management, as well as the study drug and other study materials supply, are covered by Dompé farmaceutici s.p.a. as described in the contract between IPHARMA and Dompé farmaceutici s.p.a.

Participation in the study does not require any financial expenses from the patients. All study procedures, including visits to the site, laboratory and instrumental examinations, will be free of charge. Participation in this study does not suggest payments to patients.

The life and health of patients taking part in this clinical study will be insured according to the legislation of the Russian Federation (article 44 of the Federal Law on Drugs Circulation No 61-FZ of April 12, 2010 and other regulatory requirements in force). After signing the informed Consent Form, patients will receive a health insurance certificate for the trial subjects.

### 10.8. Publication Policy

Both the complete and the partial results of the study carried out under this Protocol, and any other information provided by the Sponsor for the purposes of the study conduct, shall not be published or passed on to any third party without the consent of the study Sponsor. Any Investigator involved with this study is obligated to provide the Sponsor with complete test results and all data derived from the study.


### 11. REFERENCES

- 1. Veys EM. 20 Years' Experience with Ketoprofen. Scand J Rheumatol 1991; Suppl. 90: 3-44.
- 2. Singla NK, Desjardins PJ, Chang PD. A comparison of the clinical and experimental characteristics of four acute surgical pain models: dental extraction, bunionectomy, joint replacement, and soft tissue surgery. Pain. 2014 Mar;155(3):441-56
- 3. Seymour R A, Kelly P J, Hawkesford J E. The efficacy of ketoprofen and paracetamol (acetaminophen) in postoperative pain after third molar surgery. Br J Clin Pharmacol 1996; 41: 581–585.
- 4. SAS 9.2 http://support.sas.com/documentation/92/
- 5. MeDRA. https://www.meddra.org/
- 6. Grichnik K P, FERRANTE F M. The Difference between Acute and Chronic Pain The E Mount Sinai Journal of Medicine 1991, 58:3 217-219
- 7. Kantor TG. A Review of Its Pharmacologic and Clinical Properties. Pharmacotherapy 1986; 6(3): 93-103.
- 8. Martindale: the Complete Drug Reference: Ketoprofen. Available at: <a href="http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference">http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference</a> Accessed 13 July 2015.
- 9. KSL0112 (CRO-PK-11-262) Two-way crossover, randomised, single dose bioequivalence phase I study of ketoprofen lysine salt as orodispersible granules (40 mg administered without water) versus ketoprofen lysine salt as granules for oral solution (80 mg bipartite sachet, half sachet) after oral administration to healthy volunteers of both sexes. 30 April 2012.
- 10. Panerai A E, Lanata L, Ferrari M, Bagnasco M. A new ketoprofen lysine salt formulation: 40 mg orodispersible granules Trends in Medicine 2012 October, 12:159-167.
- 11. RBM 930475. Single dose toxicity study in mice treated by oral route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofen Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, July 7, 1994.
- 12. RBM 930473. Single dose toxicity study in rats treated by oral route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofene Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, June 23, 1994.
- 13. RBM 930476. Single dose toxicity study in mice treated by intraperitoneal route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofen Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, July 7, 1994
- 14. RBM 930474. Single dose toxicity study in rats treated by intraperitoneal route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofen Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, June 23, 1994.
- 15. RBM 930477 KLS, S-ketoprofen Lysine salt, R-ketoprofen Lysine salt and ketoprofen. 2-week toxicity studies in rats treated by oral route. RBM, Colleretto Giacosa (TO), Italy, July 21, 1994.
- 16. RBM 910102. 13-week repeated dose toxicity study in Sprague Dawley Crl:CD (SD) BR rats treated with the test article Ketoprofen lysine salt administered by oral route at the doses of 0, 2.5, 7.5 and 15 mg/kg/day followed by a 6-week recovery period. RBM, Colleretto Giacosa (TO), Italy, March 2,1993


- 17. DOM/007/AKL Repeat dose dermal toxicity to rats. A 13-week study. Life Science Research Israel Ltd., Israel, Januray 7, 1991.
- 18. Cimini A, Brandolini L, Gentile R, Cristiano L, et al. Gastroprotective Effects of Lysine Salification of Ketoprefen in Ethanol-Injured Gastric Mucosa. J Cell Physiol. 2015 230: 813-820
- 19. DOM/008/AKL Repeat dose dermal toxicity to rabbits. A l3-week study. Life Science Research Israel Ltd., Israel, Januray 6, 1991.
- RBM 930478 KLS, S-ketoprofen Lysine salt, R-ketoprofen Lysine salt and ketoprofen. Dose Range finding study by oral route in dogs - RBM, Colleretto Giacosa (TO), Italy, July 20, 1994.
- 21. RBM 880004. 13-week repeated dose toxicity study in marmosets treated with the test article Ketoprofen lysine salt administered by oral route at the doses of 0, 2.5, 7.5 and 15 mg/kg/day followed by a 6-week recovery period. RBM, Colleretto Giacosa (TO), Italy, 14 April 1989.
- 22. RBM 880006. Ketoprofen lysine salt. Ames test. RBM, Colleretto Giacosa (TO), Italy, February 29, 1988.
- 23. RBM 890666. Ketoprofen lysine salt. Chromosome aberrations in human lymphocytes. RBM, Colleretto Giacosa (TO), Italy, May 26, 1990.
- 24. RBM 880007. Ketoprofen lysine salt. Gene conversion test in S. cerevisiae D4. RBM, Colleretto Giacosa (TO), Italy, March 30, 1988.
- 25. RBM 920773. Ketoprofen lysine salt. Unscheduled DNA synthesis in cultured HeLa cells. RBM, Colleretto Giacosa (TO), Italy, Febbruary 16, 1993.
- 26. RBM 880008. Ketoprofen lysine salt. Micronucleus test in rat bone marrow. RBM, Colleretto Giacosa (TO), Italy, April 18, 1988
- 27. RBM 880005. Ketoprofen lysine salt. Preliminary teratogenesis study by oral route in rabbits. RBM, Colleretto Giacosa (TO), Italy, December 21, 1989.
- 28. RBM 910272 4-week toxicity study in rabbis by vaginal route. RBM, Colleretto Giacosa (TO), Italy, November 14, 1991.
- 29. Sarzi-Puttini P, Atzeni F, Lanata L et al. Pain and ketoprofen: what is its role in clinical practice? Reumatismo, 2010; 62(3): 172-188.
- 30. Geisslinger G, Menzel S, Wissel K, K. Brune K. Pharmacokinetics of ketoprofen enantiomers after different doses of the racemate. Br J Clin Pharmacol 1995; 40: 73-75
- 31. Bannwarth B, Lapicque F, Netter P, Monot C, Tamisier JN, Thomas P, Royer RJ. The effect of food on the systemic availability of ketoprofen. Eur J Clin Pharmacol. 1988;33(6):643-5.
- 32. Martindale: the Complete Drug Reference: Ketoprofen. Available at: <a href="http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference">http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference</a> Accessed 13 July 2015.
- 33. Netter P, Lapicque F, Bannwarth B, Tamisier JN, et al. Diffusion of Intramuscular Ketoprofen Into the Cerebrospinal Fluid. Eur J Clin Pharmacol. 1985; 29:319-21.
- 34. Advenier C, Roux A, Gobert C et al. Pharmacokinetics of ketoprofen in the elderly. Br J Clin Pharmacol 1983; 16: 65-70.


- 35. Skeith KJ, Dasgupta M, Lange R, Jamali F. The influence of renal function on the pharmacokinetics of unchanged and acyl-glucuroconjugated ketoprofen enantiomers after 50 and 100 mg racemic ketoprofen. Br J Clin Pharmacol 1996; 42: 163–169.
- 36. Stafanger G, Larsen HW, Hansen H, Sorensen K. Pharmacokinetics of ketoprofen in patients with chronic renal failure. Scand J Rheumatology 1981; 10: 189-192.
- 37. Vallés J, Artigas J R, Bertolotti M, Crea3 A, Müller F, Paredes I, Capriati A Single and Repeated Dose Pharmacokinetics of Dexketoprofen Trometamol in Young and Elderly Subjects. Methods Find Exp Clin Pharmacol 2006, 28(Suppl. A): 13-19.
- 38. Upton, RA, Buskin, JN, Williams, RL, Holford, NHG, Riegelman, S. Negligible excretion of unchanged ketoprofen, naproxen and probenecid in urine, J Pharm Sci 1980 69: 1254-1257.
- 39. Dawood, M.Y. Nonsteroidal antiinflammatory drugs and reproduction. Am. J. Obstet. Gynecol., 1993, 169, 1255-1265.
- 40. Van der Weiden, R.M.; Helmerhorst, F.M.; Keirse, M.J. Influence of prostaglandins and platelet activating factor on implantation. Hum. Reprod., 1991, 6, 436-442
- 41. Van der Weiden, R.M.; Helmerhorst, F.M.; Keirse, M.J. Prostanoid excretion in incipient singleton and twin pregnancies. Am. J. Obstet. Gynecol., 1996, 174, 1614-1617.
- 42. Van der Weiden, R.M.; Wouters, J.M. Infertility may sometimes be associated with nonsteroidal anti-inflammatory drug consumption. Br. J. Rheumatol., 1997, 36, 605.
- 43. Siu, S.S.; Yeung, J.H.; Lau, T.K. An in-vivo study on placental transfer of naproxen in early human pregnancy. Hum. Reprod., 2002, 17, 1056-1059.
- 44. Antonucci R, Zaffanello M, Puxeddu E, Porcella A et al. Use of Non-steroidal Antiinflammatory Drugs in Pregnancy: Impact on the Fetus and Newborn. Curr Drug Metab. 2012; 13(4):474-90.
- 45. Ofori, B.; Oraichi, D.; Blais, L.; Rey, E.; Bérard, A. Risk of congenital anomalies in pregnant users of non-steroidal anti-inflammatory drugs: A nested case-control study. Birth Defects Res. B. Dev. Reprod. Toxicol., 2006, 77(4), 268-279.
- 46. Ericson A, Källén BA. Nonsteroidal anti-inflammatory drugs in early pregnancy. Reprod. Toxicol. 2001 Jul-Aug; 15(4):371-5 2001.
- 47. Dollery C, ed. Therapeutic Drugs. Second Edition. Churchill Livingstone. Edinburgh 1999.
- 48. Becker J C, Domschke W, Pohle T. Current approaches to prevent NSAID-induced gastropathy COX selectivity and beyond Br J Clin Pharmacol 58:6 587–600 587.
- 49. PhVWP EMEA/12148/04/Final: Wording of the Summaries of Products Characteristics of Acetylsalicylic acid and Non-Steroidal Anti-inflammatory Drugs with regard to Use during Pregnancy and Risk of Miscarriage and Congenital Malformations
- 50. INVESTIGATOR'S BROCHURE -Ketoprofen L-lysine Salt 40 mg granules Version No. 3 FINAL 29 August 2017


### 12. APPENDIX

### 12.1. Visual analogue scale "Pain intensity"

Please put a mark on the below scale based on the current intensity of your pain symptoms.

| No pain | Worst pain |
|---|---|
| | imaginable |
| 12.2. Visual analogue scale "Pain relief" | |
| ease put a mark on the below scale based on the curre | ent relief of your pain symptoms. |
| No relief | Maximum re |

**NB:** Please use only VAS provided by IPHARMA and avoid to perform any copy of the form.

In case you need to perform a reproduction of the form (for any reason) before using it you must verify the length of the VAS: the line must be 100 mm.

### 12.3. Patient's overall assessment (5-point scale)

Considering all the ways that the pain affects you, how well are you doing?

| 1 = very good | 2 = good | 3= satisfactory | 4 = poor | 5 = very poor |
|---------------|----------|-----------------|----------|---------------|


### ПРОТОКОЛ КЛИНИЧЕСКОГО ИССЛЕДОВАНИЯ

#### KSL0117

**Наименование** Многоцентровое, двойное-слепое, рандомизированное исследования: исследование в параллельных группах оценки

эффективности и переносимости однократного приема гранул кетопрофена лизиновой соли 40 мг в сравнении с Плацебо у мужчин и женщин с острым болевым синдромом

после удаления моляров

**Номер исследования:** KSL0117

Фаза разработки: III

Исследуемый

ОКІТАЅК<sup>®</sup> гранулы по 40 мг для перорального приема

препарат:

Исследуемое Острый болевой синдром после удаления моляров

показание к применению:

**Спонсор:** Dompé farmaceutici s.p.a.

Контактное лицо и

адрес:

Mauro P. Ferrari

Via Santa Lucia, 6 20122 Milano, Italy

Телефон +39 02 58383271

1

версия и дата: января 2018 года)

Финальная Версия 1.0 – 26 сентября 2017 (в редакции от 25

В спучае несоответс

В случае несоответствия между Русской и Английской версиями, Английская версия протокола является основной.

Основная версия

Оригинальная

### Заявление о конфиденциальности

Настоящий документ является конфиденциальной информацией, принадлежащей компании «Dompé farmaceutici s.p.a». Запрещается прямая или непрямая публикация, передача или иное раскрытие содержимого этого документа, равно как и передача любой части этого документа третьим лицам. Разрешается использовать данный документ только в тех целях, для которых он был предоставлен. Информацию из него можно раскрывать только после получения письменного разрешения от компании «Dompé farmaceutici s.p.a», или представителям соответствующих регуляторных органов, или по судебному решению. О любом случае раскрытия информации из этого документа, как разрешенном, так и не разрешенном, необходимо незамедлительно сообщить в компанию «Dompé farmaceutici s.p.a».

# СТРАНИЦА ОДОБРЕНИЯ ПРОТОКОЛА

| CHOHCOP: Dompé farmaceutici s.p.a». | Дата: |
|---------------------------------------------------------|-------|
| Подпись: | |
| Имя и должность: Marcello Allegretti, ChemD | |
| Директор по науке | |
| Подпись: | Дата: |
| Имя и должность: Mauro P. Ferrari, PharmD | |
| Менеджер разработки клинических исследований ранних фаз | |
| Подпись: | Дата: |
| Имя и должность: Luigi Lanata, MD | |
| Медицинский директор | |
| КИО: OOO «ИФАРМА» | |
| Подпись | Дата |
| Имя и должность: Наталья Востокова, PharmD. | |
| Исполнительный директор, ООО ИФАРМА | |
| Подпись | Дата |
| Имя и должность: Юлия Трахтенберг, к.м.н. | |
| Медицинский директор, ООО ИФАРМА | |

КОНФИДЕНЦИАЛЬНО Страница 2 из 76

Dompé farmaceutici s.p.a. 26 сентября 2017 года (в редакции от 25 января 2018 года)

### ЗАЯВЛЕНИЕ ГЛАВНОГО ИССЛЕДОВАТЕЛЯ

### полное имя:

Я, нижеподписавшийся, подтверждаю, что я прочел этот протокол исследования и понял его. Я согласен следовать требованиям протокола исследования "Многоцентровое, двойное-слепое, рандомизированное исследование в параллельных группах оценки эффективности и переносимости однократного приема гранул кетопрофена лизиновой соли 40 мг в сравнении с Плацебо у мужчин и женщин с острым болевым синдромом после удаления моляров".

Я буду проводить это исследование в соответствии с требованиями стандарта Надлежащей клинической практики Международной конференции по гармонизации (Good Clinical Practice Guidelines of International Conference on Harmonization, ICH GCP) и Евразийского Экономического Союза (EAЭС), а также с принципами, указанными в Хельсинкской декларации и действующими законами Российской федерации.

| Хельсинкской декларации и действующими законами Российской федерации. | |
|---|---|
| Дата: | Подпись: |

# КОНТАКТНЫЕ ДАННЫЕ

| СПОНСОР<br>ИССЛЕДОВАНИЯ | Компания "Dompe farmaceutici s.p.a."<br>Via Santa Lucia, 20122 Milano, Italy |
|---|---|
| Mauro P. Ferrari | Менеджер разработки клинических исследований ранних фаз |
| | Телефон +39 02 58383271 |
| | Электронная почта: mauro.ferrari@dompe.com |
| Luigi Lanata | Медицинский директор |
| | Телефон +39 02 58383473 |
| | Электронная почта: <a href="mailto:luigi.lanata@dompe.com">luigi.lanata@dompe.com</a> |
| Laura Boga | Старший менеджер по безопасности – безопасность препарата |
| | Телефон +39 02 58383568 |
| | Факс +39 02 36026913 |
| | Электронная почта: laura.boga@dompe.com |
| | Адрес электронной почты для отчетов по СНЯ: <a href="mailto:farmacovigilanza@dompe.com">farmacovigilanza@dompe.com</a> |
| Подача отчетов по СНЯ/ | Dompé Drug Safety |
| случаям беременности | Факс +39 02 36026913 |
| | Электронная почта: farmacovigilanza@dompe.com |
| КОНТРАКТНАЯ | ООО ИФАРМА |
| ИССЛЕДОВАТЕЛЬСКАЯ | 143026, Россия, г. Москва |
| ОРГАНИЗАЦИЯ<br>(МОНИТОРИНГ, | Инновационный центр "Сколково" |
| медицинский | Улица Нобеля, дом 7 |
| мониторинг) | |
| Наталья Востокова | Исполнительный Директор |
| | Телефон: +7 (495) 276-11-43 |
| | Факс: +7 (495) 276-11-47 |
| | Электронная почта: nv@ipharma.ru |
| Юлия Трахтенберг | Медицинский директор |
| | Телефон: +7 (495) 276-11-43 |
| | Факс: +7 (495) 276-11-47 |
| | Электронная почта: jat@ipharma.ru |
| Виктория Яворская | Медицинский советник |
| | Телефон: +7 (495) 276-11-43 |
| <u> </u> | I |

| | Факс: +7 (495) 276-11-47 |
|---|---|
| | Электронная почта: yvv@ipharma.ru |
| Валерий Поддубный | Менеджер проекта |
| | Телефон: +7 (495) 276-11-43 |
| | Факс: +7 (495) 276-11-47 |
| | Электронная почта: vap@ipharma.ru |
| Регистрация СНЯ/ случаев | Медицинский отдел компании "ИФАРМА" |
| беременности (24 часа в сутки) | Факс: +7 (495) 276-11-47 |
| Cythny | Электронная почта: SAE@ipharma.ru |
| ОБРАБОТКА ДАННЫХ, | ООО "КейСтат" |
| БИОСТАТИСТИКА | 214000, Россия, г. Смоленск |
| П | ул 2-я линия Красноармейской слободы, д. 3 |
| Дмитрий Хамцов | Биостатистика и общее управление<br>Телефон: +7 (915) 644-47-13 |
| | Электронная почта: |
| | dmitry.khamtsov@keystatsolutions.com |
| ЦЕНТРАЛЬНАЯ | Не применимо |
| ЛАБОРАТОРИЯ | |
| ЛОКАЛЬНЫЙ СКЛАД | VORTEX CLINICAL SERVICES |
| STOKASIBITBINI CKSIAZI | 143405, Россия, Московская область, |
| | Красногорский район, деревня Гольево, |
| | Центральная ул., д. 3 |
| D | <u> </u> |
| Владимир Нестерин | Руководитель отдела контроля качества |
| | Телефон: + 7 (495) 785-65-78 |
| | Телефон: + 7 (495) 783-76-53 |
| | Электронная почта: Vladimir.Nesterin@vortexcs.com |
| КЛИНИЧЕСКИЕ | В соответствии с утвержденным списком клинических |
| ЦЕНТРЫ | центров |

#### СИНОПСИС

Спонсор исследования: компания "Dompé farmaceutici s.p.a.", Италия

**Исследуемый препарат:** ОКИТАСК<sup>®</sup> гранулы по 40 мг

Действующее вещество: кетопрофена лизиновая соль 40 мг

**Наименование исследования:** Многоцентровое, двойное-слепое, рандомизированное исследование в параллельных группах оценки эффективности и переносимости однократного приема гранул кетопрофена лизиновой соли 40 мг в сравнении с Плацебо у мужчин и женщин с острым болевым синдромом после удаления моляров.

**Номер исследования:** KSL0117

Фаза разработки: III

#### Основная цель:

Основной целью данного исследования является оценка эффективности препарата ОКИТАСК® в гранулах по 40 мг в сравнении с плацебо у пациентов с острым болевым синдромом после удаления одного моляра, проводимая путем сравнения AUC0-6ч профиля боли после терапии, измеряемой с помощью визуально-аналоговой шкалы.

### Дополнительные цели:

Оценка следующих параметров эффективности и безопасности препарата  $OKUTACK^{®}$  в гранулах по 40 мг в сравнении с плацебо у пациентов с острой болью после удаления одного моляра:

- Профиль боли в зависимости от времени и профиль снижения интенсивности боли с течением времени по результатам заполнения визуально-аналоговой шкалы
- Время до первого ощутимого снижения интенсивности боли (ВПСБ) и время до значительного снижения интенсивности боли (ВЗСБ)
- Доля пациентов, которым требуется терапия спасения (обезболивание) и время до приема терапии спасения
- Общая оценка, проведенная самими пациентами
- Частота нежелательных явлений (НЯ)

### Общая информация:

Компания "Dompé farmaceutici s.p.a." планирует зарегистрировать в России препарат  $OKUTACK^{\otimes}$  в гранулах по 40 мг, который является новой лекарственной формой лизиновой соли кетопрофена.

Кетопрофен является высокоактивным нестероидным противовоспалительным препаратом, относящимся к группе производных пропионовой кислоты. Кетопрофен применяется в стандартной клинической практике с 1973 года, в настоящее время является одним из наиболее широко применяемых нестероидных противовоспалительных препаратов и считается эффективным противовоспалительным средством с хорошей переносимостью. Получение аминокислотных солей кетопрофена значительно повысило его растворимость в воде, что позволило разработать жидкие лекарственные формы кетопрофена для перорального приема и позволило получить три основных клинических преимущества: 1) более быстрое всасывание из желудочно-кишечного тракта (ЖКТ) по сравнению с исходным веществом; 2) более быстрое

Dompé farmaceutici s.p.a. 26 сентября 2017 года (в редакции от 25 января 2018 года)

противовоспалительное и обезболивающее действие; 3) более кратковременное пребывание активного вещества в желудке и, следовательно, более низкий потенциал раздражающего действия и/или эффектов, приводящих к возникновению язв [11].

Лизиновая соль кетопрофена в форме гранул для приготовления раствора для перорального приема (ОКі® в пакетиках по 80 мг, содержащих 80 мг лизиновой соли кетопрофена в сдвоенном пакетике, по 40 мг лизиновой соли кетопрофена в каждой из частей) уже зарегистрирована и продается компанией Dompé в Италии с 1994 года, а в России с 1998 года в качестве средства для кратковременного лечения симптомов воспалительных состояний, сопровождающихся болью.

В ходе настоящего исследования планируется провести оценку эффективности и безопасности препарата ОКИТАСК® в гранулах по 40 мг в сравнении с плацебо у пациентов с острым болевым синдромом после удаления одного моляра.

### Дизайн исследования:

Данное исследование является многоцентровым, двойным слепым, рандомизированным плацебо-контролируемым исследованием в параллельных группах пациентов, которое проводится с целью оценки эффективности и безопасности препарата ОКИТАСК® в гранулах по 40 мг у пациентов с острым болевым синдромом после удаления моляра. Это исследование будет проводиться в 4-6 исследовательских центрах в России. Ожидается, что в него будет включено в совокупности 70 пациентов (по 35 в каждой группе). Набор пациентов в центрах является конкурентным.

Исследование будет состоять из трех периодов: период скрининга, период исследуемой терапии и период наблюдения.

В периоде скрининга после подписания информированного согласия у пациента будут в рамках определения критериев включения/невключения собраны демографические данные, медицинский анамнез и данные по сопутствующей лекарственной терапии, выполнен осмотр ротовой полости, проведены взвешивание и оценка показателей жизненных показателей, а кроме того, пациентам женского пола будет выполнен тест на беременность. Процедуры скрининга могут занять до 4 дней перед плановым удалением зуба, включая сам день, в который будет удален зуб.

В День 1 пациенту будет выполнено удаление моляра в соответствии с показаниями, обусловленными состоянием зубов. Удаление зуба будет проведено с применением стандартной методики и методов обезболивания (рекомендованные типы анестезии представлены в Разделе 5.9 "Сопутствующая терапия и терапия спасения" данного протокола исследования). После этого пациент останется в исследовательском центре для лечения болевого синдрома в соответствии с протоколом исследования.

Оценка интенсивности боли будет проводиться с применением визуальноаналоговой шкалы (ВАШ) в течение 3 часов после процедуры удаления зуба. Кроме того, будет регистрироваться оценка, которую будет проводить сам пациент. Если интенсивность боли по визуально-аналоговой шкале будет выше 30 мм и потребуется обезболивание, то пациент будет рандомизирован в это исследование.

При рандомизации пациенты распределяются в соотношении 1:1 в одну из двух групп:

Группа 1. Терапия препаратом ОКИТАСК $^{\text{®}}$  в дозе 40 мг – 35 пациентов

Группа 2. Терапия плацебо – 35 пациентов.

До получения исследуемого препарата (момент времени 0') пациент проведет оценку боли по визуально-аналоговой шкале.

Сразу же при приеме исследуемого препарата пациенты должны запустить два секундомера. Один из них должен быть остановлен сразу же, как только пациент почувствует заметное снижение боли, а второй — после того как пациент почувствует значительное снижение боли.

Пациент будет оставаться в исследовательском центре в течение 6 часов после приема исследуемого препарата для оценки боли и нежелательных явлений. Интенсивность боли будет оцениваться по визуально-аналоговой шкале через 5 минут, 10 минут, 15 минут, 30 минут, 45 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) минут после приема препарата.

Оценка снижения интенсивности боли будет проводиться по визуально-аналоговой шкале через 5 минут, 10 минут, 15 минут, 30 минут, 45 минут, 60 минут (1 час), 90

минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) минут после приема препарата.

Пациенты должны указывать действительное время проведения оценки по визуально-аналоговой шкале. Отклонения от запланированных временных точек не будут считаться отклонениями от протокола исследования. Отклонением от протокола исследования будет считаться только пропуск оценок.

Непосредственно перед тем, как пациент покинет исследовательский центр, ему предложат провести оценку своего состояния по шкале Общей оценки, проведенной самими пациентами.

В День 3 (через 48 часов после применения исследуемого препарата) будет проведен телефонный разговор с пациентом для оценки нежелательных явлений. Любые серьезные нежелательные явления, о которых пациент спонтанно сообщит в течение 30 дней после приема исследуемого препарата, должны быть зарегистрированы.

Если пациенту потребуется применение дополнительной лекарственной терапии в любое время в течение 6 часов после приема исследуемого препарата, то последняя оценка боли по визуально-аналоговой шкале и общая оценка лечения пациентом своего состояния по шкале Общей оценки, проведенной самими пациентами, должны быть выполнены перед получением препаратов терапии спасения (Раздел 7.3).

### Популяция пациентов:

Взрослые пациенты мужского и женского пола, которым запланировано удаление моляра.

#### Критерии включения и невключения:

### Критерии включения в исследование:

- 1. Подписанная форма информированного согласия;
- 2. Мужчины и женщины в возрасте от 18 до 65 лет (включительно);
- 3. Лица, которым было выполнено удаление не ретинированного моляра в течение 3 часов до рандомизации;
- 4. Лица с хорошим состоянием здоровья (понятие базируется на основе критериев безопасного применения амбулаторного обезболивания);
- 5. Лица, которым в течение 3 часов после экстракции зуба требуется прием препарата для уменьшения боли (ВАШ ≥ 30 мм);
- 6. Лица, которые согласны оставаться под наблюдением в течение до 9 часов после удаления зуба;
- 7. Лица, способные заполнить 100-миллиметровую визуально-аналоговую шкалу и категориальную шкалу в течение периода наблюдения (около 9 часов);
- 8. Полное понимание: способность понимать суть и цели исследования, включая возможные риски и побочные эффекты; способность сотрудничать с Исследователем и выполнять все требования исследования;
- 9. Контрацепция (для женщин): женщины, способные к деторождению, должны использовать как минимум один надежный метод контрацепции из числа перечисленных ниже:
  - а. гормональные пероральные, имплантируемые, трансдермальные или
#### инъекционные контрацептивы;

b. негормональное внутриматочное устройство (ВМУ), или женский презерватив со спермицидом, или контрацептивная губка со спермицидом, или диафрагма со спермицидом, или шеечный колпачок со спермицидом;

или:

- с. мужчина половой партнер женщины должен быть согласен на использование мужского презерватива со спермицидом;
- d. половой партнер, которому была выполнена стерилизация.

#### Критерии невключения:

- 1. Лица, которым были выполнены: удаление ретинированного и дистопированного зуба, зубосохраняющие операции, апикальное перемещение лоскута/ вестибулопластика со свободным трансплантатом десны, взятым из твердого неба;
- 2. Лица, которым в течение одной процедуры было удалено больше одного зуба;
- 3. Лица, которым одновременно с удалением зуба была выполнена установка импланта;
- 4. Аллергия: известная или предполагаемая гиперчувствительность к активным компонентам (кетопрофен и парацетамол, применяемый в качестве терапии спасения) и/или вспомогательным веществам в составе препарата; наличие в анамнезе гиперчувствительности к лекарственным препаратам (в особенности, к нестероидным противовоспалительным препаратом) или аллергических реакций в целом, которые, по мнению Исследователя, могут повлиять на результаты исследования;
- 5. Заболевания: наличие в анамнезе значимых заболеваний почек, печени, сердечно-сосудистой системы, дыхательной системы (в том числе бронхиальной астмы), кожи, системы крови, органов внутренней секреции, желудочно-кишечного тракта и мочевыводящих путей и половой системы, либо нервной системы или аутоиммунных заболеваний, которые могут повлиять на цели исследования;
- 6. Лекарственные препараты: прием нестероидных противовоспалительных препаратов и других обезболивающих препаратов (в особенности, кетопрофена, парацетамола и ацетилсалициловой кислоты (АСК)), антигистаминных препаратов, седативных препаратов, в том числе растительных препаратов и биологически активных пищевых добавок в течение 48 часов до удаления зуба;
- 7. Исследования других лекарственных препаратов: участие в исследовании любого другого препарата в течение 3 месяцев до начала скрининга (включая последнюю процедуру исследования);
- 8. Алкогольная и наркотическая зависимость в анамнезе;
- 9. Положительные результаты теста на беременность у женщин, способных к деторождению (включая женщин, находящихся в постменопаузе менее 2 лет).

# Дозировка исследуемого препарата и способ его применения:

Действующее вещество: Кетопрофена лизиновая соль (КЛС)

Клинико-фармацевтический класс: противовоспалительные и противоревматические препараты, нестероидные (код ATX: M01AE03).

Лекарственная форма: гранулы кетопрофена лизиновой соли по 40 мг (соответствует 25 мг кетопрофена)

Применение препарата: 1 пакетик – 40 мг – однократно

Условия хранения: хранить при температуре не выше + 25°C

Производитель: компания "Dompé farmaceutici s.p.a." (Италия)

Повторная упаковка (первичная и вторичная): компания "Monteresearch" (Италия)

Контроль и выпуск партии: компания "Dompé farmaceutici" (Италия)

# Контрольная группа: плацебо

Лекарственная форма: гранулы по 0 мг кетопрофена лизиновой соли

Применение препарата: 1 пакетик – однократно

Условия хранения: хранить при температуре не выше + 25°C

Производитель: компания "Monteresearch" (Италия)

Контроль и выпуск партии: компания "Dompé farmaceutici" (Италия)

## Конечные точки оценки эффективности:

#### Первичная конечная точка оценки эффективности:

- AUC<sub>0-6ч</sub> профиля боли от момента 0 (исходное значение на ВАШ) и до 6 часов после начала терапии

Оценка боли будет проводиться по горизонтальной 100-миллиметровой визуальноаналоговой шкале (ВАШ): от 0 (отсутствие боли) до 100 (самая сильная боль, которую только можно представить) в 0 минут (непосредственно перед приемом исследуемого препарата показатель по ВАШ долен быть >30 мм), а также через 5 минут, 10 минут, 15 минут, 30 минут, 45 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) минут после приема препарата.

Пациенты должны указывать действительное время проведения оценки по визуально-аналоговой шкале. Отклонения от запланированных моментов времени не будут считаться отклонениями от протокола исследования. Отклонениями от протокола исследования будет считаться только пропуск оценок.

Расчет  $AUC_{0-64}$  будет проводиться по правилу трапеций. Если пациенту потребуется терапия спасения в любое время в течение 6 часов после приема исследуемого препарата, то будет использоваться последняя оценка по визуально-аналоговой шкале, полученная перед этим. Для расчета  $AUC_{0-64}$  будут использоваться данные последнего наблюдения (перенос вперед данных последнего наблюдения).

## Вторичные конечные точки оценки эффективности:

- Профиль боли в зависимости от времени и профиль снижения интенсивности боли с течением времени

Оценка боли будет проводиться по горизонтальной 100-миллиметровой визуально-

аналоговой шкале (ВАШ): от 0 (отсутствие боли) до 100 (самая сильная боль, которую только можно представить) в 0 минут (непосредственно перед приемом исследуемого препарата показатель по ВАШ должен быть >30 мм), а также через 5 минут, 10 минут, 15 минут, 30 минут, 45 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) минут после приема препарата.

Пациенты должны указывать действительное время проведения оценки по визуально-аналоговой шкале. Отклонения от запланированных моментов времени не будут считаться отклонениями от протокола исследования. Отклонениями от протокола исследования будет считаться только пропуск оценок.

Оценка снижения интенсивности боли будет проводиться по горизонтальной 100-миллиметровой визуально-аналоговой шкале: от 0 (интенсивность боли не снизилась) до 100 (максимальное снижение боли) через 5 минут, 10 минут, 15 минут, 30 минут, 45 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) минут после приема препарата.

Если пациенту потребуется терапия спасения в любое время в течение 6 часов после приема исследуемого препарата, то будет использоваться последняя оценка по визуально-аналоговой шкале, полученная перед этим. Все остальные оценки эффективности (если такие останутся) будут исключены из анализа.

# - Время до первого ощутимого снижения интенсивности боли (ВПСБ) и время до значительного снижения интенсивности боли (ВЗСБ)

Измерение времени до первого ощутимого снижения интенсивности боли (ВПСБ) и времени до значительного снижения интенсивности боли (ВЗСБ) будет проводиться с помощью секундомеров. Сразу же при приеме исследуемого препарата пациенты должны запустить два секундомера. Один из них должен быть остановлен сразу же, как только пациент почувствует заметное снижение боли, а второй – после того как пациент почувствует значительное снижение боли.

# - Доля пациентов, которым требуется терапия спасения (обезболивание) и время до проведения терапии спасения

В случае недостаточного контроля боли пациент получит лекарственную терапию спасения для обезболивания (т.е., парацетамол в таблетках в дозе 500-1000 мг). Время до приема обезболивающего препарата терапии спасения, если такое произойдет, также будет регистрироваться (NB: участникам будет предложено воздерживаться от приема резервных препаратов в течение первого часа после приема исследуемого препарата). Если парацетамол в дозе 500 или 1000 мг не окажет нужного эффекта, пациенту будет разрешено принять еще одну дозу парацетамола 500 мг или 1000 мг. Интервал между приемами должен быть не менее 4 часов. максимальная суточная доза составляет 4000 мг.

# Общая оценка, проведенная самими пациентами

Общая оценка, проведенная самими пациентами (5-балльная шкала): 1 = очень хорошо, 2 = хорошо, 3 = удовлетворительно, 4 = плохо, 5 = очень плохо.

Эта оценка будет проводиться после исходного заполнения визуально-аналоговой шкалы и непосредственно перед тем как пациент покинет исследовательский центр. Если пациент получает терапию спасения, то он должен провести общую оценку после последнего заполнения визуально-аналоговой шкалы.

#### Конечные точки оценки безопасности:

## - Частота нежелательных явлений (НЯ)

Регистрация нежелательных явлений будет проводиться в соответствии с жалобами участника исследования, данными обследования ротовой полости и оценки показателей функций жизненно-важных органов.

#### Методы статистической обработки:

Все данные по пациентам, собранные в электронных индивидуальных регистрационных картах (эИРК), будут сведены по пациентам, группам терапии и исследовательским центрам. В соответствии с показателями будут применены подходящие методы описательной статистики. Для непрерывных данных будут представлены средние показатели, стандартное отклонение (СО), медиана, диапазон (минимум и максимум) и 95% доверительный интервал (ДИ). Для категорийных данных будут представлены частота и проценты. Если это применимо, то для пропорций будут представлены 95% доверительные интервалы. Если не указано иное, то уровнем значимости, используемым для статистического тестирования, будет 0,05, а используемые тесты будут двухсторонними. Будет выпущен план статистического анализа, в котором будут подробно описаны все статистические методы и анализы, которые будут применяться к результатам исследования.

## Анализ первичной конечной точки оценки эффективности:

Первичной переменной будет  $AUC_{0-64}$  профиля боли от момента 0 (исходное значение на визуально-аналоговой шкале) до 6 часов после начала терапии.

Анализ  $AUC_{0-64}$  будет основан на фактических, а не на запланированных моментах времени, а расчет будет проводиться по правилу трапеций. Если фактическое время не записано, то будет использовано запланированное время.

Будет проведено сравнение показателей AUC при терапии со средними данными t-теста Стьюдента для независимых данных. Если средняя  $AUC_{0-64}$  при применении препарата OKИTACK® будет меньше средней  $AUC_{0-64}$  при применении плацебо при p<0,05, то нуль-гипотеза (H<sub>0</sub>), утверждающая, что препарат OKИTACK® не отличается от плацебо, будет отклонена и вместо нее будет принята альтернативная гипотеза (H<sub>1</sub>), утверждающая, что препарат OKИTACK® превосходит плацебо.

# Анализ конечных точек безопасности:

Все нежелательные явления, зарегистрированные в электронной ИРК, будут кодироваться по классам систем и органов (System Organ Class, SOC) и предпочтительным терминам (ПТ) на основе Медицинского словаря для нормативноправовой деятельности в сфере лекарственных препаратов (Medical Dictionary for Drug Regulatory Affairs, MedDRA [5]). Они будут валидированы и просуммированы в зависимости от терапии, взаимосвязи с исследуемой терапией и степенью тяжести.

#### Размер выборки:

Расчет размера выборки исследования был основан на статье Seymour 1996 [3], в которой идет речь о рандомизированном, двойном слепом, плацебо-контролируемом исследовании с терапией плацебо, парацетамолом (500 и 1000 мг) и кетопрофеном (12,5 и 25 мг).

Неоткорректированные показатели AUC0-6ч для плацебо и кетопрофена составили приблизительно 263 и 173 мм ч-1 соответственно. Соответствующие показатели стандартного отклонения составили 106 мм ч-1 (приблизительно 40% от среднего значения для AUC при применении плацебо) и 121 мм ч-1 (приблизительно 70% от среднего значения для AUC при применении кетопрофена в дозе 25 мг).

Тестируемой гипотезой для этого исследования является превосходство кетопрофена в сравнении с плацебо, что в статистических терминах будет выглядеть следующим образом:

H0: среднее при применении плацебо ≥ среднего при применении кетопрофена (без различий между разными видами терапии)

H1: среднее при применении плацебо < среднего при применении кетопрофена (клинически и статистически значимое различие между группами)

Всего для достижения разницы в 90 мм ч-1 между группами при мощности 80%, а = 0,05, CO = 121 мм ч-1 и при соотношении рандомизации 1:1 потребуется 58 пациентов (по 29 пациентов в группе). Расчет размера популяции был проведен с помощью программы SAS 9.2 [4].

С учетом уровня досрочного выбытия из исследования, который составляет 15%, включение в исследование должено составить 70 пациентов (по 35 пациентов в каждой из групп). С учетом того, что доля пациентов, не прошедших скрининг, составит приблизительно 30%, планируется, что в ходе этого исследования будет скринировано до 100 пациентов.

# Рандомизация:

Участники исследования будут в случайном порядке распределены в одну из двух равных по размеру групп в соотношении 1:1. Рандомизация будет проводиться с применением системы интерактивного взаимодействия через сеть Интернет (interactive web response system, IWRS).

#### Версия протокола и дата выпуска:

KSL0117 Финальная версия 1.0 от 26 сентября 2017 года (в редакции от 25 января 2018 года).

# ОГЛАВЛЕНИЕ

| ЗАЯВЛЕНИЕ ГЛАВНОГО ИССЛЕДОВАТЕЛЯ | 3 |
|-----------------------------------------------------------|----|
| КОНТАКТНЫЕ ДАННЫЕ | 4 |
| СПИСОК СОКРАЩЕНИЙ | 18 |
| 1. ВВЕДЕНИЕ | 21 |
| 2. ЦЕЛИ ИССЛЕДОВАНИЯ | 24 |
| 2.1. Основная цель | 24 |
| 2.2. Дополнительные цели | 24 |
| 3. ДИЗАЙН ИССЛЕДОВАНИЯ | 24 |
| 3.1. Общий дизайн и план исследования | 24 |
| 3.1.1. Дизайн исследования | 24 |
| 3.2. Обоснование дизайна исследования | 29 |
| 3.3. Длительность исследования | 30 |
| 3.4. Ранее полученный опыт применения препарата ОКИТАСК® | 30 |
| 3.4.1. Доклинические данные | 32 |
| 3.4.2. Клинические данные | 34 |
| 3.5. Обоснование выбора дозы и соотношение риска и пользы | 44 |
| 4. ИССЛЕДУЕМАЯ ПОПУЛЯЦИЯ | 44 |
| 4.1. Исследуемая популяция | 45 |
| 4.2. Критерии включения | 45 |
| 4.3. Критерии невключения | 45 |
| 4.4. Критерии невключения | 46 |
| 5. ИССЛЕДУЕМЫЙ ПРЕПАРАТ | 47 |
| 5.1. Описание | 47 |
| 5.2. Режим терапии | 48 |
| 5.3. Рандомизация и закрытие кодов терапии | 48 |
| 5.4. Процедура раскрытия кодов терапии | 48 |
| 5.5. Комплаентность в отношении исследуемой терапии | 48 |
| 5.6. Упаковка и маркировка препарата | 48 |
| 5.7. Учет исследуемого препарата | 49 |
| 5.8. Хранение исследуемого препарата | 49 |
| 5.9. Сопутствующая и резервная терапия | 49 |
| 5.10. Запрещенная предшествующая и сопутствующая терапия | 50 |
| 6. ПРОЦЕДУРЫ ИССЛЕДОВАНИЯ | 51 |
| 6.1. Информированное согласие | 51 |
| 6.2. Регистрация пациента | 51 |
| 6.3. Демографические данные и медицинский анамнез | 51 |
| 6.4. Обследование ротовой полости | 51 |
| 6.5. Показатели жизненных функций, масса тела и рост | 51 |
| 6.6. Оценочные шкалы | 52 |

КОНФИДЕНЦИАЛЬНО

| 6.7. | Определение времени до первого ощутимого снижения интенсивности боли | |
|---|---|---|
| (ВПС | Б) и времени до значительного снижения интенсивности боли (ВЗСБ) | 52 |
| 6.8. | Безопасность и нежелательные явления | 53 |
| 6.8. | 1. Определения | 53 |
| 6.8. | 2. Беременность | 54 |
| 6.8. | 3. Регистрация нежелательных явлений и серьезных нежелательных явлений | 55 |
| 6.8. | 4. Оценка тяжести | 56 |
| 6.8. | 5. Взаимосвязь с исследуемым препаратом | 56 |
| 6.8. | 6. Оценка ожидаемости | 57 |
| 6.8. | 7. Регистрация серьезных нежелательных явлений и случаев беременности | 57 |
| 6.8. | 8. Передозировка препарата | 58 |
| 6.9. | Досрочное исключение участника из исследования | 58 |
| 7. B | ВИЗИТЫ ИССЛЕДОВАНИЯ | 60 |
| 7.1. | Скрининг (Дни от -3 до 1) | 60 |
| 7.2. | Исследуемая терапия (День 1) | 60 |
| 7.3. | Досрочное прекращение участия в исследовании (День 1) | 61 |
| 7.4. | Период Наблюдения (День 3 ±1 день) | 61 |
| 7.5. | Незапланированные визиты | 62 |
| 8. K | СОНТРОЛЬ КАЧЕСТВА | 63 |
| 9. Г | ІЛАН СТАТИСТИЧЕСКОЙ ОБРАБОТКИ | 64 |
| 9.1. | Общие соображения | 64 |
| 9.2. | Определение размера популяции | 64 |
| 9.3. | Рандомизация | 64 |
| 9.4. | Популяции пациентов для анализа | 65 |
| 9.4. | 1. Популяция назначенной терапии (ITT популяция) | 65 |
| 9.4. | 2. Популяция изучения безопасности | 65 |
| 9.4. | 3. Популяция по протоколу | 65 |
| 9.4. | · | 65 |
| 9.5. | Демографические данные и исходные характеристики | 66 |
| 9.6. | Анализы эффективности | 66 |
| 9.6. | | 66 |
| 9.6. | | 66 |
| 9.7. | Анализы безопасности | 67 |
| Cep | оъезные нежелательные явления | 68 |
| 10. | АДМИНИСТРАТИВНЫЕ ПРОЦЕДУРЫ | 69 |
| 10.1. | | 69 |
| 10.2. | | 69 |
| 10.3. | Процедуры мониторинга | 69 |
| 10.4. | | 70 |
| 10.5. | Хранение записей | 70 |
| 10.6. | • | 70 |
| 10.6 | | 70 |

| | л исследования KSL0117 Финальная 26 сентября 2017 года (в редакции | naceutici s.p.a.<br>от 25 января<br>2018 года) |
|---|---|---|
| 10.6 | 2. Некоторые вопросы, касающиеся этики | 70 |
| 10.6 | 3. Информированное согласие | 71 |
| 10.7. | Финансирование | 71 |
| 10.8. | Политика в отношении публикаций | 71 |
| 11. | ЛИТЕРАТУРНЫЕ ССЫЛКИ | 73 |
| 12. | ПРИЛОЖЕНИЕ | 76 |
| 12.1. | Визуально-аналоговая шкала "Интенсивность боли" | 76 |
| 12.2. | Визуально-аналоговая шкала "Снижение интенсивности боли" | 76 |
| 12.3. | Общая оценка, проведенная самими пациентами (по 5-балльной шкале | ) 76 |
| СПИС | ОК ТАБЛИЦ | |
| Табли | а 1 Расписание визитов и процедур | 27 |
| Табли | | |
| получ | нные в ходе исследования KSL0112 | 37 |
| СПИС | ОК РИСУНКОВ | |
| Рисун | к 1. Профили средних концентраций кетопрофена в плазме крови (м | ікг/мл) с |
| течени | ем времени после приема 40 мг лизиновой соли кетопрофена в форме г | ранул, |
| - | римых в полости рта (T) (• непрерывная линия), и 40 мг лизиновой сол | |
| | офена в форме гранул для приготовления раствора для перорального пр | |
| пункт | рная линия), показанные на полулогарифмической шкале | |
| Рисун | | |
| Рисун | к 3 Маркировка пакетика с исследуемым препаратом | 49 |

КОНФИДЕНЦИАЛЬНО Страница 17 из 76

# СПИСОК СОКРАЩЕНИЙ

| ADME | Всасывание, распределение, метаболизм и выведение (Absorption, distribution, metabolism and excretion) |
|---|---|
| AUC | Площадь под кривой изменения концентрации в зависимости от времени |
| CFS | Надосадочная жидкость, не содержащая клеток (Cell-free supernatant) |
| GLP | Надлежащая лабораторная практика (Good laboratory practice) |
| IASP | Международная ассоциация по изучению боли (International Association for the Study of Pain) |
| ICSRs | Индивидуальные отчеты по безопасности (Individual case safety reports) |
| MedDRA | Медицинский словарь нормативно-правовой деятельности (Medical Dictionary for Regulatory Activities) |
| NZW | Новозеландский белый (New Zealand White) |
| OA | Остеоартрит |
| PID | Различие в интенсивности боли (Pain intensity different) |
| SAP | План статистического анализа (Statistical analysis plan) |
| SDV | Проверка первичных данных (Source Data Verification) |
| SmPC | Краткая характеристика лекарственного препарата (Summary of Product Characteristics) |
| SOC | Класс систем и органов |
| TC | Телефонный контакт (Telephone contact) |
| TEAEs | Нежелательные явления, возникшие на фоне проводимой терапии (Treatment-Emergent Adverse Events) |
| TK | Токсикокинетика |
| АД | Артериальное давление |
| AK | Арахидоновая кислота |
| АЛТ | Аланиновая трансаминаза аланинаминотрансфераза |
| АСК | Ацетилсалициловая кислота |
| Б/р | Безрецептурный |
| БАД | Биологически активные добавки |
| в/в | Внутривенно |
| ВАШ | Визуально-аналоговая шкала |
| ВДП | Визит досрочного прекращения |
| ВЗСБ | Время до значимого снижения боли |
| ВПСБ | Время до первого ощутимого снижения боли |

| ДИ | Доверительный интервал |
|------|------------------------------------------------------|
| ДНК | Дезоксирибонуклеиновая кислота |
| ДП | Досрочное прекращение (видит досрочного прекращения) |
| EC | Европейский Союз |
| ЖКТ | Желудочно-кишечный тракт |
| 3T | Завершение терапии |
| ИЛП | Исследуемый лекарственный препарат |
| ИМТ | Индекс массы тела |
| ИРК | Индивидуальная регистрационная карта |
| КИО | Контрактная исследовательская организация |
| КК | Кетопрофеновая кислота |
| КЛС | Кетопрофена лизиновая соль |
| КП | Кетопрофен |
| КФК | Креатинфосфокиназа |
| M3 | Министерство здравоохранения |
| МКБ | Международная классификация болезней |
| НЛР | Нежелательная лекарственная реакция |
| НПВП | Нестероидные противовоспалительные препараты |
| НЭК | Независимый этический комитет (локальный) |
| RH | Нежелательные явления |
| ПГ | Простагландины |
| ПД | Пищевая добавка |
| ПРТ | Препараты для резервной терапии |
| PA | Ревматоидный артрит |
| РΠ | Рецептурные препараты |
| СНЛР | Серьезная нежелательная лекарственная реакция |
| СНЯ | Серьезное нежелательное явление |
| СОП | Стандартные операционные процедуры |
| CCC | Сердечно-сосудистая система |
| ФД | Фармакодинамика, фармакодинамический |
| ФЖЕЛ | Форсированная жизненная емкость легких |
| ФК | Фармакокинетика, фармакокинетический |
| ЦНС | Центральная нервная система |
| ЦОГ | Циклооксигеназа |
| Ч | Час |

| ЧСС | Частота сердечных сокращений |
|------|--------------------------------------------------|
| эИРК | Электронная индивидуальная регистрационная карта |
| ЭКГ | Электрокардиограмма/электрокардиография |

#### 1. ВВЕДЕНИЕ

Нестероидные противовоспалительные препараты (НПВП) представляют собой химически неоднородную группу веществ, часто не связанных между собой химически, которые обладают общими терапевтическими эффектами и нежелательными реакциями. Основные терапевтические эффекты нестероидных противовоспалительных препаратов происходят из их способности ингибировать синтез простагландинов, подавляя важный фермент в пути синтеза простагландинов, циклооксигеназу или ЦОГ. Все нестероидные противовоспалительные препараты обладают жаропонижающими, обезболивающими и противовоспалительными свойствами и часто применяются для лечения воспалительных заболеваний особенной нарушений со стороны опорно-двигательного аппарата, для которых характерны боль и воспаление. Наиболее частыми нежелательными реакциями на нестероидные противовоспалительные препараты являются эффекты со стороны желудочно-кишечного тракта и сердечно-сосудистой системы [1].

Лизиновая соль кетопрофена (КЛС), которая была представлена в Италии в 1980 году, обладает подтвержденными противовоспалительными и жаропонижающими свойствами, которые более выражены по сравнению с кетопрофеном, что обусловлено ее более высокой растворимостью, которая позволяет применять препарат во множестве разных лекарственных форм, использовать разные высокие дозы и дает стабильный профиль переносимости [3].

Получение аминокислотных солей кетопрофена значительно повысило его растворимость в воде, что позволило разработать жидкие лекарственные формы кетопрофена для перорального приема и получить три основных клинических преимущества: 1) более быстрое всасывание из желудочно-кишечного тракта (ЖКТ) по сравнению с исходным веществом; 2) более быстрое противовоспалительное и обезболивающее действие; 3) более кратковременное пребывание активного вещества в желудке и, следовательно, более низкий потенциал раздражающего действия и/или эффектов, приводящих к возникновению язв.

В сравнительных исследованиях кетопрофен не уступал по эффективности другим противовоспалительным и обезболивающим препаратам [3]. Для кетопрофена характерны те же побочные эффекты, что и для других нестероидных противовоспалительных препаратов, при этом наиболее часто отмечаются нарушения со стороны желудочнокишечного тракта: тошнота, рвота, диарея, вздутие живота, запор, диспепсия, боль в животе, реже – пептические язвы, перфорация, гастрит или желудочно-кишечное кровотечение [3]. Приблизительно у 30% лиц, получающих кетопрофен, возникают побочные эффекты со стороны желудочно-кишечного тракта легкой степени, частота и интенсивность которых снижаются, если препарат принимать вместе с пищей или антацидами [3]. К другим, менее частым нежелательным эффектам кетопрофена, относятся нарушения со стороны кожи (крапивница, эритема, кожная сыпь), общие нарушения (аллергические и анафилактоидные реакции), нарушения со стороны нервной системы (головокружение и вертиго), нарушения со стороны сердечно-сосудистой системы (ощущения учащенного сердцебиения, тахикардия, артериальная гипотензия и артериальная гипертензия), нарушения со стороны дыхательной системы (бронхоспазм, одышка), нарушения со стороны почек (задержка воды в организме), а также нарушения кроветворения и нарушения со стороны мочевыводящих путей. В большинстве случаев симптомы преходящие и разрешаются при приостановке терапии, а также при применении специфической лекарственной терапии.

Лизиновая соль кетопрофена в форме гранул для приготовления раствора для перорального приема  $(OKi^{®})$  в пакетиках по 80 мг, содержащих 80 мг лизиновой соли кетопрофена в сдвоенном пакетике, по 40 мг лизиновой соли кетопрофена в каждой из

частей) уже зарегистрирована и продается компанией "Dompé" в Италии с 1994 года и в России с 1998 года в качестве средства для кратковременного лечения симптомов воспалительных состояний, сопровождающихся болью.

Кетопрофен в форме гранул в пакетиках по 40 мг был зарегистрирован в Италии в 2001 году для лечения боли разного типа и происхождения (головная боль, зубная боль, невралгия, боль при менструациях, боль в мышцах и боль, вызванная остеоартритом), но не распространялся на рынке.

В сниженной дозе, составлявшей 25 мг (что соответствует 40 мг лизиновой соли кетопрофена в форме гранул), препарат изучался у человека в качестве обезболивающего. Разные формы кетопрофена в дозе 25 мг для перорального приема зарегистрированы в Европейском Союзе разными владельцами регистрационных удостоверений под разными торговыми марками (например, Toprec<sup>®</sup> производства компании "Sanofi-Aventis", Франция; Торгек<sup>®</sup> производства компании "Sanofi-Aventis", Италия; Fastum<sup>®</sup> производства компании "Menarini", Италия).

Новая лекарственная форма кетопрофена в виде лизиновой соли в дозировке 40 мг для перорального приема (что соответствует 25 мг кетопрофена) аналогична по содержанию активного вещества уже зарегистрированной лекарственной форме кетопрофена в дозировке 25 мг для перорального приема. Препарат ОКИТАСК в гранулах по 40 мг (лизиновая соль кетопрофена 40 мг, что соответствует 25 мг кетопрофена) была выведена на рынок в Италии в 2012 году для применения по следующим показаниям: боль разных видов и происхождения, в особенности головная боль, зубная боль. невралгия, а также менструальная и мышечная боль и боль, вызванная остеоартритом. Кроме того, препарат ОКИТАСК в гранулах по 40 мг с мая 2015 года распространяется на рынке в Албании, а с июля 2016 года — в Косово; новая лекарственная форма препарата ОКИТАСК в таблетках по 40 мг была зарегистрирована в Италии в феврале 2017 года.

Установленная в ходе клинических исследований токсикологии безопасность лизиновой соли кетопрофена сравнима с таковой у кетопрофена; более того, в связи с более быстрым всасыванием время пребывания препарата в желудочно-кишечном тракте должно быть снижено, а следовательно, у человека ожидается боле низкая вероятность раздражения желудочно-кишечного тракта.

Оценка безопасности гранул препарата  $OKi^{\&}$  для приготовления раствора для перорального приема и капель  $OKi^{\&}$  у человека была проведена в рамках клинических исследований, выполненных с применением лизиновой соли кетопрофена для перорального приемка (как в ходе исследований фармакокинетики, так и в ходе исследований клинической эффективности) при тщательном мониторинге всех нежелательных явлений (НЯ) и нежелательных лекарственных реакций (НЛР), возникавших в ходе этих исследований. Кроме того, было проведено специфическое исследование безопасности с целью изучения способности лизиновой соли кетопрофена вызывать раздражение и/или образование язв в желудочно-кишечном тракте.

Исключительно низкая частота нежелательных явлений после терапии с применением лизиновой соли кетопрофена и развитие таких нежелательных явлений у участников исследований, получавших плацебо, указывают на очень хороший профиль безопасности как у гранул  $OKi^{\text{®}}$ , так и у капель  $OKi^{\text{®}}$  [3].

Опыт постмаркетингового применения разных лекарственных форм препарата  $OKi^{\otimes}$  показывает, что нежелательные явления развиваются довольно редко. Тем не менее, частоту нежелательных эффектов можно свести к минимуму, применяя самые низкие эффективные дозы новой лекарственной формы лизиновой соли кетопрофена в дозировке 40 мг в виде гранул для перорального приема, растворимых в ротовой полости. В

Исследуемый препарат ОКИТАСК® Протокол исследования KSL0117 Финальная версия 1.0

Dompé farmaceutici s.p.a. 26 сентября 2017 года (в редакции от 25 января 2018 года)

действительности соответствующая доза кетопрофена в виде кислоты составляет 25 мг вместо 50 мг, содержащейся в одном пакетике препарата  $OKi^{\mathbb{R}}$  в гранулах по 80 мг для приготовления раствора для перорального приема.

Настоящее исследование было разработано для того чтобы установить эффективность препарата  $OKUTACK^{\mathbb{R}}$  в гранулах по 40 мг для перорального приема на модели боли легкой и умеренной степени в целях дальнейшей регистрации указанного препарата в России.

# 2. ЦЕЛИ ИССЛЕДОВАНИЯ

#### 2.1. Основная цель

Основной целью данного исследования является оценка эффективности препарата ОКИТАСК<sup>®</sup> в гранулах по 40 мг в сравнении с плацебо у пациентов с острым болевым синдромом после удаления одного моляра, проводимая путем сравнения  $AUC_{0-64}$  профиля боли после терапии, измеряемой с помощью визуально-аналоговой шкалы.

#### 2.2. Дополнительные цели

K дополнительным целям данного исследования относится оценка следующих параметров эффективности и безопасности препарата ОКИТАСК<sup>®</sup> в гранулах по 40 мг в сравнении с плацебо у пациентов с острой болью после удаления одного моляра:

- Профиль боли в зависимости от времени и профиль снижения интенсивности боли с течением времени по результатам заполнения визуально-аналоговой шкалы
- Время до первого ощутимого снижения интенсивности боли (ВПСБ) и время до значительного снижения интенсивности боли (ВЗСБ)
- Доля пациентов, которым требуется терапия спасения (обезболивание) и время до приема терапии спасения
- Общая оценка, проведенная самими пациентами
- Частота нежелательных явлений (НЯ)

# 3. ДИЗАЙН ИССЛЕДОВАНИЯ

#### 3.1. Общий дизайн и план исследования

Это многоцентровое двойное слепое рандомизированное, плацебо-контролируемое исследование в параллельных группах с целью оценки эффективности и переносимости кетопрофена лизиновой соли в форме гранул в дозе 40 мг в сравнении с плацебо у мужчин и женщин с острым болевым синдромом после удаления моляра.

Исследование будет проводиться в 4-6 исследовательских центрах в России. Ожидается, что в него будет включено в совокупности 70 пациентов (по 35 в каждой группе). Набор пациентов в исследовательских центрах является конкурентным.

#### 3.1.1. Дизайн исследования

Само исследование будет состоять из трех периодов: период скрининга, период исследуемой терапии и период наблюдения.

# *3.1.1.1.* Скрининг

В период скрининга после подписания информированного согласия у пациента в рамках определения критериев включения/невключения будут собраны демографические данные, медицинский анамнез и данные по сопутствующей лекарственной терапии, выполнен осмотр ротовой полости, проведены взвешивание и оценка показателей функций жизненно-важных органов, а кроме того, пациентам женского пола будет выполнен тест на беременность. Процедуры скрининга могут занять до 4 дней перед плановым удалением зуба, включая сам день, в который будет удален зуб.

В День 1 пациенту будет выполнено удаление моляра в соответствии с показаниями, обусловленными состоянием зубов. Удаление зуба будет проведено с применением стандартной методики и методов анестезии (рекомендованные типы анестезии представлены в Разделе 5.9 "Сопутствующая терапия и терапия спасения" данного

протокола исследования). После этого пациент останется в исследовательском центре для лечения болевого синдрома в соответствии с протоколом исследования.

Оценка интенсивности боли будет проводиться с применением визуально-аналоговой шкалы в течение 3 часов после процедуры удаления зуба. Кроме того, будет регистрироваться оценка, которую будет проводить сам пациент. Если интенсивность боли по визуально-аналоговой шкале будет выше 30 мм и потребуется обезболивание, то пациент будет рандомизирован в это исследование.

#### 3.1.1.2. Исследуемая терапия

При рандомизации пациенты распределяются в соотношении 1:1 в одну из двух групп:

Группа 1. Терапия препаратом ОКИТАСК ${\Bbb R}$  в дозе 40 мг – 35 пациентов

Группа 2. Терапия плацебо – 35 пациентов.

До получения получения исследуемого препарата (момент времени 0') пациент проведет оценку боли по визуально-аналоговой шкале.

Сразу же при приеме исследуемого препарата пациенты должны запустить два секундомера. Один из них должен быть остановлен сразу же, как только пациент почувствует заметное снижение боли, а второй — после того как пациент почувствует значительное снижение боли.

Пациент будет оставаться в исследовательском центре в течение 6 часов после приема исследуемого препарата для оценки боли и нежелательных явлений. Интенсивность боли будет оцениваться по визуально-аналоговой шкале через 5 минут, 10 минут, 15 минут, 30 минут, 45 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) минут после приема препарата.

Оценка снижения интенсивности боли будет проводиться по визуально-аналоговой шкале через 5 минут, 10 минут, 15 минут, 30 минут, 45 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) минут после приема препарата.

Пациенты должны указывать действительное время проведения оценки по визуальноаналоговой шкале. Отклонения от запланированных временных точек не будут считаться отклонениями от протокола исследования. Отклонением от протокола исследования будет считаться только пропуск оценок.

Непосредственно перед тем, как пациент покинет исследовательский центр, ему предложат провести оценку своего состояния по шкале Общей оценки, проведенной самими пациентами.

Если пациенту потребуется применение дополнительной лекарственной терапии в любое время в течение 6 часов после приема исследуемого препарата, то последняя оценка боли по визуально-аналоговой шкале и общая оценка лечения пациентом своего состояния по шкале Общей оценки, проведенной самими пациентами, должны быть выполнены перед получением препаратов терапии спасения.

# 3.1.1.3. Контрольное наблюдение

В День 3 (через 48 часов после приема исследуемого препарата) будет проведен телефонный разговор с пациентом для оценки нежелательных явлений. Необходимо будет зарегистрировать любые серьезные нежелательные явления, о которых пациент спонтанно

Исследуемый препарат ОКИТАСК  $^{\text{®}}$  Протокол исследования KSL0117 Финальная версия 1.0

Dompé farmaceutici s.p.a. 26 сентября 2017 года (в редакции от 25 января 2018 года)

сообщит в течение 30 дней после приема исследуемого препарата. Расписание процедур исследования приведено в Таблице 1.

Таблица 1 Расписание визитов и процедур исследования

| | | Исследуемая терап | ия | | | | | | | | | | | | | ДЗ <sup>3</sup> | Период<br>наблюдения |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Тест/ обследование | Скрининг | Исходный уровень <sup>1</sup><br>(до приема препарата) | | Время (после приема) | | | | | | | | Телефонный<br>контакт | | | | | |
| День | День -4 -1 | День 1 | | День 1 | | | | | | | | День 1 | День 3±1 | | | | |
| Часы | | 0 | | 0,08 | 0,17 | 0,25 | 0,5 | 0,75 | 1 | 1,5 | 2 | 3 | 4 | 5 | 6 | > 1 | 48 |
| Минуты | | 0 | | 5 | 10 | 15 | 30 | 45 | 60 | 90 | 120 | 180 | 240 | 300 | 360 | > 60 | |
| Информированное согласие и присвоение<br>скринингового номера | X | | | | | | | | | | | | | | | | |
| Демографические данные | X | | | | | | | | | | | | | | | | |
| Медицинский анамнез и сопутствующие<br>заболевания | X | | 0 | | | | | | | | | | | | | | |
| Обследование ротовой полости | X | | (eQ | | | | | | | | | | | | | | |
| Poct <sup>6</sup> | X | | плацебо | | | | | | | | | | | | | | |
| Масса тела | X | | / п. | | | | | | | | | | | | | | |
| Жизненные показатели | X | | Та | | | | | | | | | | | | | | |
| Тест на беременность | X | | apa | | | | | | | | | | | | | | |
| Удаление моляра | Х (День 1) | | еп | | | | | | | | | | | | | | |
| Оценка интенсивности боли по ВАШ (0-100 мм) <sup>7</sup> | X | X | исследуемого препарата/ | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Критерии включения/ невключения <sup>2</sup> | X | | емо | | | | | | | | | | | | | | |
| Присвоение рандомизационного номера | | X | еду | | | | | | | | | | | | | | |
| Шкала Общей оценки, проведенной самими пациентами (5-балльная шкала) <sup>7</sup> | | X | иссл | | | | | | | | | | | | X | X | |
| Оценка снижения интенсивности боли по ВАШ (0-100 мм) <sup>7</sup> | | | Прием | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Время до первого ощущения снижения интенсивности боли (ВПСБ), измеренное с помощью секундомера <sup>4</sup> | | | T X | | | | | | | | | | | | | | |
| Время до значительного снижения интенсивности боли (ВЗСБ), измеренное с помощью секундомера <sup>4</sup> | | X | | | | | | | | | | | | | | | |
| Терапия спасения (если применимо) <sup>6</sup> | | | | | | | | | X <sup>5</sup> | | | | | | | | |
| Сопутствующая терапия | X | X | | | | | | | X | | | | | | | X | X |
| Предыдущая терапия | X | X | | | | | | | | | | | | | | | |
| Нежелательные явления | X | X X X | | | | | | X | | | | | | | | | |

1. После удаления зуба, перед приемом исследуемого препарата

2. Подтверждение критериев включения/ невключения перед рандомизацией

3. Если пациенту потребуется применение терапии спасения в любое время в течение 6 часов после приема исследуемого препарата, то последняя оценка боли по визуально-аналоговой шкале и общая оценка, проведенная самими пациентами, должны быть выполнены перед получением препаратов терапии спасения.

КОНФИДЕНЦИАЛЬНО Страница 27 из 76

Участникам исследования будет предложено воздерживаться от приема терапии спасения в течение одного часа после приема исследуемого препарата. Оценки при досрочном прекращении исследования будут проведены до получения пациентом терапии спасения; должно быть зарегистрировано действительное время заполнения визуально-аналоговой шкалы.

- 4. Время, зарегистрированное секундомером, должно быть записано в эИРК
- 5. В случае плохого контроля боли пациентам будет разрешено получить терапия спасения для обезболивания (Парацетамол в дозе 500-1000 мг). Время до приема резервного обезболивающего препарата, если такое произойдет, также должно быть зарегистрировано. Участникам исследования будет предложено воздерживаться от приема терапии спасения в течение одного часа после приема исследуемого препарата. Если парацетамол в дозе 500-1000 мг окажется неэффективным, пациенту будет разрешено принять еще по 500-1000 мг парацетамола каждые 6-8 часов; максимальная суточная доза составляет 4000 мг.
- 6. Рост регистрируется со слов пациента.
- 7. Пациенты должны указывать фактическое время проведения оценки по визуально-аналоговой шкале. Отклонения от запланированных временных точек не будут считаться отклонениями от протокола исследования. Отклонениями от протокола исследования будут считаться только пропуски оценок.

КОНФИДЕНЦИАЛЬНО Страница 28 из 76

#### 3.2. Обоснование дизайна исследования

Это многоцентровое двойное слепое рандомизированное исследование в параллельных группах с целью оценки эффективности и переносимости кетопрофена лизиновой соли в форме гранул в дозе 40 мг в сравнении с плацебо у мужчин и женщин с острым болевым синдромом после удаления моляров.

Исследование было разработано для определения эффективности и безопасности препарата ОКИТАСК<sup>®</sup> в гранулах по 40 мг для перорального приема на модели боли легкой и умеренной степени тяжести. Удаление моляра является моделью острой хирургической боли, которая позволяет проводить сбор данных для определения профиля боли в клиническом центре в заданном периоде времени [2]. Демонстрация превосходства исследуемого препарата в сравнении с плацебо служит в качестве подтверждения чувствительности данной модели боли.

Демонстрация эффективности и безопасности препарата ОКИТАСК в гранулах по 40 мг в виде части клинического досье для регистрации новой лекарственной формы лизиновой соли кетопрофена в России была выбрана в качестве наиболее подходящего дизайна исследования. Данные по биоэквивалентности по этому препарату доступны из исследования препарата ОКИТАСК в гранулах по 40 мг в сравнении с гранулами ОКі для приготовления раствора для перорального приема, проведенного в Швейцарии в 2015 году [9].

Дизайн многоцентрового двойного слепого рандомизированного исследования в параллельных группах с плацебо-контролем является стандартным дизайном адекватных и хорошо контролируемых исследований.

Препарат ОКИТАСК представляет собой лизиновую соль кетопрофена; 40 мг препарата ОКИТАСК соответствуют 25 мг кетопрофена, которые являются рекомендованной начальной дозой для обезболивания при безрецептурном применении препарата.

Использование плацебо в данной модели является приемлемым и этически оправдано, поскольку 1) нет риска для безопасности и благополучия пациента и 2) в случаях, когда исследуемый препарат или плацебо не позволят достичь достаточного уровня снижения интенсивности боли, пациентам будет предоставлена терапия спасения. Участникам исследования будет предложено воздерживаться от приема терапии спасения в течение одного часа после приема исследуемого препарата. Парацетамол в дозе 500-1000 мг был выбран в качестве препарата терапии спасения, поскольку от относится к другой фармацевтической группе обезболивающих препаратов, что позволит избежать взаимодействия между препаратами. Если прием Парацетамола не даст нужного эффекта, пациентам будет разрешено принимать парацетамол в дозе 500-1000 мг каждые 6-8 часов; интервал между приемами не должен быть меньше 4 часов; максимальная суточная доза составляет 4000 мг.

В ходе этого исследования будет проводиться оценка снижения интенсивности боли после удаления моляра. Поскольку боль всегда субъективна, ее наиболее точное измерение получается при использовании шкал, заполняемых самими пациентами. В настоящее время нет валидированных объективных способов измерения боли, которые моно было бы использовать в условиях клинических исследований. Интенсивность боли (pain intensity, PI) остается ключевым показателем эффективности обезболивающих препаратов и будет регистрироваться в ходе этого исследования. Для оценки интенсивности боли и ее снижения в этом исследовании будет использоваться визуально-аналоговая шкала (ВАШ). Первичной конечной точкой будет AUC<sub>0-64</sub> профиля боли от момента 0 (исходное значение на визуально-аналоговой шкале) до 6 часов после начала

КОНФИДЕНЦИАЛЬНО Страница 29 из 76

терапии. Оценка в течение 6 часов соответствует профилю фармакокинетики лизиновой соли кетопрофена с  $T_{max}$  в пределах 0,75-1 часа и  $T_{1/2}$  1,5-2 часов.

В качестве вторичных конечных точек в ходе данного исследования будут оцениваться профиль боли и профиль снижения интенсивности боли с течением времени, измеряемые по шкале ВАШ, время до первого ощутимого снижения интенсивности боли (ВПСБ), время до первого значительного снижения боли (ВЗСБ), доля пациентов, которым потребовалась терапия спасения, время до получения терапии спасения и общая оценка, проводимая самими пациентами. Измерение времени до первого ощутимого снижения интенсивности боли и времени до первого значительного снижения боли будет проводиться с помощью двух секундомеров.

Предполагается, что лизиновая соль кетопрофена будет безопасной. Наблюдение за пациентами будет проводиться в течение 48 часов после приема исследуемого препарата, что превышает 7 периодов полувыведения лизиновой соли кетопрофена. Любые серьезные нежелательные явления, о которых пациент спонтанно сообщит в течение 30 дней после приема исследуемого препарата, должны быть зарегистрированы.

Гипотеза исследования и размер выборки основаны на данных, полученных в ходе плацебо-контролируемого исследования кетопрофена (разница между группами по средней AUC 90 мм ч-1 и стандартном отклонении 121 мм ч-1), в ходе которого  $\alpha = 0.05$ , а мощность составила 80% [3].

#### 3.3. Длительность исследования

Длительность участия каждого из пациентов в этом исследовании составит до  $7\pm1$  день и будет включать следующие этапы: скрининг (до 4 дней), удаление зуба, рандомизация и прием исследуемой терапии (1 день) и период наблюдения (2 дня).

Начало набора пациентов в исследование планируется на октябрь 2017 года. Также планируется, что все пациенты выполнят все визиты исследования до марта 2018 года. Окончанием исследования считается дата последнего визита последнего пациента. Отчет по клиническому исследованию будет закончен в июне 2018 года.

# 3.4. Ранее полученный опыт применения препарата ОКИТАСК®

Боль является наиболее частым симптомом, в связи с которым пациенты обращаются за медицинской помощью. При том, что точного определения боли не существует, она может быть определена как неприятные ощущение и эмоциональный опыт, связанные с имеющимся или возможным повреждением тканей или описываемые как такое повреждение (определение IASP). Острая и хроническая боль являются разными клиническими проблемами. Острая боль вызывается специфическим заболеванием или повреждением, служит полезным биологическим предупреждением, связана со спазмом скелетных мышц и активацией симпатической нервной системы и сама прекращается [6].

Нестероидные противовоспалительные препараты играют установленную роль в снижении интенсивности слабой или умеренной боли, малых лихорадочных состояний, а также при острых и хронических воспалительных нарушениях, таких как остеоартрит, ревматоидный артрит, ювенильный идиопатический артрит и анкилозирующий спондилит. Ацетилсалициловая кислота, диклофенак, ибупрофен и напроксен являются известными нестероидными противовоспалительными препаратами подтвержденной эффективностью при самостоятельном лечении заболеваний, сопровождающихся болью слабой или умеренной интенсивности и лихорадкой. Максимальные концентрации наиболее быстро действующих из этих активных веществ при применении в безрецептурных лекарственных формах достигаются ( $T_{max}$ ) через 20-60 минут (таблетки диклофенака натрия), значения  $T_{max}$  совпадают с началом снижения боли

КОНФИДЕНЦИАЛЬНО Страница 30 из 76

и могут значительно варьироваться, например,  $T_{max}$  для напроксена составляет от 2 до 4 часов. Количество лекарственных форм и форм выпуска этих препаратов ограничено, при этом для приема большинства из них требуется вода. Существует потребность в безрецептурном обезболивающем препарате, который бы быстро действовал и обладал уникальной формой, дающей эффект "на ходу".

Кетопрофен, производное пропионовой кислоты, является хорошо известным и применяемым нестероидным противовоспалительным препаратом с доказанной анальгетической, противовоспалительной и жаропонижающей активностью. Он был впервые одобрен для клинического применения во Франции и в Великобритании в 1973 году. В настоящее время он применяется во всем мире во множестве разных лекарственных форм, таких как капсулы, растворы для инъекций, свечи и гели для местного нанесения [7].

Он часто прописывается для лечения заболеваний опорно-двигательного аппарата и суставов, таких как анкилозирующий спондилит, остеоартрита и ревматоидный артрит, а также при заболеваниях околосуставных структур, таких как бурсит и тендинит. Кроме того, он применяется при дисменорее, при послеоперационной боли, для лечения болезненных и воспалительных заболеваний, таких как острая подагра или заболевания мягких тканей, а также для подавления лихорадки.

В качестве безрецептурного препарата кетопрофен одобрен для лечения большого количества заболеваний, сопровождающихся болью слабой или умеренной интенсивности, а также для облегчения лихорадки [8].

Химическое наименование кетопрофена следующее: 2-(3-бензоилфенил)-пропионовая кислота, а молекулярная формула  $C_{16}H_{14}O_3$ . Кетопрофену присвоен код ATX M01AE03. Фармакопейные лекарственной формы кетопрофена по Британской фармакопее (BP) от 2014 года следующие: кетопрофен в капсулах; кетопрофен гель; по Фармакопее США версии 36: кетопрофен в капсулах с замедленным высвобождением.

Лизиновая соль кетопрофена (КЛС) является солью кетопрофена, для которой наличие противовоспалительных, обезболивающих подтверждено тех же жаропонижающих свойств, что и у исходного вещества, кетопрофена. Образование соли аминокислотой кетопрофена с лизином значительно повышает растворимость кетопрофена в воде, повышает скорость и объем всасывания (Ттах 15 минут) по сравнению с обычной кислотой кетопрофена, а также с применяемыми безрецептурными нестероидными противовоспалительными препаратами; в ходе исследований было установлено что образование лизиновой соли кетопрофена дает гастропротективный эффект, что подтверждается данными полученными при применении лизиновой соли кетопрофена в стандартной практике, когда при применении этой лекарственной формы отмечалось меньше реакций со стороны желудочно-кишечного тракта, чем при применении ибупрофена и, следовательно, это дает основу для разработки гранул для перорального приема, растворимых в ротовой полости [10].

Лизиновая соль кетопрофена представлена в лекарственной форме гранул по 40 мг, растворимых в ротовой полости (далее в этом документе будут упоминаться как лизиновая соль кетопрофена (КЛС) в гранулах по 40 мг), которые эквивалентны 25 мг кетопрофена, что было подтверждено при эффективности более низкой дозы положительном соотношении профиля пользы и риска для безрецептурной лекарственной формы кетопрофена. Содержимое пакетика помещается прямо на язык. Гранулы растворятся в слюне и, таким образом, могут удобно применяться без воды, что дает хорошую альтернативу людям с нарушениями глотания, которым трудно глотать обычные капсулы и таблетки. Было установлено, что лизиновая соль кетопрофена в форме гранул

КОНФИДЕНЦИАЛЬНО Страница 31 из 76

по 40 мг эффективна в отношении контроля слабой или умеренной боли, при этом снижение интенсивности боли начиналось через 5 минут после приема.

Согласно Краткой характеристике лекарственного препарата для лизиновой соли кетопрофена в гранулах по 40 мг, показания, утвержденные для этого препарата в Италии, следующие: боль разных типов и происхождения, особенно головная боль, зубная боль, невралгия, менструальная боль, ревматическая боль и мышечные боли.

Лизиновая соль кетопрофена показана к применению у взрослых лиц и подростков в возрасте 15 лет и старше.

Предполагаемая дозировка составляет 40 мг лизиновой соли кетопрофена (что эквивалентно 25 мг кетопрофена) до 3 раз в стуки у взрослых лиц и подростков в возрасте 15 лет и старше.

Все предлагаемые показания характеризуются кратковременной, острой болью и могут быть диагностированы самими пациентами.

#### 3.4.1. Доклинические данные

При остром воздействии лизиновой соли кетопрофена у крыс и мышей при пероральном или внутрибрющинном введении достигались очень высокие дозы (средняя доза, вызывающая гибель 50% подопытных животных ( $LD_{50}$ ) составила более 100 мг/кг у крыс и более 400 мг/кг у мышей) [11], [12], [13], [14], [15].

В ходе исследований фармакологии и по данным литературы было установлено, что лизиновая соль кетопрофена обладает противовоспалительной, обезболивающей и жаропонижающей активностью, описанной ранее для исходного вещества, кетопрофена в форме свободной кислоты, и подтверждает терапевтические показания для применения регистрируемого препарата (лизиновая соль кетопрофена 40 мг в гранулах, растворимых в ротовой полости).

В исследовании с моделированием отека в конечности крысы, вызванного каррагинаном, лизиновая соль кетопрофена применялась либо местно в виде пены, наносившейся на кожу, либо перорально в дозах 0,5, 1 и 2 мг/кг (за 1 час до инъекции каррагинана) статистически значимо снижала образование отека, при этом наиболее выраженный эффект отмечался при пероральном введении лизиновой соли кетопрофена в дозе 2 мг/кг.

В дальнейшем исследовании с оценкой жаропонижающей активности у крыс, лизиновая соль кетопрофена применялась перорально в дозах до 3 мг/кг, что приводило к зависимому от дозы снижению повышенной температуры тела, вызванному дрожжами (самая высокая жаропонижающая активность была отмечена при дозе 3 мг/кг). На модели in vitro с культивированными клетками слизистой оболочки желудка человека, поврежденными под действием этанола, лизин и лизиновая соль кетопрофена явно защищали клетки, поврежденные этанолом, в отличие от кетопрофена в форме свободной кислоты, а кроме того, лизин и лизиновая соль кетопрофена снижали уровни малоового диальдегида (МДА), повышенные под действием этанола, а также подавляли активацию ядерного фактора каппа В (NFkB) и интерлейкина-8 (IL-8). Уровни малонового диальдегида не снижались под действием кетопрофена в форме свободной кислоты, которая лишь в с меньшей активностью снижала уровни NFkB и IL-8. Эти результаты, полученные in vitro, четко показывают защитную роль лизина и лучший профиль переносимости лизиновой соли кетопрофена по сравнению с кетопрофеном в форме свободной кислоты [18].

КОНФИДЕНЦИАЛЬНО Страница 32 из 76

Фармакологические эффекты, полученные на разных моделях на животных, также как и данные, полученные in vitro, однозначно подтверждают предполагаемое клиническое применение и дозы лизиновой соли кетопрофена в форме гранул, растворимых в ротовой полости.

Абсорбция лизиновой соли кетопрофена была изучена на животных после перорального (собаки) и местного (на кожу) применения препарата в форме пены. У собак биодоступность и фармакокинетика лизиновой соли кетопрофена, S-кетопрофена, R-кетопрофена и кетопрофена в ходе 2-недельного исследования с пероральным введением были сравнимы. При эквимолярных дозах активных веществ у лизиновой соли кетопрофена и кетопрофена были выявлены одинаковые профили распределения препарата за 2-часвой период времени, однако средние уровни в плазме крови в первые два момента взятия образцов были существенно выше для лизиновой соли кетопрофена, чем у кетопрофена в виде свободной кислоты, что явно указывает на заметно более раннее начало фармакологической активности лизиновой соли кетопрофена.

Местное нанесение лизиновой соли кетопрофена приводило к незначительным концентрациям кетопрофена в плазме крови (нг/мл) по сравнению с концентрациями, получаемыми после внутривенного введения (мкг/мл); часто эти концентрации были ниже наименьшего предела количественного определения (т.е., ниже 0,05 мкг/мл). В результате был сделан вывод, что после нанесения на кожу значительной системной абсорбции лизиновой соли кетопрофена не происходило.

Эффекты лизиновой соли кетопрофена в отношении сердечно-сосудистой системы были изучены на собаках. Переносимость препарата после внутримышечного или внутривенного введения в дозах до 10 мг/кг была хорошей. Более высокие дозы, введенные внутривенно (25-50 мг/кг) вызывали преходящее повышение артериального давления, а при самой высокой дозе отмечалась легкая артериальная гипотензия. У кроликов лизиновая соль кетопрофена при внутривенном ведении в дозах до 100 мг/кг не вызывала значимых эффектов со стороны сердечно-сосудистой системы. Эта безопасная доза у кроликов дает 16-кратный фактор безопасности при сравнении со 120 мг/сут лизиновой соли кетопрофена в форме, растворимой в полости рта, при применении у человека.

Токсикология лизиновой соли кетопрофена была тщательно изучена в ходе исследований токсичности при однократном и многократном введении, продолжавшемся до 13 недель. Кроме того, были проведены исследования генетической токсичности, репродуктивной токсичности и местной переносимости. У грызунов и животных других отрядов были изучены разные пути введения (в том числе пероральный). Все исследования были выполнены признанными медико-биологическими исследовательскими организациями (Ricerche Biomediche RBM в Италии и Life Science Research в Израиле) и в соответствии с требованиями стандарта Надлежащей лабораторной практики (GLP) [11], [13], [12], [14], [15], [16], [17], [18], [19], [20], [22], [21], [23], [24], [25], [26], [27], [28].

Как и ожидалось для нестероидных противовоспалительных препаратов, основными органами-мишенями у всех изученных видов были желудочно-кишечный тракт и почки. Дозы 2,5 мг/кг/сут и 7,5 мг/кг/сут у крыс и мартышек, соответственно, были дозами, при которых не было отмечено токсических эффектов. Эти результаты аналогичны результатам, представленным в опубликованных результатах токсикологических исследований, проведенных с кетопрофеном в форме свободной кислоты на животных, не относящихся к грызунам.

КОНФИДЕНЦИАЛЬНО Страница 33 из 76

Оценка потенциала мутагенности и генетической токсичности лизиновой соли кетопрофена была проведена в соответствии со стандартным набором исследований in vitro и in vivo. Генотоксической и мутагенной активности у лизиновой соли кетопрофена выявлено не было.

Тератогенных эффектов или эффектов в отношении фертильности или функций системы размножения у кроликов при пероральном введении препарата в дозах 15, 30 и 60 мг/кг/сут выявлено не было. Было отмечено несколько случаев смерти, возможно связанных с эффектами препарата в отношении желудочно-кишечного тракта.

На основе полученных данных по фармакологии и токсикологии, доклинические данные по лизиновой соли кетопрофена подтверждают, что доклинический профиль этого вещества аналогичен таковому для кетопрофена в форме свободной кислоты и полностью подтверждают выбранные дозировки и показания к применению у человека. Потенциально улучшенный профиль переносимости (хорошо подтвержденный при исследовании in vitro с клетками слизистой оболочки желудка человека), более быстрое начало действия и оптимизированная форма лекарственного препарата делают его особенно подходящим для безрецептурного применения.

# 3.4.2. Клинические данные

# Всасывание и распределение

Как было указано Sarzi-Puttini, лизиновая соль кетопрофена обладает более высокой растворимостью по сравнению с кетопрофеном в форме свободной кислоты. Это приводит к более быстрому всасыванию активного вещества с более высокой максимальной концентрацией, которая достигается уже через 15 минут по сравнению с 60 минутами после приема кетопрофена. Быстрое повышение максимальной концентрации лизиновой соли кетопрофена в плазме крови приводит к более быстрому наступлению фармакологической активности, что важно, поскольку быстрота наступления обезболивания является одним из наиболее важных факторов для потребителей, которым требуется облегчение боли [29].

Взаимосвязь между концентрацией и обезболивающими эффектом кетопрофена была установлена в ходе исследования обезболивания кетопрофеном при вмешательствах на ротовой полости. Концентрация кетопрофена, которая приводила к снижению боли на 50% от максимальной ( $Ce_{50}$ ) составила 0,3 мкг/мл (95% доверительные интервалы от 0,1 до 0,5) [10]. В ходе второго исследования биофармацевтических свойств, проведенного с препаратом ОКИТАСК<sup>®</sup> в гранулах по 40 мг при участии 69 человек было установлено, что через 5 минут после приема уровни кетопрофена в плазме крови составляли 0,15 мкг/мл (стандартное отклонение 0,19 мкг/мл). С учетом доверительных пределов для  $Ce_{50}$  (0,1-0,5 мкг/мл) клинически значимые анальгетические эффекты лизиновой соли кетопрофена в гранулах по 40 мг могут наступить через 5 минут после первого перорального приема.

Линейность всасывания была установлена для разных доз кетопрофена, составлявших от 12,5 мг до 200 мг [30].

При приеме кетопрофена вместе с пищей его биодоступность (AUC) не изменялась, однако максимальная концентрация ( $C_{max}$ ) была ниже, а время до наступления максимальной концентрации ( $T_{max}$ ) было дольше. Количество принятой пищи оказывало лишь слабый эффект на объем всасывания кетопрофена [31]. Кетопрофен на 99% связывается с белками плазмы крови, при этом его существенные концентрации выявлены в синовиальной жидкости [32].

КОНФИДЕНЦИАЛЬНО Страница 34 из 76

Лизиновая соль кетопрофена быстро и легко распределяется в центральной нервной системе и может быть выявлена в спинномозговой жидкости через 15 минут после внутримышечного введения кетопрофена в дозе 100 мг. Быстрая диффузия может быть объяснена высоким уровнем растворимости лизиновой соли кетопрофена в липидах, приводящим к быстрому прохождению гематоэнцефалического барьера [33].

#### Метаболизм

Кетопрофен быстро и широко метаболизируется в печени, в основном путем конъюгирования. Кроме того, препарат подвергается гидроксилированию и последующей конъюгации с глюкуроновой кислотой. Глюкуроновый конъюгат кетопрофена и его гидроксилированные метаболиты фармакологически неактивны; активных метаболитов выявлено не было.

## Выделение и полувыведение

Период полувыведения из плазмы крови составляет около 1,5 часов. Метаболизм кетопрофена происходит, в основном, путем конъюгации с глюкуроновой кислотой, а выделение происходит, в основном, с мочой [32].

После однократного перорального приема кетопрофена здоровыми взрослыми лицами приблизительно 60-80% от принятой дозы выделалось с мочой; основная часть вещества выделалась с мочой в течение 24 часов [38]. Выведение препарата у пожилых лиц было снижено [34], что является важным при оценке безопасности лизиновой соли кетопрофена в гранулах по 40 мг в данной популяции пациентов. Связанное с возрастом накопление кетопрофена у лиц пожилого возраста, обусловленное сниженным клиренсом, также было отмечено Skeith и соавторами [35]. В связи с этим в Краткой характеристике лекарственного препарата рекомендуется с осторожностью применять данный препарат у лиц пожилого возраста.

Почечная и, в дальнейшем, печеночная недостаточность приводит к стереоселективному снижению почечного клиренса ацилглюкуроновых конъюгатов кетопрофена (CLrconj), и это, по-видимому, является этапом, на котором происходит ограничение скорости клиренса кетопрофена, что приводит к увеличению концентрации лекарственного вещества в плазме крови [37], [35], [36]. В связи с этим лизиновая соль кетопрофена противопоказана к применению у пациентов с тяжелой почечной или печеночной недостаточностью.

#### Исследование биоэквивалентности

Было проведено открытое перекрестное исследование однократного приема натощак с целью определения сравнительной фармакокинетики лизиновой соли кетопрофена в форме гранул, растворимых в ротовой полости (40 мг с приемом без запивания водой) в сравнении с лизиновой солью кетопрофена в форме гранул для приготовления раствора для перорального приема (80 мг в пакетике из двух частей, половина пакетика, препарат Oki<sup>®</sup> 80 мг) после перорального приема у здоровых добровольцев [9].

Семьдесят один участник исследования (34 женского пола и 37 мужского) получили не менее одной дозы исследуемого препарата (ОКИТАСК<sup>®</sup> в дозе 40 мг в форме гранул без воды и ОКі<sup>®</sup> 80 мг в форме гранул для приготовления раствора для перорального приема, половина пакетика с водой (240 мл)). После первого приема исследуемого препарата один участник исследования отозвал согласие на участие в этом исследовании по личным причинам, но ни один из участников не был исключен из исследования Исследователем в связи с приемом запрещенных сопутствующих препаратов в ходе периода отмывки. Таким образом, при анализе фармакокинетики 69 участников

КОНФИДЕНЦИАЛЬНО Страница 35 из 76

исследования были пригодны для изучения данных (популяция исследования: 34 женщины и 35 мужчин (средний возраст  $\pm$  стандартное отклонение  $= 33,6 \pm 9,0$ )).

Здоровые добровольцы были в случайном порядке распределены для приема:

**Тестируемое вещество** (T) = ОКИТАСК<sup>®</sup> в гранулах по 40 мг (соответствует 25 мг кетопрофена): содержимое всего пакетика исследуемого препарата было помещено на язык и растворилось во рту в течение приблизительно 3 минут без приема воды. Непосредственно перед помещением гранул на язык ротовая полость была увлажнена при употреблении 20 мл минеральной воды. После этого прием жидкости не был разрешен в течение 2 часов.

Референсный препарат (R) = OKi® в гранулах по 80 мг в пакетиках из двух частей для приготовления раствора: половина пакетика = 40 мг лизиновой соли кетопрофена (соответствует 25 мг кетопрофена): содержимое половины пакетика референсной лекарственной формы было растворено в 190 мл минеральной воды. Участник исследования сразу же выпивал весь раствор целиком. После этого проводилось ополаскивание стакана 50 мл минеральной воды и эта жидкость тоже немедленно выпивалась. После этого прием жидкости не был разрешен в течение 2 часов.

Прием препарата проводился однократно утром натощак, при отсутствии приема пищи в течение всей ночи, а через 4 часа после приема препарата участники исследования получали стандартный завтрак.

В каждом из периодов исследования проводился сбор образцов крови у добровольцев для оценки уровней кетопрофена в следующие моменты времени: перед приемом препарата (0), через 0,08 (5 минут), 0,25 минут, 0,5 минут, 0,75 минут, 1,0 час, 1,5 часа, 2,0 часа, 3,0 часа, 4,0 часа, 5,0 часов, 6,0 часов и 8,0 часов после приема препарата.

Определение кетопрофена в плазме крови проводилось с помощью валидированного метода высокоэффективной жидкостной хроматографии ВЭЖХ-У/Ф.

В соответствии с Европейскими руководствами были определены следующие параметры фармакокинетики:  $AUC_{0-\tau}$ ,  $AUC_{0-\infty}$  и  $C_{max}$ , которые были проанализированы с применением вариационного анализа. Перед анализом данные были трансформированы с применением логарифмической трансформации неперов. Статистический метод тестирования биоэквивалентности (БЭ) был основан на 90% доверительных интервалах (ДИ) для соотношения средних популяционных (тестируемое вещество/ референсное вещество) для учитываемых параметров фармакокинетики. Этот метод эквивалентен соответствующим двум односторонним процедурам теста при нулевой гипотезе о биоэквивалентности при 5% уровне значимости (были применены два односторонних t-теста Schuirmann). Критерием приемлемости для биоэквивалентности было то, что 90% доверительные интервалы соотношения средних геометрических были в диапазоне 80,00-125,00.

В качестве фиксированных эффектов статистический анализ учитывал терапию, период, последовательность и субъекта внутри последовательности.  $T_{max}$  было проанализировано с применением непараметрического теста Friedman.

Выявленные профили фармакокинетики тестируемого препарата (ОКИТАСК в гранулах по 40 мг и  $\mathrm{Oki}^{\$}$  в гранулах по 80 мг для приготовления раствора, половина пакетика) показали, что обе лекарственные формы быстро всасываются с  $\mathrm{T}_{\mathrm{max}}$  приблизительно 0,5 часа и обе лекарственные формы приводят к одинаковым уровням системной экспозиции кетопрофена.

КОНФИДЕНЦИАЛЬНО Страница 36 из 76

С учетом 90% доверительного интервала соотношения (тестируемый препарат/ референсный препарат) средних геометрических все значения для каждого из параметров фармакокинетики были в пределах приемлемого диапазона (80-125%) биоэквивалентности. Таким образом, можно сделать выводы, что препарат ОКИТАСК в гранулах по 40 мг при приеме без воды является биоэквивалентным препарату  $OKi^{\otimes}$  в гранулах по 80 мг для приготовления раствора (половина пакетика: 40 мг), прием которого осуществляется с 240 мл воды, как в отношении скорости ( $C_{max}$ ), так и объема (AUC) всасывания кетопрофена.

Сводные данные, полученные в ходе оценки фармакокинетики и биоэквивалентности в исследовании KSL0112 представлены ниже.

Таблица 2. Сводные данные по фармакокинетике и 90% доверительные интервалы, полученные в ходе исследования KSL0112

| mirepawin, north termine a node neoregopullin 11820112 | | | | | |
|---|---|---|---|---|---|
| Терапия | С <sub>тах</sub><br>(мкг/мл) | Т <sub>тах</sub> (ч) | AUC <sub>0-t</sub><br>(мкг•ч/мл) | AUC <sub>0-∞</sub><br>(мкг•ч/мл) | t <sub>1/2</sub> (ч) |
| Т | 2,77 ± 0,82 | 0,46 ± 0,19 | 4,82 ± 1,02 | 4,93 ± 1,07 | $1.66 \pm 0.23$ |
| R | 3,16 ± 0,75 | $0.30 \pm 0.13$ | $4,62 \pm 1,08$ | 4,77 ± 1,13 | $\begin{array}{c} 1.87 \pm \\ 0.31 \end{array}$ |
| Статисти | ческий анализ | | | | |
| 90% доверительный интервал соотношения средних геометрических | | | | | |
| | | AUC <sub>0-t</sub> | 104,71 | 102,63 | 106,84 |
| Терапия Т в сравнении с R | | AUC <sub>0-∞</sub> | 104,61 | 102,46 | 106,80 |
| | | $\mathbf{C}_{max}$ | 86,28 | 82,24 | 90,52 |

На графике ниже показано, что профили изменения концентраций кетопрофена в плазме крови с течением времени при двух вариантах терапии, изучавшихся в ходе исследования KSL0112, виртуально накладываются друг на друга.

КОНФИДЕНЦИАЛЬНО Страница 37 из 76



Рисунок 1. Профили средних концентраций кетопрофена в плазме крови (мкг/мл) с течением времени после приема 40 мг лизиновой соли кетопрофена в форме гранул, растворимых в полости рта (Т) (● непрерывная линия), и 40 мг лизиновой соли кетопрофена в форме гранул для приготовления раствора для перорального приема (R) (□ пунктирная линия), показанные на полулогарифмической шкале

По оси Х: время (ч)

По оси Ү: [Кетопрофен] (мкг/мл)

Вторичной конечной точкой данного исследования являлась оценка безопасности. Случаев смерти или тяжелых нежелательных явлений, возникших на фоне проводимой терапии, или серьезных нежелательных явлений в ходе периода исследования не было. Переносимость исследуемого и референсного веществ у участников исследования была хорошей. У 10 участников исследования из 71 (14%) возникло по одному нежелательному явлению (НЯ). В частности, у 8 участников исследования (11,3%) возникло по одному нежелательному явлению после приема тестируемого препарата, а у 2 участников исследования – после приема референсного препарата. Исследователь расценил 5 зарегистрированных нежелательных явлений из 10 как связанные с исследуемой терапией. В частности, у 4 участников исследования (5,6%) возникло одно нежелательное явление после приема тестируемого препарата, а у одного участника исследования (1,4%) – после приема референсного препарата. Наиболее часто регистрируемыми нежелательными явлениями был головная боль, отмеченная у 3 участников исследования (4,2%), получавших исследуемую терапию. Другие зарегистрированные нежелательные явления отмечались не более чем у оного участника исследования каждое. Клинически значимых эффектов кетопрофена в отношении показателей функций жизненно-важных органов, массы тела, данных ЭКГ или параметров стандартных лабораторных тестов не отмечалось.

Таким образом, можно сделать выводы, что препарат ОКИТАСК $^{\text{®}}$  в гранулах по 40 мг при приеме без воды является биоэквивалентным препарату ОКі $^{\text{®}}$  в гранулах по 80 мг для приготовления раствора (половина пакетика: 40 мг), прием которого осуществлялся с 240

КОНФИДЕНЦИАЛЬНО Страница 38 из 76

мл воды, как в отношении скорости ( $C_{max}$ ), так и объема (AUC) системного всасывания кетопрофена у здоровых добровольцев мужского и женского пола.

#### Беременность и грудное вскармливание

Использование нестероидных противовоспалительных препаратов может привести к снижению фертильности у женщин и не рекомендуется женщинам, планирующим беременность, как и применение любых других препаратов, ингибирующих циклооксигеназу/ синтез простагландина. Применение нестероидных противовоспалительных препаратов должно быть прекращено у женщин с нарушениями фертильности или у женщин, которые обследуются по поводу бесплодия.

Нестероидные противовоспалительные препараты могут проникать через плаценту; воздействие нестероидных противовоспалительных препаратов в ранние сроки беременности повышает риск невынашивания и пороков развития у плода, который увеличивается вместе с увеличением дозы и длительности терапии. Ингибирование синтеза простагландина [39], [40], [41], [42] под действием любых ингибиторов может повлиять на нерожденного ребенка, поскольку воздействие таких препаратов в течение третьего триместра беременности повышает частоту преждевременного закрытия артериального протока в матке, нарушений функции почек, прогрессировать до почечной недостаточности с олигогидроамнионом, замедлением гестации, нарушением координации родовой деятельности и поздним родоразрешением [43], [44], [45], [46]. Таким образом, как и для всех нестероидных противовоспалительных препаратов и в соответствии с руководящим документом ЕМЕА/12148/04, применение лизиновой соли кетопрофена в гранулах по 40 мг в третьем триместре беременности противопоказано; применение лизиновой соли кетопрофена в гранулах по 40 мг не рекомендовано в течение первых двух триместров беременности; в этом периоде рекомендуется применять лизиновую соль кетопрофена только если это крайне необходимо.

Кетопрофен после приема может быть обнаружен в женском молоке. В ходе трехдневного исследования в послеродовом периоде кормящие матери получали кетопрофен в дозе 100 мг внутривенно болюсно каждые 12 часов. Между третьим и четвертым введениями были взяты образцы молока. Анализ этих образцов и экстраполяция результатов показали, что младенец, получающий грудное вскармливание, может получить среднюю дозу  $8,5\pm5,5$  мкг/кг/сут, максимально  $13,6\pm7,6$  мкг/кг/сут. Относительная доза для младенца составляет  $0,31\pm0,17\%$  от дозы для матери, откорректированной по массе тела. В ходе этого исследования относительная доза кетопрофена для младенца была меньше, чем для другого изучавшегося препарата, налбуфина  $(0,59\pm0,27\%)$ .

Авторы пришли к выводу, что грудное вскармливание в случаях, когда матери получают кетопрофен для лечения боли в послеродовом периоде, допустимо. Тем не менее, применение лизиновой соли кетопрофена в гранулах по 40 мг противопоказано, что отмечено в Краткой характеристике лекарственного препарата.

#### Объем применения лизиновой соли кетопрофена у пациентов

Препараты лизиновой соли кетопрофена зарегистрированы и распространяются компанией Dompé farmaceutici S.p.A. под четырьмя разными торговыми наименованиями: Artrosilene (Артрозилен),  $Oki^{\text{®}}$  ( $OKU^{\text{®}}$ ),  $OKi^{\text{®}}$  Infiammazione e Dolore и  $OKITASK^{\text{®}}$  ( $OKUTACK^{\text{®}}$ ).

Компания Dompé farmaceutici S.p.A. получила первое регистрационное удостоверение на препараты, содержащие лизиновую соль кетопрофена, под наименованием **Artrosilene** 

КОНФИДЕНЦИАЛЬНО Страница 39 из 76

(Артрозилен) в Италии 13 июня 1979 года для препарата в форме свечей. В настоящее время Артрозилен зарегистрирован и продается в разных странах, в виде разных лекарственных форм и в разных дозах, с разными способами системного применения:

- Перорально (твердые капсулы с замедленным высвобождением по 320 мг),
- Парентерально (раствор для инъекций 160 мг/ 2 мл)
- Ректально (свечи по 160 мг)

Указанные выше варианты лекарственного препарата в дальнейшем были зарегистрированы и начали продаваться компанией "Dompé farmaceutici S.p.A.", являющейся собственником регистрационного удостоверения, в Албании, Косово и России под тем же торговым наименованием.

Кроме того, компания "Dompé farmaceutici S.p.A." является собственником регистрационных удостоверений лекарственных форм, зарегистрированных под торговым наименованием "Артрозилен", предназначенных для местного нанесения на кожу (гель для кожи 5 г / 100 г и пена 15 г/ 100 мл), которые распространяются как в Италии, так и за ее пределами.

Лизиновая соль кетопрофена под наименованием OKi® (OKU®) была зарегистрирована компанией "Dompé farmaceutici S.p.A." (ранее "Dompé S.p.A.") в Италии 15 ноября 1994 года и в дальнейшем была зарегистрирована и начала продаваться в нескольких странах мира под разными торговыми наименованиями. Препараты лизиновой соли кетопрофена под наименованием "OKi®" или под другими торговыми марками зарегистрированы в виде ряда лекарственных форм и доз с разными способами применения:

- Для перорального приема: гранулы по  $80~\rm Mr$  для приготовления раствора, капли с концентрацией  $80~\rm mr/mn$ 
  - Для парентерального введения: раствор для инъекций 160 мг/ 2 мл;
  - Для ректального введения: свечи по 160, 30 и 60 мг.

Под наименованием "OKi® Infiammazione е Dolore" зарегистрированы две лекарственных формы для местного применения (1,6% раствор для ополаскивания полости рта и 0,16% спрей для орошения слизистых оболочек полости рта), которые продаются в Италии. Ополаскиватель для полости рта зарегистрирован также в Албании, Косово, Мальте, России (собственник регистрационного удостоверения компания «Dompé») и в Греции и Южной Корее (собственниками регистрационных удостоверений являются бизнес-партнеры компании).

Препарат ОКІТАЅК<sup>®</sup> (ОКИТАСК<sup>®</sup>) в гранулах по 40 мг впервые был зарегистрирован в Италии 12 сентября 2012 года; в дальнейшем, почти через три года, этот же продукт был зарегистрирован в Албании и в Косово. Таблетки по 40 мг, покрытые пленочной оболочкой, были зарегистрированы в Италии в феврале 2017 года.

Как сообщается в Дополнении к клиническому обзору препарата ОКИТАСК® (последние данные получены 16 сентября 2016 года), поданному в Итальянское регуляторное агентство в декабре 2016 года вместе с запросом на обновление регистрационного удостоверения, с момента начала продаж (сентябрь 2012 года) по 31 августа 2016 года компанией «Dompé» было продано 13067368 упаковок препарата ОКИТАСК® в форме гранул в странах, где этот препарат зарегистрирован. На основе имеющихся данных по продажам и одобренных показаний к применению предполагается, что одна упаковка препарата используется одним пациентом в связи с чем количество

КОНФИДЕНЦИАЛЬНО Страница 40 из 76

проданных упаковок соответствует количеству пациентов, получивших препарат. Оценочное совокупное количество пациентов, получивших препарат, на 31 августа 2016 года превышало 13 миллионов.

#### Нежелательные явления

Для всех нестероидных противовоспалительных препаратов существуют давно и хорошо известные проблемы безопасности в отношении желудочно-кишечного тракта и почек (NICE 2015). В 2006 году Европейское агентство по лекарственным препаратам (ЕМА 2006) заявило, что общий баланс риска и пользы для неселективных нестероидных противовоспалительных препаратов остается благоприятным при их применении в соответствии с инструкцией, в частности, на основе общего профиля безопасности соответствующих нестероидных противовоспалительных препаратов неизбирательного действия и с учетом индивидуальных факторов риска у конкретных пациентов (например, заболеваний желудочно-кишечного тракта, сердечно-сосудистой системы и почек).

В стандартных медицинских руководствах, таких как Martindale (2015) [32] и Dollery (1999) [47] отмечается, что острый интерстициальный нефрит связан с применением многих разных нестероидных противовоспалительных препаратов, включая и кетопрофен. Нарушения со стороны желудочно-кишечного тракта при применении кетопрофена описаны как частые и сравнимые по частоте с нарушениями, возникающими при применении других производных пропионовой кислоты, таких как напроксен. Неизбирательное ингибирование синтеза простагландина под действием нестероидных противовоспалительных препаратов, в том числе простагландинов, действующих как гастропротекторы, является главной причиной нежелательных явлений со стороны желудочно-кишечного тракта [47].

Наиболее часто отмечавшиеся нежелательные явления, возникавшие при применении лизиновой соли кетопрофена в ходе описанных выше исследований препаратов лизиновой соли кетопрофена (ОКИТАСК® и ОКИ® 80 мг), поражали желудочно-кишечный тракт. Обычно они характеризовались кратковременными эпизодами изжоги и боли легкой приеме натощак (исследования безопасным профилем даже при биоэквивалентности). Причинная взаимосвязь с препаратом  $\operatorname{OKi}^{\mathbb{R}}$  в ранулах по 80 мг для приготовления раствора, дозировка которого в 2 раза выше лизиновой соли кетопрофена в гранулах по 40 мг, была расценена как возможная для всех зарегистрированных нежелательных явлений с вовлечением желудочно-кишечного тракта. Этот опыт отражен в опубликованных данных клинических исследований, в которых нежелательные явления со стороны желудочно-кишечного тракта являются наиболее часто отмечаемыми после перорального приема кетопрофена. Нежелательные явления со стороны желудочнокишечного тракта, возникающие при применении нестероидных противовоспалительных препаратов, а, следовательно, и при применении кетопрофена, могут проявляться следующим образом: тошнота, рвота, диарея, вздутие живота, запор, диспепсия, боль в животе, мелена, рвота кровью, язвенный стоматит, обострение болезни Крона и гастрит.

Для того чтобы снизить риск нежелательных явлений со стороны желудочнокишечного тракта, для производства лизиновой соли кетопрофена в форме гранул была выбрана самая низкая эффективная доза лизиновой соли кетопрофена, 40 мг, более того, в предлагаемую Краткую характеристику лизиновой соли кетопрофена в форме гранул по 40 мг включены следующие предупреждения и меры предосторожности:

Данный лекарственный препарат запрещается применять в следующих случаях:

- У лиц с активной пептической язвой или с наличием в анамнезе любых желудочнокишечных кровотечений, язв или перфораций;

КОНФИДЕНЦИАЛЬНО Страница 41 из 76

- У лиц с язвой желудка или двенадцатиперстной кишки, хронической диспепсией и гастритом. При применении лекарственного препарата следует учитывать приведенные далее меры предосторожности;
- Следует избегать применения лизиновой соли кетопрофена в гранулах по 40 мг одновременно с другими нестероидными противовоспалительными препаратами, в том числе с селективными ингибиторами циклооксигеназы-2.
- нежелательные эффекты могут быть сведены к минимуму путем применения минимальной эффективной дозы в течение самого короткого времени, необходимого для контроля симптомов.
- Пациентам, которые в то же самое время получают лекарственные препараты, которые могут повысить риск образования язв или возникновения кровотечений, таких как кортикостероиды для перорального приема, антикоагулянты, такие как варфарин, избирательные ингибиторы обратного захвата серотонина или антитромбоцитарные препараты, такие как ацетилсалициловая кислота.

# Данные по безопасности, полученные в ходе постмаркетингового применения

Он был впервые одобрен для клинического применения во Франции и в Великобритании в 1973 году. В настоящее время он применяется во всем мире в виде разных лекарственных форм, таких как капсулы, растворы для инъекций, свечи, а также гели для местного нанесения.

Совокупные данные по препарату ОКИТАСК<sup>®</sup> в гранулах взяты из дополнения к клиническому обзору, поданному в Итальянское регуляторное агентство для обновления регистрационных данных на препарат. В совокупности по сентябрь 2016 года было выпущено 59 отчетов по нежелательным реакциям у отдельных лиц, включавших 119 случаев нежелательных лекарственных реакций, зарегистрированных у лиц, получавших лизиновую соль кетопрофена в гранулах по 40 мг, в рамках стандартной клинической практики. Среди зарегистрированных случаев 22 отчета по нежелательным реакциям у отдельных лиц (37,3%) были расценены как случаи с хотя бы одной серьезной нежелательной лекарственной реакцией: в совокупности компания получила отчеты по 53 серьезным нежелательным лекарственным реакциям (44,5%) и по 66 нежелательным лекарственным реакциям (55,5%). Все случаи были спонтанно зарегистрированы в Италии и информация о них получена как от регуляторных органов (посредством Итальянской национальной сети фармакологического надзора) или от работников здравоохранения/ пациентов.

С учетом количества лиц, получавших препарат, частота нежелательных лекарственных реакций (серьезных и не являющихся серьезными) расценивается как очень редкая (<1/10000).

Классами систем и органов, которые наиболее часто вовлекаются в нежелательные реакции, были:

- "Поражения кожи и подкожной клетчатки": в этом классе систем и органов было зарегистрировано 35 нежелательных лекарственных реакций, 15 из которых были серьезными и ожидаемыми (без неожиданных нежелательных лекарственных реакций), а 20 не были серьезными.
- "Нарушения со стороны желудочно-кишечного тракта": в этом классе систем и органов было зарегистрировано 25 нежелательных лекарственных реакций, 7 из которых были серьезными и ожидаемыми (неожиданных нежелательных лекарственных реакций не было), а 18 не были серьезными.

КОНФИДЕНЦИАЛЬНО Страница 42 из 76

- "Нарушения со стороны дыхательной системы, органов грудной клетки и средостения": в этом классе систем и органов было зарегистрировано 18 нежелательных лекарственных реакций, 13 из которых были серьезными и ожидаемыми (11 ожидаемых и 2 неожиданных), а 5 не были серьезными.

Большинство зарегистрированных нежелательных лекарственных реакций представляли собой известные аллергические реакции, включавшие проявления со стороны кожи и/или симптомы нарушений со стороны дыхательной системы или желудочно-кишечного тракта, что описано в текущей версии Краткой характеристики лекарственного препарата.

В целом, какого-либо специфического риска для этого лекарственного препарата выявлено не было: случаев, завершившихся смертью у пациентов, получавших препарат, зарегистрировано не было. Данных о случаях межлекарственного взаимодействия, передозировки, применения не по назначению или применения не по показаниям компания не получала. Отчетов по применению препарата во время беременности или грудного вскармливания компанией не получено. Были зарегистрированы один случай намеренного злоупотребления препаратом и один случай его применения по ошибке (непреднамеренно), как описано выше: в обоих случаях остаточные явления не упоминались.

#### Выводы по безопасности

В ходе клинических исследований было установлено, что лизиновая соль кетопрофена и другие препараты кетопрофена являются эффективным и хорошо переносятся при применении по показаниям, предложенным для лизиновой соли кетопрофена в гранулах по 40 мг. Профиль безопасности кетопрофена (и его лизиновой соли) хорошо изучен в ходе клинических исследований и в течение 40 лет использования в качестве рецептурного, а затем и безрецептурного препарата. Серьезные нежелательные явления при кратковременном пероральном приеме кетопрофена в дозе 25 мг (эквивалент лизиновой соли кетопрофена в дозе 40 мг) отмечаются редко. Данные по нежелательным реакциям, представленные для лизиновой соли кетопрофена в гранулах по 40 мг (ОКИТАСК®), показывают, что наиболее часто регистрируемыми нежелательные лекарственные реакции поражают кожу и подкожную клетчатку, при этом наиболее часто регистрируемой нежелательной лекарственной реакцией является крапивница.

Наиболее часто регистрируемые нежелательные явления, отмеченные кратковременном применении кетопрофена в низкой дозе (25 мг), возникали со стороны желудочно-кишечного тракта и хорошо изучены, легко диагностируются, легкой или умеренной степени тяжести и разрешаются при прекращении терапии. Тем не менее, имеющиеся данные указывают на то, что кратковременный пероральный прием лизиновой соли кетопрофена (40 мг) вызывает меньше нежелательных явлений со чем прием стороны желудочно-кишечного тракта, других нестероидных противовоспалительных препаратов, что считается следствием оптимизированной скорости всасывания. На основании исследований установлено, что образование соли кетопрофена с лизином дает дополнительную степень защиты слизистых оболочек желудка. Прием лизиновой соли кетопрофена с пищей для уменьшения частоты нежелательных явлений со стороны желудочно-кишечного тракта при кратковременном применении лизиновой соли кетопрофена не является обязательным.

Этот клинический опыт в достаточной мере отражен в соответствующей Краткой характеристике лекарственного и в инструкции по применению лизиновой соли кетопрофена в гранулах по 40 мг. Имеющиеся данные по безопасности лизиновой соли кетопрофена и других лекарственных форм кетопрофена подтверждают возможность

КОНФИДЕНЦИАЛЬНО Страница 43 из 76

кратковременного перорального приема лизиновой соли кетопрофена в дозе 40 мг до 3 раз в сутки у взрослых лиц в возрасте старше 18 лет.

Таким образом, симптоматическая польза от применения лизиновой соли кетопрофена в гранулах по 40 мг у взрослых лиц значительно превосходит известные риски.

#### 3.5. Обоснование выбора дозы и соотношение риска и пользы

Доза лизиновой соли кетопрофена в гранулах, которую предполагается использовать в этом исследовании, составляет 40 мг однократно (эквивалентно 25 мг кетопрофена). Эта доза составляет одну треть от суточной дозы, разрешенной в Италии (для взрослых лиц и подростков в возрасте старше 15 лет: 1 пакетик в качестве разовой дозы или повторно 2 или 3 раза в день при более интенсивной боли) и в европейских странах (т.е., до 3 раз в сутки у взрослых лиц в возрасте старше 18 лет), 1 пакетик в качестве разовой дозы или повторно 2 или 3 раза в день по мере необходимости.

Лизиновая соль кетопрофена широко применяется в клинической практике в течение более 35 лет и, таким образом, имеется обширный опыт применения этого препарата.

С учетом профиля безопасности уже продаваемого препарата ОКИТАСК $^{\text{®}}$  в гранулах по 40 мг, особенных рисков для безопасности не ожидается.

Препарат ОКИТАСК<sup>®</sup> в гранулах поставляется в форме отдельных пакетиков и дает легкую возможность применения данной лекарственной формы, которую удобно проглатывать без воды как обычным людям, так и лицам, которые обычно испытывают затруднения при проглатывании таблеток или капсул. В инструкции по применению лизиновой соли кетопрофена в гранулах по 40 мг представлены необходимые предупреждения, что обеспечивает правильный и безопасный самостоятельный прием препарата.

С учетом того, что планируемая доза лизиновой соли кетопрофена составляет 40 мг однократно, каких-либо проблем с безопасностью участников исследования не ожидается.

Использование плацебо в этом исследовании является приемлемым и этически оправдано, поскольку 1) нет риска для безопасности и благополучия пациента и 2) в случаях, когда исследуемый препарат или плацебо не позволят достичь достаточного уровня снижения интенсивности боли, пациентам будет предоставлена резервная терапия. Участникам исследования будет предложено воздерживаться от приема резервных препаратов в течение первого часа после приема исследуемого препарата. Парацетамол в дозе 500-1000 мг был выбран в качестве резервной терапии, поскольку от относится к другой фармацевтической группе обезболивающих препаратов, что позволит избежать взаимодействия между препаратами. Если прием парацетамола в дозе 500-1000 мг не даст нужного эффекта, пациентам будет разрешено принимать парацетамол в дозе 500-1000 мг каждые 6-8 часов; интервал между приемами не должен быть меньше 4 часов; максимальная суточная доза составляет 4000 мг.

Это исследование считается интервенционным исследованием с низким интервенционным риском, поскольку оно проводится с уже зарегистрированным лекарственным препаратом, который будет исследован в соответствии с его регистрационным удостоверением, выданным в некоторых странах Европы.

#### 4. ИССЛЕДУЕМАЯ ПОПУЛЯЦИЯ

КОНФИДЕНЦИАЛЬНО Страница 44 из 76

#### 4.1. Исследуемая популяция

В скрининг данного исследования планируется включить до 100 мужчин и женщин, у которых запланировано удаление моляра. 70 пациентов, пригодных для участия в исследовании, будут рандомизированы в одну из групп терапии в соотношении 1:1:

Группа 1. Терапия препаратом ОКИТАСК $^{\otimes}$  в дозе 40 мг – 35 пациентов

Группа 2. Терапия плацебо – 35 пациентов.

#### 4.2. Критерии включения

Пациенты, пригодные для участия в данном исследовании, должны соответствовать следующим критериям включения:

- 1. Подписанная форма информированного согласия
- 2. Мужчины и женщины в возрасте от 18 до 65 лет (включительно);
- 3. Лица, которым было выполнено удаление не ретинированного моляра в течение 3 часов до рандомизации;
- 4. Лица с хорошим состояние здоровья (понятие базируется на основе критериев безопасного применения амбулаторного обезболивания);
- 5. Лица, которым в течение 3 часов после экстракции зуба требуется прием препарата для уменьшения боли (BAШ ≥30 мм);
- 6. Лица, которые согласны оставаться под наблюдением в течение 9 часов после удаления зуба;
- 7. Лица, способные заполнить 100-миллиметровую визуально-аналоговую шкалу и категориальную шкалу в течение периода наблюдения (около 9 часов);
- 8. Полное понимание: способность понимать суть и цели исследования, включая возможные риски и побочные эффекты; способность сотрудничать с Исследователем и выполнять все требования исследования;
- 9. Контрацепция (для женщин): женщины, способные к деторождению, должны использовать в ходе исследования как минимум один надежный метод контрацепции из числа перечисленных ниже:
  - а. гормональные пероральные, имплантируемые, трансдермальные или инъекционные контрацептивы;
  - b. негормональное внутриматочное устройство (ВМУ), или женский презерватив со спермицидом, или контрацептивная губка со спермицидом, или диафрагма со спермицидом, или шеечный колпачок со спермицидом;
  - с. мужчина половой партнер женщины долен быть согласен на использование мужского презерватива со спермицидом;
  - d. половой партнер, которому была выполнена стерилизация.

# 4.3. Критерии невключения

Пациенты не будут включены в исследование, если они соответствуют хотя бы одному из критериев невключения, из числа перечисленных далее:

1. Лица, которым были выполнены: удаление ретинированного и дистопированного зуба, зубосохраняющие операции, апикальное перемещение лоскута/ вестибулопластика со свободным трансплантатом десны, взятым из твердого неба;

КОНФИДЕНЦИАЛЬНО Страница 45 из 76
- 2. Лица, которым в течение одной процедуры было удалено больше одного зуба;
- 3. Лица, которым одновременно с удалением зуба была выполнена установка импланта;
- 4. Аллергия: известная или предполагаемая гиперчувствительность к активным компонентам (кетопрофен и парацетамол, применяемый в качестве резервного препарата) и/или вспомогательным веществам в составе препарата; наличие в анамнезе гиперчувствительности к лекарственным препаратам (в особенности, к нестероидным противовоспалительным препаратом) или аллергических реакций в целом, которые, по мнению Исследователя, могут повлиять на результаты исследования;
- 5. Заболевания: наличие в анамнезе значимых заболеваний почек, печени, сердечнососудистой системы, дыхательной системы (в том числе бронхиальной астмы), кожи, системы крови, органов внутренней секреции, желудочно-кишечного тракта и мочевыводящих путей и половой системы, либо нервной системы или аутоиммунных заболеваний, которые могут повлиять на цели исследования;
- 6. Лекарственные препараты: прием нестероидных противовоспалительных препаратов и других обезболивающих препаратов (в особенности, кетопрофена, парацетамола и ацетилсалициловой кислоты (АСК)), антигистаминных препаратов, седативных препаратов, в том числе растительных препаратов и биологически активных пищевых добавок в течение 48 часов до удаления зуба;
- 7. Исследования других лекарственных препаратов: участие в исследовании любого другого препарата в течение 3 месяцев до начала скрининга (включая последнюю процедуру исследования);
- 8. Алкогольная и наркотическая зависимость в анамнезе;
- 9. Положительные результаты теста на беременность у женщин, способных к деторождению (включая женщин, находящихся в постменопаузе менее 2 лет).

#### 4.4. Критерии невключения

Допускается однократный повторный скрининг пациента, если процедура удаления зуба была отложена или отменена за пределами окна День -4 — День 1. В этом случае пациент должен подписать новую форму информированного согласия, ему присваивается новый номер, и все процедуры скрининга должны быт проведены повторно.

Запрещается повторный скрининг пациентов для второго удаления моляра или участие в исследовании два раза.

КОНФИДЕНЦИАЛЬНО Страница 46 из 76

# 5. ИССЛЕДУЕМЫЙ ПРЕПАРАТ

# 5.1. Описание

| ОКИТАСК <sup>®</sup> гранулы по 40 мг |
|---|
| Кетопрофена лизиновая соль |
| Кетопрофен: 2-(3-бензоилфенил)-пропионовая кислота; |
| $C_{16}H_{14}O_3$ ; номер в соответствии с каталогом Химической реферативной службы (CAS) 56105-81-8; молекулярная масса 254,29 |
| Лизин: 2,6-диаминогексаноевая кислота; |
| $C_6H_{14}N_2O_2$ ; номер в соответствии с каталогом Химической реферативной службы (CAS) 70-54-2; молекулярная масса 146,19 |
| Нестероидный противовоспалительный препарат, производное пропионовой кислоты. |
| Код АТХ: М01АЕ03 |
| Гранулы для перорального приема. |
| Состав: лизиновая соль кетопрофена, повидон К-25, кремний (коллоидный безводный), гипромеллоза, основной бутилированный сополимер метилакрилата (Eudragit EPO), лаурилсульфат натрия, стеариновая кислота, магния стеарат, ароматизатор лайма, ароматизатор лимона, ароматизатор Frescofort, аспартам, маннитол, ксилитол, тальк |
| Гранулы в пакетике. |
| Пакетик: непрозрачный, изготовленный из полиэтилена/ алюминия/ полиэтилентетрафатлата, содержащий 700 мг гранул (40 мг лизиновой соли кетопрофена) |
| 40 мг – 1 пакетик |
| Однократный прием |
| Хранить при температуре не выше + 25°C |
| Хранить в месте, недоступном для детей |
| Компания "Dompé farmaceutici S.p.A." (Италия) |
| http://www.biocentury.com/companies/dompe_farmaceutici_spa |
| Компания "Monteresearch" (Италия) |
| Компания "Dompé farmaceutici S.p.A." (Италия) |

| Препарат сравнения: | Плацебо, имитирующее препарат ОКИТАСК <sup>®</sup> в гранулах по 40 мг |
|---|---|
| Суточная доза | 0 мг – 1 пакетик |
| Режим терапии: | Однократный прием |
| Условия хранения: | Хранить при температуре не выше + 25°C<br>Хранить в месте недоступном для детей |
| Производитель: | Компания "Monteresearch" (Италия) |
| Контроль и выпуск<br>партии | Компания Dompé farmaceutici S.p.A. <a href="http://www.biocentury.com/companies/dompe_farmaceutici_spa">http://www.biocentury.com/companies/dompe_farmaceutici_spa</a> (Италия) |

КОНФИДЕНЦИАЛЬНО Страница 47 из 76

# 5.2. Режим терапии

Пациенты примут препарат ОКИТАСК<sup>®</sup> в гранулах по 40 мг или плацебо однократно в течение 3 часов после удаления моляра (интенсивность боли по визуально-аналоговой шкале ≥30 мм). Каждый пациент получит один пакетик, содержащий 40 мг лизиновой соли кетопрофена (эквивалент 25 мг кетопрофена) или плацебо. Все содержимое пакетика пациент должен поместить себе на язык и проглотить. Исследуемый препарат растворяется в слюне, поэтому прием воды может не потребоваться.

# 5.3. Рандомизация и закрытие кодов терапии

Это двойное слепое плацебо-контролируемое исследование. Пациенты будут распределены с помощью системы IWRS в соотношении 1:1 в одну из двух групп:

Группа 1. Терапия препаратом ОКИТАСК $^{\text{®}}$  в дозе 40 мг – 35 пациентов

Группа 2. Терапия плацебо – 35 пациентов.

Рандомизация будет проведена после удаления зуба при подтверждении критериев включения/ невключения (ВАШ ≥30 мм).

Терапия в двойном слепом режиме обеспечивается плацебо, которое идентично препарату ОКИТАСК<sup>®</sup> в гранулах по 40 мг. Препарат будет маркирован таким образом, чтобы это исключало раскрытие кода терапии. Система IWRS назначит номер упаковки исследуемого препарата, содержимое которой должен принять пациент. Руководство по рандомизации и работе с IWRS будет представлено Исследователям перед началом исследования.

# 5.4. Процедура раскрытия кодов терапии

Код каждого конкретного пациента моет быть раскрыт при неотложной медицинской ситуации, если знание того, какой препарат был назначен этому пациенту может повлиять на его лечение. назначение терапии спасения не требует раскрытия кода.

Раскрытие кода терапии пациента может быть проведено через IWRS. Причина раскрытия кода терапии должна быть указана в первичной документации. По возможности перед раскрытием кода терапии необходимо связаться с медицинским монитором; если это невозможно, то медицинский монитор должен быть уведомлен о раскрытии кода терапии в течение 24 часов после того как оно произошло.

#### 5.5. Комплаентность в отношении исследуемой терапии

Пациенты должны однократно принять исследуемый препарат под контролем Исследователя. Специфической оценки комплаентности в ходе этого исследования не предполагается.

# 5.6. Упаковка и маркировка препарата

Исследуемый препарат будет предоставляться Спонсором. Упаковка и маркировка препарата будет проводиться в соответствии с действующим российским законодательством и действующими требованиями.

Маркировка коробки, в которой содержится пакетик с исследуемым препаратом, показана на Рисунке 2.

#### Рисунок 2 Маркировка коробки, содержащей пакетик с препаратом

Маркировка пакетика показана на Рисунке 3

КОНФИДЕНЦИАЛЬНО Страница 48 из 76

# Рисунок 3 Маркировка пакетика с исследуемым препаратом

Для клинических исследований- Клиническое исследование: KSL0117

Упаковка № XXX\* Гранулы OkiTask® 40 мг или Плацебо Дозировка: 1 пакет, соответствующий 40 мг или 0 мг соли кетопрофена лизина

КИО: ООО «ИФАРМА», Россия, тел. + 7 (495) 276-1143

Серия: XXXXX\*\* Срок годности: до XXXXXX

Хранить в недоступном для детей месте

# 5.7. Учет исследуемого препарата

Исследователь несет ответственность за ведение записей по учету исследуемого препарата для того чтобы избежать ошибок при получении, хранении, выдаче и возврате исследуемого препарата. Использованные пакетики должны храниться в исследовательском центре для мониторинга и подтверждения их выдачи пациентам. В случае повреждения пакетика, которое не дает пациенту принять исследуемый препарат, необходимо сделать соответствующую запись в первичной документации и журнале учета препарата, после чего пакетик должен быть заменен с помощью системы IWRS.

#### 5.8. Хранение исследуемого препарата

Исследователь несет ответственность за адекватный прием, хранение, выдачу и возврат исследуемого препарата, а также за ведение инвентарных записей и регистрацию в IWRS.

Исследователь должен обеспечить ограниченный доступ к препарату и необходимый температурный режим для его хранения. Хранение исследуемого препарата осуществляется при комнатной температуре не выше +25°С. Контроль температуры должен проводиться с применением термометров, регистрирующих максимальную и минимальную температуру за отчетный период. Информация по мониторингу температуры должна регулярно регистрироваться в журнале контроля температуры (т.е., каждый день за исключением выходных и праздничных дней).

### 5.9. Сопутствующая и резервная терапия

Все сопутствующие лекарственные препараты, в том числе растительные препараты и биологически активные пищевые добавки (БАД) должны быть зарегистрированы в первичной документации и в эИРК. К этим препаратам относятся все лекарственные препараты и биологически активные добавки.

К сопутствующей терапии также относится анестезия и терапия спасения, разрешенная протоколом исследования, которая применяется для снижения интенсивности боли (если это применимо).

Для анестезии можно использовать Ультракаин Д (артикаин 40 мг), Ультракаин ДС форте (артикаин + адреналин 40 мг + 0,01 мг/мл), Ультракаин ДС (артикаин + адреналин 40 мг + 0,005 мг/мл) в количестве 1-2 карпул. Исследователь моет выбрать препарат для анестезии с учетом состояния пациента, медицинского анамнеза и других обстоятельств. Количество использованных карпул и тип анестезии у каждого из пациентов должны быть зарегистрированы в первичной документации и в эИРК.

В случае недостаточного контроля над болью пациент получит терапию спасения для обезболивания (т.е., Парацетамол в таблетках в дозе 500-1000 мг). Участникам исследования будет предложено воздерживаться от приема резервных препаратов в течение одного часа после приема исследуемого препарата. Если прием Парацетамола в

КОНФИДЕНЦИАЛЬНО Страница 49 из 76

<sup>\*</sup> Номера наборов будут подготовлены в соответствии с рандомизационным листом и пронумерованы от 001 до 150.

дозе 500-1000 мг не даст нужного эффекта, пациентам будет разрешено принимать парацетамол в дозе 500-1000 мг каждые 6-8 часов; интервал между приемами не должен быть меньше 4 часов; максимальная суточная доза составляет 4000 мг.

Наименование препарата (предпочтительнее наименование активного вещества), дозировка, частота и способ применения, показания к применению (включая основное заболевание, сопутствующие заболевания, нежелательные явления или профилактику), дата начала и окончания применения препарата сопутствующей терапии должны быть зарегистрированы в первичной документации и в индивидуальной регистрационной карте.

Если на момент завершения исследования сопутствующая терапия продолжается, то в ИРК должна быть сделана соответствующая отметка.

# 5.10. Запрещенная предшествующая и сопутствующая терапия

К препаратам, прием которых запрещен в течение 48 часов до скрининга и в течение Дня 1 относятся:

- Антигистаминные препараты;
- Седативные препараты (в том числе растительные и БАДы).

Препараты, применение которых запрещено в течение Дня 1:

- Лекарственные препараты для анестезии, помимо указанных протоколом исследования (например, прокаин, лидокаин);
- Нестероидные противовоспалительные препараты и комбинированные препараты, в состав которых входят нестероидные противовоспалительные препараты (за исключением исследуемого препарата);
- Обезболивающие препараты: опиоиды, ацетилсалициловая кислота и ее производные, пиразолоны, другие обезболивающие и жаропонижающие препараты (за исключением препаратов терапии спасения, указанных протоколом, если применимо);
- Антитромботические лекарственные препараты;
- Гемостатическая губка.

Кроме того, запрещено участие в оценках любых исследуемых препаратов в течение 3 месяцев до начала скрининга и в течение самого исследования.

КОНФИДЕНЦИАЛЬНО Страница 50 из 76

# 6. ПРОЦЕДУРЫ ИССЛЕДОВАНИЯ

Все процедуры исследования должны проводиться в соответствии с требованиями и рекомендациями Надлежащей клинической практики Международной конференции по гармонизации (ICH GCP Раздел Е6 (R2) Руководство по надлежащей клинической практике (ЕМА/СНМР/ICH/135/1995 – 1 December 2016)) и Евразийского Экономического Союза (ЕАЭС), принципами, указанными в Хельсинкской декларации, а также в соответствии с действующим законодательством и нормативами Российской Федерации. Исследователь должен быть согласен на проведение мониторингов, аудитов и инспекций в клиническом центре и предоставить прямой доступ к материалам исследования для Спонсора и его представителей, Независимого этического комитета и представителей регуляторных органов.

#### 6.1. Информированное согласие

Информированное согласие необходимо получить на скрининге перед проведением любых процедур, относящихся к исследованию. Один экземпляр подписанного информированного согласия долен быть передан пациенту, а второй подписанный экземпляр долен быть оставлен в исследовательском центре вместе с документацией пациента по исследованию.

#### 6.2. Регистрация пациента

| Каждому пациенту, подписавшему форму информированного согласия, будет |
|---|
| присвоен индивидуальный регистрационный номер, состоящий из четырех цифр: |
| - первые две цифры соответствуют номеру центра, а вторые две – порядковому |
| номеру пациента в этом центре (01, 02, 03 и т.д.). Затем пациенту будет присвоен |
| рандомизационный номер, который распределяет система IWRS. Он состоит из буквы R и |
| двух цифр (R ). Исследователь должен перенести этот номер на этикетку |
| исследуемого препарата, распределенного пациенту (смотри раздел 5.6). |

Инструкция по регистрации пациентов в IWRS будет представлена Исследователям перед началом исследования.

# 6.3. Демографические данные и медицинский анамнез

Для оценки соответствия пациентов критериям включения/ невключения необходимо собрать демографические данные пациента (пол, дата рождения/ возраст, раса) и полный медицинский анамнез, включая значимые острые и хронические заболевания и состояния (например, постменопауза), данные по хирургическим вмешательствам и аллергическим реакциям. Кроме этого необходимо опросить пациента о госпитализациях и/или хирургических вмешательствах, запланированных на время проведения исследования (если применимо). Все новые диагнозы и состояния, выявленные в ходе скрининга, должны быть внесены в медицинский анамнез пациента.

#### 6.4. Обследование ротовой полости

Обследование ротовой полости включает оценку общего вида, состояния слизистых оболочек, зубов и горла.

Изменения по сравнению с исходным состоянием, которые расцениваются как нежелательные явления, должны быть зарегистрированы в первичной документации и в эИРК.

#### 6.5. Показатели жизненных функций, масса тела и рост

Врачебный осмотр включает измерение артериального давления, подсчет пульса и частоты дыхательных движений в положении сидя после 10 минут отдыха. Изменения по

КОНФИДЕНЦИАЛЬНО Страница 51 из 76

сравнению с исходным состоянием, которые расцениваются как нежелательные явления, должны быть зарегистрированы в первичной документации и в эИРК.

Взвешивание проводится без обуви. Рост регистрируется на основании слов пациента.

#### 6.6. Оценочные шкалы

Оценочные шкалы представлены в Приложении (Раздел 12).

# 1) Интенсивность боли

Оценка интенсивности боли проводится с помощью визуально-аналоговой шкалы (ВАШ), которая состоит из 100-миллиметровой шкалы с диапазоном от 0 мм (нет боли) до 100 мм (самая сильная боль, которую можно представить) (Раздел 12.1). Пациенту будет предложено оставить метку на шкале на основании текущей интенсивности боли.

Исследователь долен измерить расстояние от 0 до отметки на шкале с помощью стандартизованной линейки и записать результат в первичной документации и в ИРК.

#### 2) Снижение интенсивности боли

Оценка снижения интенсивности боли проводится с помощью визуально-аналоговой шкалы, которая состоит из шкалы длиной 100 мм с диапазоном от 0 мм (интенсивность боли не снизилась) до 100 мм (максимальное снижение интенсивности боли) (Раздел 12.2). Пациенту будет предложено оставить метку на шкале на основании текущего снижения интенсивности боли.

Исследователь долен измерить расстояние от 0 до отметки на шкале с помощью стандартизованной линейки и записать результат в первичной документации и в ИРК.

### 3) Общая оценка, проведенная самим пациентом

Пациенту будет предложено провести общую оценку своего состояния, ответив на вопрос: "С учетом воздействия боли, насколько хорошо Вы себя чувствуете?". Пациент должен дать ответ на шкале из 5 пунктов: 1 = очень хорошо, 2 = хорошо, 3 = удовлетворительно, 4 = плохо, 5 = очень плохо (Раздел 12.3).

Оценка по данной шкале проводится после оценки боли по визуально-аналоговой шкале до приема исследуемого препарата (исходный уровень) и в точке 6 часов после приема исследуемого препарата. Если пациент будет принимать терапию спасения, то оценка по данной шкале производится после последнего измерения по ВАШ (перед приемом терапии спасения).

Исследователь должен записать указанный пациентом балл в первичной документации и в ИРК.

# 6.7. Определение времени до первого ощутимого снижения интенсивности боли (ВПСБ) и времени до значительного снижения интенсивности боли (ВЗСБ)

Сразу же при приеме исследуемого препарата пациенты должны запустить два секундомера. Один из них должен быть остановлен сразу же, как только пациент почувствует заметное снижение боли, а второй — после того как пациент почувствует значительное снижение боли. Время до первого ощутимого снижения интенсивности боли (ВПСБ) и время до значительного снижения интенсивности боли (ВЗСБ) должны быть зарегистрированы в первичной документации и в эИРК.

КОНФИДЕНЦИАЛЬНО Страница 52 из 76

#### 6.8. Безопасность и нежелательные явления

# 6.8.1. Определения

**Нежелательное явление** (**НЯ**) — любое неблагоприятное медицинское событие, которое произошло с пациентом или испытуемым, получившим исследуемый препарат, которое не обязательно связано с проводимой терапией. Таким образом, нежелательное явление может быть любым неблагоприятным и неожиданным изменением (в т.ч., и отклонением в лабораторных показателях), симптомом или заболеванием, связанными по времени с использованием лекарственного (исследуемого) препарата, вне зависимости от того, связаны они с этим (исследуемым) препаратом или нет. В данном исследовании нежелательные явления необходимо регистрировать с момента подписания формы информированного согласия (перед получением первой дозы исследуемого препарата) до визита наблюдения (День 3±1) после последнего визита пациента или последней процедуры в рамках протокола исследования.

Боль после удаления зуба в данном исследовании не будет расцениваться, как нежелательное явление.

**Нежелательная лекарственная реакция (НЛР)** – любое нежелательное явление, для которого имеется обоснованная возможность того, что оно вызвано лекарственным препаратом. Слова "обоснованная возможность" означают, что есть какие-либо данные, подтверждающие наличие причинной взаимосвязи между препаратом (в любой дозе) и рассматриваемым нежелательным явлением.

**Серьезное нежелательное явление** – любое неблагоприятное медицинское событие, которое при любой дозе:

- привело к смерти или представляет угрозу для жизни (т.е., если во время развития нежелательного явления был риск смерти пациента. Это не относится к событиям, которые могли бы привести к смерти, если бы они были более тяжелыми)
- требует госпитализации или продления госпитализации
- привело к значительному длительному или постоянному снижению трудоспособности, пороку развития или к врожденному дефекту
- является важным медицинским событием

К важным медицинским событиям относятся те, которые могут не являться непосредственно угрожающими жизни, но имеют очевидную или выраженную клиническую значимость. Они могут привести к ухудшению состояния пациента/ участника исследования и могут потребовать вмешательства для предотвращения одного из других серьезных исходов, указанных выше. Например, передозировка препарата или злоупотребление им, судороги, которые не привели к госпитализации в стационар, или интенсивная терапия бронхоспазма в отделении неотложной помощи обычно могут быть расценены как серьезные нежелательные явления.

ПРИМЕЧАНИЕ: Госпитализация по социальным показаниям, визиты в дневной стационар, госпитализация или оперативное лечение, которые были запланированы до включения пациента в исследование для лечения основного заболевания не считаются серьезными нежелательными явлениями.

**Неожидаемая нежелательная лекарственная реакция** — нежелательная реакция, природа и тяжесть которой не соответствуют применяемой информации по препарату (например, данных из Брошюры Исследователя по не зарегистрированному препарату или инструкции по применению препарата/ краткой характеристике лекарственного препарата

КОНФИДЕНЦИАЛЬНО Страница 53 из 76

в случае зарегистрированного препарата). Эта группа также включает нежелательные лекарственные реакции, указанные в Брошюре Исследователя как характерные для данного класса препаратов или ожидаемые в связи с фармацевтическими свойствами исследуемого препарата, которые ранее отмечены не были.

Подозреваемая неожидаемая серьезная нежелательная реакция: любая подозреваемая нежелательная реакция, являющаяся как серьезной, так и неожиданной (suspected unexpected serious adverse reaction, SUSAR). Определение ожидаемости реакции должно проводиться на основе Брошюры Исследователя.

# 6.8.2. Беременность

Женщины, способные к деторождению, не исключаются из исследования в случае, если они используют надежные методы контроля рождаемости. Женщинами, способными к деторождению, считаются все женщины, физиологически способные забеременеть, в том числе женщины, находящиеся в постменопаузе менее 2 лет.

Для участия в этом исследовании его потенциальные участники должны согласиться на использование надежных методов контрацепции. Надежными методами контрацепции являются:

- а. гормональные пероральные, имплантируемые, трансдермальные или инъекционные контрацептивы;
- b. негормональное внутриматочное устройство (ВМУ), или женский презерватив со спермицидом, или контрацептивная губка со спермицидом, или диафрагма со спермицидом, или шеечный колпачок со спермицидом; или должны иметь:
- с. мужчина половой партнер женщины долен быть согласен на использование мужского презерватива со спермицидом;
- d. половой партнер, которому была выполнена стерилизация.

Участницы исследования женского пола, неспособные к деторождению или находящиеся в постменопаузе не менее 2 лет будут включаться в исследование. У всех участниц исследования женского пола должен быть отрицательный результат теста на беременность.

Беременность не является серьезным нежелательным явлением, но относится к событиям, о которых необходимо срочно уведомлять Спонсора. В случае беременности, выявленной в течение до 30 дней после приема исследуемого препарата, наступившей как у пациентки женского пола, так и у женщины-партнера пациента мужского пола, данные по беременности должны быть немедленно переданы Спонсору. За пациентками женского пола будет проводиться наблюдение в течение всего срока беременности и 30 дней после ее окончания. Состояние здоровья любых новорожденных также должно отслеживаться в течение до 30 дней после рождения (включая случаи беременности партнеров пациентов мужского пола). Важную информацию необходимо регистрировать в первичной документации, эИРК и в форме отчета по беременности. Отчеты по беременности должны быть заполнены и переданы по электронной почте/ факсу в соответствии с процедурой, описанной в Разделе 6.8.7 "Регистрация серьезных нежелательных явлений и случаев беременности".

КОНФИДЕНЦИАЛЬНО Страница 54 из 76

# 6.8.3. Регистрация нежелательных явлений и серьезных нежелательных явлений

Во время исследования и на визитах контрольного наблюдения пациенты должны докладывать о любых нежелательных явлениях, в особенности в ответ на открытые, прямые вопросы, заданные Исследователем. Исследователи также должны регистрировать любые серьезные нежелательные явления, о которых пациенты спонтанно сообщили в течение 30 дней после получения ими исследуемого препарата. Для каждого нежелательного явления/ серьезного нежелательного явления, о котором сообщил пациент, Исследователь должен собрать и зарегистрировать в первичной документации и в эИРК всю необходимую информацию, включая диагноз и симптомы, дату начала и дату разрешения, исход, степень тяжести, критерии серьезности, обстоятельства, которые могут указывать на возможную взаимосвязь с исследуемым препаратом и сопутствующей терапией, сопутствующие заболевания и состояния, процедуры исследования или другие причины, действия произведенные с исследуемым препаратом, лекарственную терапию, медицинские вмешательства, результаты лабораторных и инструментальных тестов по поводу нежелательного явления, другие обстоятельства, которые могут дополнить описание данного нежелательного явления.

Датой начала серьезного нежелательного явления является дата появления критерия серьезности. Предшествующее состояние, если это применимо, должно быть зарегистрировано как нежелательное явление, не являющееся серьезным.

Если нежелательное явление является серьезным, Исследователь также должен подать отчет по серьезному нежелательному явлению (с указанием критериев серьезности) в течение 24 часов после первого получения информации о нем медицинскому монитору компании ИФАРМА. Кроме того, Спонсор должен получить заверенные копии первичных документов по этому серьезному нежелательному явлению (выписная справка из стационара, заключение по результатам вскрытия, справка о смерти и т.п.). Данные в первичных документах и форме отчета по серьезному нежелательному явлению должны быть надлежащим образом анонимизированы.

Если у пациента наблюдается более одного серьезного нежелательного явления, Исследователь долен установить, какое из них является первичным основным, т.е., определить наиболее значимое. Если в том же отчете перечислены и другие явления, то Исследователь, вместе с указанием взаимосвязи с исследуемым препаратом, должен определить, какие нежелательные явления являются серьезными, а какие серьезными не являются. В любом случае от Исследователя требуется, чтобы он записал свое мнение о взаимосвязи наблюдаемых явлений с исследуемым лекарственным препаратом.

Нежелательные явления надлежит регистрировать и наблюдать за ними, начиная с даты подписания информированного согласия и до даты последнего визита или выполнения процедуры, связанной с исследованием (телефонный контакт в периоде наблюдения).

Регистрация серьезных нежелательных явлений, полученных спонтанно, проводится в течение 30 дней после применения исследуемого препарата: регистрация и оценка таких нежелательных явлений проводится точно также, как и регистрация и оценка серьезных нежелательных явлений, возникших в ходе исследования.

В соответствии с предписаниями ICH E2A по событиям в периоде после окончания исследования, несмотря на то что поиск и сбор такой информации не проводится Спонсором в стандартном порядке, информация по серьезным нежелательным явлениям, которые возникли после того, как пациент завершил участие в клиническом исследовании, может передаваться Исследователем непосредственно Спонсору. Такие

КОНФИДЕНЦИАЛЬНО Страница 55 из 76

случаи нежелательных явлений, возникших после окончания исследования, должны рассматриваться как требующие ускоренной регистрации, как если бы они были возникли в ходе исследования. В связи с этим для принятия решения о том, требуется ли ускоренная регистрация такого нежелательного явления, необходимо провести оценку причин его возникновения и определить его ожидаемость.

Монитор исследования отвечает за проверку соответствия записей в эИРК и отчетов по серьезным нежелательным явлениям данным в первичной документации.

Исследователь отвечает за то, чтобы участники исследования с нежелательными явлениями получили необходимое лечение любых нежелательных явлений, если такое требуется.

#### 6.8.4. Оценка тяжести

Для каждого нежелательного явления Исследователь должен провести оценку степени тяжести. С этой целью будет использоваться следующая классификация степени тяжести:

| 1. Легкой степени | Степень 1 – не влияет на обычные функции пациента (отмечаются симптомы и жалобы, которые легко переносятся (приемлемое)). |
|---|---|
| 2. Средней степени | Степень 2 – влияет в некотором объеме на обычные функции пациента (оказывают достаточно дискомфортное влияние на обычную активность (беспокоят)). |
| 3. Тяжелой<br>степени | Степень 3 — значительно влияет на обычные функции пациента (пациент неспособен к работе или не может осуществлять обычную деятельность (не приемлемое)) |

Для каждого эпизода следует регистрировать самую высокую достигнутую степень тяжести.

Обратите внимание, что нежелательные явления тяжелой степени не всегда соответствую критериям серьезности, и, наоборот, серьезное нежелательное явление не всегда должно быть нежелательным явлением тяжелой степени. Срочность регистрации серьезного нежелательного явления не зависит от степени тяжести этого явления.

#### 6.8.5. Взаимосвязь с исследуемым препаратом

Для каждого нежелательного явления Исследователь должен провести оценку его возможной взаимосвязи с исследуемым препаратом в соответствии с категориями, приведенными в Таблице далее.

| Категория нежелательного явления | Определение |
|---|---|
| 1. Взаимосвязь отсутствует (сопутствующее событие) | Явление, которое не связано и не сможет быть связано с исследуемым препаратом, например, пациент был пассажиром во время дорожно-транспортного происшествия. |
| 2. Взаимосвязь маловероятна (без прямого отношения) | Взаимосвязь маловероятна, например, клиническое событие, включая отклонения в лабораторных показателях, так связано по времени с применением препарата, что причинная взаимосвязь становится невероятной и для которого взаимосвязь с другими препаратами, веществами или заболеванием является более вероятным объяснением |
| 3. Взаимосвязь<br>возможна | Взаимосвязь может быть, но явление также могло быть вызвано состоянием пациента или другой терапией, или иной причиной |
| 4. Взаимосвязь<br>вероятна | Взаимосвязь вероятна, нежелательное явление прекращается при прекращении применения исследуемого препарата и не может быть следствием состояния пациента |
| 5. Взаимосвязь очень вероятна | Сильная взаимосвязь, явление прекращается при прекращении применения исследуемого препарата и, если это имело место, вновь возникает при возобновлении |

КОНФИДЕНЦИАЛЬНО Страница 56 из 76

| применения исследуемого препарата |
|-----------------------------------|

# 6.8.6. Оценка ожидаемости

Ожидаемость в этом исследовании определяется на основе данных из Брошюры Исследователя

| Явление<br>ожидаемо | Нежелательная реакция, природа и тяжесть которой соответствует существующей информации по препарату (например, данным из Брошюры Исследователя) |
|---|---|
| Явление<br>неожиданное | Нежелательная реакция, природа и тяжесть которой не соответствует информации из соответствующего документа по препарату (например, данным из Брошюры Исследователя) |

# 6.8.7. Регистрация серьезных нежелательных явлений и случаев беременности

Обо всех серьезных нежелательных явлениях, вне зависимости от их степени тяжести и взаимосвязи с исследуемым препаратом, а также обо всех случаях беременности необходимо сообщать на английском языке медицинскому монитору компании ИФАРМА и в отдел по безопасности препарата компании «Dompé» по факсу или по электронной почте в течение 24 часов с момента, когда Исследователю впервые стало известно об этом нежелательные явления. Информация по серьезным нежелательным явлениям должна передаваться в специальной форме отчета по серьезным нежелательным явлениям. Информация по беременности должна передаваться в специальной форме отчета по беременности. При необходимости Исследователь может связаться с Медицинским монитором для консультаций или разъяснений.

# Регистрация серьезных нежелательных явлений/ беременности

Наименование компании: ООО ИФАРМА

Медицинский монитор: Виктория Яворская

Телефон: +7 (925) 400-01-34

Факс: +7 (495) 276-1147

Электронная почта: SAE@ipharma.ru

Отдел по безопасности препарата Dompé Drug Safety:

Laura Boga, менеджер по безопасности

Прямая линия: +39 02 58383462;

Факс: +39 02 36026913

Электронная почта: farmacovigilanza@dompe.com

Медицинский монитор компании ИФАРМА будет нести ответственность за проверку соответствия переданной информации и данных, включенных в форму отчета по СНЯ/ беременности, получение и передачу любой дополнительной информации, переданной Исследователями, а также за передачу полностью заполненных форм отчетов по СНЯ/ беременности в Dompé Drug Safety незамедлительно по электронной почте и любым способом в течение 24 часов с момента, когда стало известно о явлении.

Исследователь должен проинструктировать пациентов о необходимости сообщать о серьезных нежелательных явлениях и беременности в течение исследования и 30 дней после последнего визита в исследовательский центр. В форме отчета по СНЯ/ беременности Исследователь должен предоставить всю информацию по явлению. Каждая форма отчета по СНЯ должна включать как минимум следующую информацию: данные

КОНФИДЕНЦИАЛЬНО Страница 57 из 76

пациентов, название явления, критерий серьезности, взаимосвязь с исследуемым препаратом и исход на момент создания отчета.

При составлении первичного отчета Исследователь должен указать в отчете, что этот отчет первичный ("Primary report"). При получении дополнительной информации по серьезному нежелательному явлению (например, новой информации о состоянии пациента или результатов лабораторных анализов) Исследователь должен заполнить новую форму отчета по СНЯ с пометкой о том, что это дополнительный отчет ("Additional report"). Оригинал отчета по СНЯ должен храниться в папке Исследователя.

Исследователь (или уполномоченный член персонала) несет ответственность за сообщение о любых серьезных нежелательных явлениях/ подозреваемых неожиданных серьезных нежелательных реакциях в локальный Этический комитет и в локальные учреждения в соответствии с действующими правилами и нормативами.

Спонсор будет нести ответственность за подготовку и передачу Периодических отчетов по безопасности и отчеты по SUSAR и за передачу их на рассмотрение в компанию ИФАРМА. Компания ИФАРМА будет нести ответственность за периодическую передачу отчетов по безопасности в регуляторные органы на территории России и Исследователям, а также за ускоренное сообщение о подозреваемых неожиданных серьезных нежелательных реакциях в локальные регуляторные органы в соответствии с действующими правилами и нормативами. Спонсор будет нести ответственность за сообщение необходимой информации в регуляторные органы за пределами Российской Федерации.

#### 6.8.8. Передозировка препарата

О случаях передозировки (случайной или намеренной), которые могут привести или не могут привести к серьезным нежелательным реакциям, Исследователь должен сообщать в компанию ИФАРМА и в Dompé Drug Safety с применением той же самой процедуры, то и для серьезных нежелательных явлений, в течение 24 часов после того как Исследователю стало известно о таком случае. Сюда относятся отчеты о приемах и передозировках препарата с суицидальными намерениями.

Передозировка препарата  $OKUTACK^{\otimes}$  определяется как применение более 3 пакетиков препарата в заданный день терапии.

Исследователь должен предоставить в форме отчета по СНЯ информацию о симптомах, корригирующей терапии и исходах передозировки.

### 6.9. Досрочное исключение участника из исследования

Пациент имеет право выйти из исследования в любой момент без объяснения причин. Пациент должен быть исключен из исследования в следующих случаях:

- Ему требуется терапия спасения (как предусмотрено протоколом исследования)
- Ему требуется применение запрещенных лекарственных препаратов
- Исследователь считает, что это важно с медицинской точки зрения
- Пациент отозвал сове согласие на участие в исследовании
- Пациент не выполняет процедуры, относящиеся к исследованию
- Нежелательное явление или серьезное нежелательное явление, которое влияет на безопасность или благополучие пациента

КОНФИДЕНЦИАЛЬНО Страница 58 из 76

- Пациент включен в исследование с нарушением критериев включения/ невключения, или есть значительные отклонения от протокола, которые могут повлиять на безопасность пациента и целостность данных исследования.

По возможности Исследователь должен обсудить необходимость исключения пациента с медицинским монитором или проинформировать об исключении пациента из исследования (кроме случаев прекращения исследования из-за применения резервной терапии, которые предусмотрены протоколом исследования). Причина исключения пациента из исследования должна быть указана в первичной документации и в эИРК. Если пациент прекращает свое участие в исследование более чем по одной причине, следует указать только основную причину. Если пациент исключается из исследования из-за нежелательного явления или серьезного нежелательного явления, то в качестве причины прекращения участия пациента в исследование должно быть указано это нежелательное явление или серьезное нежелательное явление.

Кроме того, Спонсор в любое время может прекратить исследование. Исследователь имеет право в любое время прекратить исследование по медицинским или регуляторным причинам. Исследование может быть прекращено только после совместных консультаций между Исследователем и Спонсором.

Серьезные нежелательные явления и случаи беременности, продолжающиеся на момент прекращения исследования, должны отслеживаться в соответствии с протоколом, если между исследователем и Спонсором не достигнуто иное соглашение.

Ни пациенты, которые будут принимать терапию спасения, ни выбывшие пациенты не будут замещены в исследовании.

КОНФИДЕНЦИАЛЬНО Страница 59 из 76

### 7. ВИЗИТЫ ИССЛЕДОВАНИЯ

# 7.1. Скрининг (Дни от -3 до 1)

- Процедура получения информированного согласия
- Присвоение скринингового номера пациенту
- Сбор демографических данных, медицинского анамнеза и данных по текущему заболеванию
- Оценка ранее полученной и сопутствующей терапии
- Обследование ротовой полости
- Определение показателей жизненных функций, массы тела и роста (по данным пациента)
- Тест на беременность
- Удаление моляра
- Оценка интенсивности боли (в течение 3 часов после удаления зуба)
- Оценка нежелательных явлений
- Оценка критериев включения/невключения

Скрининг и удаление зуба могут быть проведены в один и тот же день - День 1.

Допускается однократный повторный скрининг пациента, если процедура удаления зуба была отложена или отменена за пределами окна День -4 — День 1. В этом случае пациент должен подписать новую форму информированного согласия и ему присваивается новый номер.

Запрещается повторный скрининг пациентов для второго удаления моляра или участие в исследовании два раза.

#### 7.2. Исследуемая терапия (День 1)

#### До приема препарата

- Оценка нежелательных явлений и сопутствующей лекарственной терапии
- Рандомизация и распределение номера набора исследуемого препарата
- Оценка интенсивности боли по визуально-аналоговой шкале (0-100 мм) в момент времени 0' (непосредственно до приема исследуемого препарата)
- Общая оценка, проведенная самими пациентами (5-балльная шкала)
- Прием исследуемого препарата

Сразу же при приеме исследуемого препарата пациенты должны запустить два секундомера. Один из них должен быть остановлен сразу же, как только пациент почувствует заметное снижение боли, а второй — после того как пациент почувствует значительное снижение боли.

КОНФИДЕНЦИАЛЬНО Страница 60 из 76

#### После приема препарата

- Оценка интенсивности боли по визуально-аналоговой шкале (0-100 мм) через 5 минут, 10 минут, 15 минут, 45 минут, 30 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) после приема препарата.
  - Оценка снижения интенсивности боли по визуально-аналоговой шкале (0-100 мм) через 5 минут, 10 минут, 15 минут, 45 минут, 30 минут, 60 минут (1 час), 90 минут (1,5 часа), 120 минут (2 часа), 180 минут (3 часа), 240 минут (4 часа), 300 минут (5 часов) и 360 минут (6 часов) после приема препарата<sup>2</sup>.
- Общая оценка, проведенная самими пациентами (5-балльная шкала) после последней оценки по визуально-аналоговой шкале
- Оценка нежелательных явлений и сопутствующей лекарственной терапии

Пациент выписывается из клинического центра после завершения всех процедур визита.

# 7.3. Досрочное прекращение участия в исследовании (День 1)

В случае досрочного исключения пациента из исследования, следующие процедуры будут проведены (если применимо):

- Оценка интенсивности боли по визуально-аналоговой шкале (0-100 мм)<sup>2</sup>
- Оценка снижения интенсивности боли по визуально-аналоговой шкале  $(0-100 \text{ мм})^2$
- Общая оценка, проведенная самими пациентами (по 5-балльной шкале) после последней оценки по визуально-аналоговой шкале
- Оценка нежелательных явлений и сопутствующей лекарственной терапии

В случае недостаточного контроля над болью пациент получит терапию спасения для обезболивания (т.е., парацетамол в таблетках в дозе 500-1000 мг). Участникам исследования будет предложено воздерживаться от приема резервных препаратов в течение одного часа после приема исследуемого препарата. NB: если пациент примет терапию спасения, то вышеперечисленные процедуры должны быть проведены перед назначением терапии спасения.

Если прием парацетамола в дозе 500-1000 мг не даст нужного эффекта, пациентам будет рекомендовано принять еще одну дозу Парацетамола 500-1000 мг каждые 6-8 часов; интервал между приемами не должен быть меньше 4 часов; максимальная суточная доза составляет 4000 мг.

# 7.4. Период Наблюдения (День 3 ±1 день)

• Оценка нежелательных явлений (телефонный контакт)

КОНФИДЕНЦИАЛЬНО Страница 61 из 76

\_

<sup>&</sup>lt;sup>1</sup> Пациенты должны указывать фактическое время проведения оценки по визуально-аналоговой шкале. Отклонения от запланированных временных точек не будут считаться отклонениями от протокола исследования. Отклонениями от протокола исследования будут считаться только пропуски оценок.

Исследуемый препарат ОКИТАСК<sup>®</sup> Протокол исследования KSL0117 Финальная версия 1.0

Dompé farmaceutici s.p.a. 26 сентября 2017 года (в редакции от 25 января 2018 года)

# 7.5. Незапланированные визиты

По усмотрению Исследователя пациенты могут быть приглашены на незапланированный визит в любое время в ходе клинического исследования по требованиям безопасности, если необходимо провести осмотр или выполнить процедуру. на незапланированных визитах Исследователь может выполнить необходимые процедуры. незапланированные визиты должны быть зарегистрированы в первичной документации и в эИРК. Внеплановые визиты не должны приводить к изменениям визитов, запланированных по протоколу.

КОНФИДЕНЦИАЛЬНО Страница 62 из 76

#### 8. КОНТРОЛЬ КАЧЕСТВА

Данное исследование проводится в соответствии со стандартными операционными процедурами ООО ИФАРМА, Руководствами по Надлежащей клинической практике (GCP ICH E6 (R2)) и ЕАЭС, принципами, указанными в Хельсинкской декларации и действующими законами и нормативами Российской Федерации. Соответствие этим принципам будет проверяться при аудите клинических центров и данных исследования.

Исследователь должен ввести все необходимые данные исследования в соответствии с тем, как это указано в протоколе исследования, в эИРК, предоставленную Спонсором или его представителем. Специалисты по клиническим исследованиям (мониторы исследования) будут посещать каждый клинический центр с частотой, указанной в плане мониторинга, для проверки эИРК на предмет полноты и точности. При любом несоответствии между первичной документацией и заполненными эИРК выставляются запросы на уточнение информации и Исследователь должен ответить на них и/или устранить несоответствия. После заполнения эИРК и разрешения всех запросов Исследователь должен подписать и датировать эИРК для каждого пациента. Заполненные страницы эИРК просматриваются в ходе визитов мониторинга и передаются в базу данных исследования. При завершении исследования оригинальные эИРК будут сохранены в архиве Спонсора, а копии эИРК будут сохранены в исследовательских центрах. Удаленный мониторинг в ходе этого исследования не предусмотрен. В данном исследовании предусмотрена 100% верификация первичных данных в исследовательских центрах.

КОНФИДЕНЦИАЛЬНО Страница 63 из 76

# 9. ПЛАН СТАТИСТИЧЕСКОЙ ОБРАБОТКИ

#### 9.1. Общие соображения

Все данные по пациентам, собранные в электронных индивидуальных регистрационных картах (эИРК), будут сведены по пациентам, группам терапии и исследовательским центрам. В соответствии с показателями будут применены подходящие методы описательной статистики. Для непрерывных данных будут представлены средние показатели, стандартное отклонение (СО), медиана, диапазон (минимум и максимум) и 95% доверительный интервал (ДИ). Для категорийных данных будут представлены частота и проценты. Если это применимо, то для пропорций будут представлены 95% доверительные интервалы. Если не указано иное, то уровнем значимости, используемым для статистического тестирования, будет 0,05, а используемые тесты будут двухсторонними. Будет выпущен план статистического анализа, в котором будут подробно описаны все статистические методы и анализы, которые будут применяться к результатам исследования.

#### 9.2. Определение размера популяции

Расчет размера выборки исследования был основан на статье Seymour 1996 [3] в которой идет речь о рандомизированном, двойном слепом, плацебо-контролируемом исследовании с терапией плацебо, парацетамолом (500 и 1000 мг) и кетопрофеном (12,5 и 25 мг).

Неоткорректированные показатели  $AUC_{0-64}$  для плацебо и кетопрофена составили приблизительно 263 и 173 мм ч-1 соответственно. Соответствующие показатели стандартного отклонения составили 106 мм ч-1 (приблизительно 40% от среднего значения для AUC при применении плацебо) и 121 мм ч-1 (приблизительно 70% от среднего значения для AUC при применении кетопрофена в дозе 25 мг).

Тестируемой гипотезой для этого исследования является превосходство кетопрофена в сравнении с плацебо, что в статистических терминах будет выглядеть следующим образом:

 $H_0$ : среднее при применении плацебо  $\geq$  среднего при применении кетопрофена (без различий между разными видами терапии)

 $H_1$ : среднее при применении плацебо < среднего при применении кетопрофена (клинически и статистически значимое различие между группами),  $\Delta$ =90 мм ч-1

Всего для достижения разницы в 90 мм ч-1 между группами при мощности 80%,  $\alpha = 0.05$ , CO = 121 мм ч-1 и при соотношении рандомизации 1:1 потребуется 58 пациентов (по 29 пациентов в группе). Расчет размера популяции был проведен с помощью программы SAS 9.2 [4].

С учетом уровня досрочного выбывания из исследования, который составляет 15%, включение в исследование должно составить 70 пациентов (по 35 пациентов в каждой из групп). С учетом того что доля пациентов, не прошедших скрининг, составит приблизительно 30%, планируется, что в ходе этого исследования будет скринировано до 100 пациентов.

#### 9.3. Рандомизация

Участники исследования будут в случайном порядке распределены в одну из двух равных по размеру групп в соотношении 1:1. Рандомизация будет проводиться с применением системы интерактивного взаимодействия через сеть Интернет (interactive web response system, IWRS). Система IWRS назначит номер упаковки исследуемого

КОНФИДЕНЦИАЛЬНО Страница 64 из 76

препарата, которую надо будет выдать пациенту. Раскрытие кодов терапии для статистического анализа будет проведено после закрытия базы данных.

Набор пациентов в исследование является конкурентным между исследовательскими центрами.

#### 9.4. Популяции пациентов для анализа

Диспозиция всех пациентов будет определена перед закрытием базы данных и раскрытием кодов терапии.

# 9.4.1. Популяция назначенной терапии (ITT популяция)

Популяция назначенной терапии (Intent-to-treat, ITT) будет включать всех рандомизированных пациентов, получивших хотя бы одну дозу исследуемого препарата прошедших хотя бы одну оценку эффективности после этого; она будет основана на рандомизированной терапии, вне зависимости от реальной полученной терапии. Данные из популяции назначенной терапии будут использованы для всех анализов эффективности. Данные пациентов будут обобщены в соответствии с группами терапии, в которые они были рандомизированы.

# 9.4.2. Популяция изучения безопасности

Популяция изучения безопасности определяется, как все рандомизированные пациенты, получившие хотя бы одну дозу исследуемого препарата. Таким образом, популяция изучения безопасности будет идентична популяции назначенной терапии, если все рандомизированные пациенты получат хотя бы одну дозу исследуемого препарата. Популяция оценки безопасности будет использоваться для представления всех вводов по безопасности в зависимости от фактически полученной терапии.

#### 9.4.3. Популяция по протоколу

Популяция назначенной терапии совпадает с популяцией по протоколу, если все пациенты из нее завершат период исследуемой терапии, пройдут все оценки для первичного анализа эффективности и будут признаны комплаентными. Пациенты считаются комплаентными, если у них нет значимых отклонений от протокола в ходе исследования. Значимые отклонения от протокола будут подробно описаны в плане статистического анализа и выявлены перед закрытием базы данных.

#### 9.4.4. Обработка пропущенных данных

С учетом того что основная переменная  $AUC_{0-64}$  выводится на основании измерения интенсивности боли по визуально-аналоговой шкале, то для того чтобы избежать отклонений при непрямом тестировании эффектов терапии будут использоваться анализы первичной и вторичных переменных с замещением пропущенных данных с применением переноса вперед данных последнего наблюдения.

Анализ вторичной чувствительности будет проведен с использованием метода множественного условного замещения для пропущенных данных. В соответствии с ICH-E9, определение методов будет уточняться в плане статистического анализа в ходе изучения закрытых данных.

Замещение пропущенных данных будет возможно только у тех пациентов, которые имеют хотя бы одно обследование по ВАШ после исходного (пациент соответствует характеристике ІТТ популяции). В Плане Статистического Анализа будут представлены детали методологии, которая будет применяться при расчетах.

КОНФИДЕНЦИАЛЬНО Страница 65 из 76

# 9.5. Демографические данные и исходные характеристики

Демографические данные и исходные характеристики будут представлены для всех пациентов из популяции оценки безопасности по группам терапии и обработаны с применением методов описательной статистики.

# 9.6. Анализы эффективности

# 9.6.1. Анализ первичных конечных точек эффективности

Первичной переменной будет  $AUC_{0-64}$  профиля интенсивности боли от момента времени 0 (исходное значение на визуально-аналоговой шкале) до 6 часов после начала терапии.

Анализ  $AUC_{0.64}$  будет основан на фактических, а не на запланированных временных точках, а расчет будет проводиться по правилу трапеций. Если фактическое время не записано, то будет использовано запланированное время. Будет использован метод переноса вперед данных последнего наблюдения, как описано в Разделе 9.4.4.

Будет проведено сравнение показателей AUC при терапии со средними данными t-теста Стьюдента для независимых данных. Если средняя  $AUC_{0-64}$  при применении препарата ОКИТАСК будет меньше средней  $AUC_{0-64}$  при применении Плацебо при p<0,05, то нуль-гипотеза ( $H_0$ ), утверждающая, что препарат ОКИТАСК не отличается от плацебо, будет отклонена и вместо нее будет принята альтернативная гипотеза ( $H_1$ ), утверждающая, что препарат ОКИТАСК превосходит Плацебо.

# 9.6.2. Анализы вторичных конечных точек эффективности

Профиль боли – анализ профиля интенсивности боли будет проведен с помощью дисперсионного анализа для результатов многократных измерений (ANOVA). Данная модель будет включать фиксированные эффекты, которыми являются клинический центр, временные точки и группа терапии. Временные точки будут расценены, как повторные измерения. Для выбора соответствующей матрицы для результатов наблюдений у каждого отдельного пациента будут применены три модели, использующие составную симметрию, Huynh-Feldt и неструктурированные структуры. Матрица для итоговой модели будет выбрана с применением информационного критерия Akaike, в котором самое низкое значение означает максимальное соответствие. Будет изучена важность взаимодействия терапии в зависимости от центра, однако если она не будет значимой при 10% уровне, она будет исключена из итоговой модели. Для каждой комбинации момента времени и терапии будет проведена оценка откорректированных наименьших квадратичных. Рассчитанная разница в терапии между препаратом ОКИТАСК и плацебо в каждой из временных точек будет представлена вместе с соответствующим 95% доверительным интервалом.

Снижение интенсивности боли — анализ снижения интенсивности боли будет проведен с помощью дисперсионного анализа для результатов многократных измерений (ANOVA). Данная модель будет включать фиксированные эффекты, которыми являются клинический центр, временные точки и группа терапии. Временные точки будут расценены, как повторные измерения. Для выбора соответствующей матрицы для результатов наблюдений у каждого отдельного пациента будут применены три модели, использующие составную симметрию, Huynh-Feldt и неструктурированные структуры. Матрица для итоговой модели будет выбрана с применением информационного критерия Akaike, в котором самое низкое значение означает максимальное соответствие. Будет изучена важность взаимодействия терапии в зависимости от центра, однако если она не

КОНФИДЕНЦИАЛЬНО Страница 66 из 76

будет значимой при 10% уровне, она будет исключена из итоговой модели. Для каждой комбинации момента времени и терапии будет проведена оценка откорректированных наименьших средних квадратичных. Рассчитанная разница в терапии между препаратом ОКИТАСК и плацебо в каждый из моментов времени будет представлена вместе с соответствующим 95% доверительным интервалом.

**Время до первого ощутимого снижения боли (ВПСБ)** — для описания и определения различий в профилях в зависимости от терапии будут использованы кривые Каплана-Майера и логарифмический ранговый тест.

**Время до значимого снижения боли (ВЗСБ)** – для описания и определения различий в профилях в зависимости от терапии будут использованы кривые Каплана-Майера и логарифмический ранговый тест.

**Время до приема препарата терапии спасения** — время до приема препарата терапии спасения будет рассчитано для каждого пациента, а представлена будет только медиана. Если количество пациентов будет достаточным, то для описания и определения различий в профилях в зависимости от терапии будут использованы кривые Каплана-Майера и логарифмический ранговый тест.

**Общая оценка состояния, проведенная самими пациентами** — для определения различий между ответами на терапию будет использован тест Кохрана-Мантеля-Гензеля.

#### 9.7. Анализы безопасности

**Осмотр ротовой полости** — данные будут представлены по группам терапии для каждого момента времени с соответствующими показателями описательной статистики.

**Показатели жизненных функций** — показатели жизненных функций (артериальное давление, пульс и частота дыхательных движений) будут представлены по группам терапии для каждого момента времени с соответствующими показателями описательной статистики.

**Масса тела и рост** будут представлены по группам терапии с соответствующими показателями описательной статистики.

#### Нежелательные явления

Сводные данные по нежелательным явлениям, возникшим на фоне проводимой терапии и зарегистрированным после приема препарата, включая общее количество зарегистрированных нежелательных явлений, количество и процент пациентов, у которых было выявлено хотя бы одно нежелательное явление, количество и процент пациентов, у которых было выявлено хотя бы одно тяжелое нежелательное явление, количество и процент пациентов, досрочно вышедших из исследования из-за нежелательных явлений, количество и процент пациентов, у которых было выявлено хотя бы одно серьезное нежелательное явление и количество и процент случаев смерти будут представлены для каждой из групп терапии. Кроме того, для нежелательных явлений и для серьезных нежелательных явлений будут представлены описания явлений в каждой из категорий взаимосвязи с исследуемым препаратом.

Будет представлен разбор количества и процента пациентов с каждым из нежелательных явлений, распределенных по группам по классам систем и органов и по предпочтительным терминам в соответствии со словарем MedDRA (самой новой версией, имеющейся на момент окончания исследования). Обратите внимание, что будет вестись подсчет пациентов, а не явлений, при этом внутри каждого предпочтительного термина пациенты будут учитываться только один раз.

КОНФИДЕНЦИАЛЬНО Страница 67 из 76

Эти данные будут дополнительно представлены в таблицах в зависимости от взаимосвязи с исследуемым препаратом с разнесением по классам систем и органов и предпочтительным терминам. Взаимосвязь с исследуемым препаратом будет определяться в соответствии с тем, как она указана в эИРК.

Кроме того, с разнесением по классам систем и органов и предпочтительным терминам будет представлен краткий обзор зарегистрированных нежелательных явлений, разделенных по степени тяжести (легкая, средняя, тяжелая степень).

Будет представлен краткий обзор нежелательных явлений, в результате которых пациенты досрочно вышли из исследования, сгруппированных по классам систем и органов и предпочтительным терминам.

Будут перечислены все нежелательные явления, зарегистрированные в эИРК.

#### 9.7.1. Серьезные нежелательные явления

Будет представлен разбор количества и процента пациентов с каждым из серьезных нежелательных явлений, возникших после приема исследуемого препарата, распределенных по классам систем и органов и по предпочтительным терминам в соответствии со словарем MedDRA.

Эти данные будут дополнительно представлены в таблицах в зависимости от взаимосвязи с исследуемым препаратом с разнесением по классам систем и органов и предпочтительным терминам.

Кроме того, в зависимости от классов систем и органов и предпочтительных терминов будет представлен краткий обзор зарегистрированных серьезных нежелательных явлений, разделенных по степени тяжести (легкая, средняя, тяжелая степень).

Будет представлен краткий обзор серьезных нежелательных явлений, в результате которых пациенты досрочно вышли из исследования, сгруппированных по классам систем и органов и предпочтительным терминам.

КОНФИДЕНЦИАЛЬНО Страница 68 из 76

### 10. АДМИНИСТРАТИВНЫЕ ПРОЦЕДУРЫ

#### 10.1. Законодательные аспекты

Имена всех пациентов должны храниться в строгой секретности. Идентификация пациента проводится по присвоенному ему номеру и дате рождения. Пациенты должны быть проинформированы о том, что любая информация, хранящаяся в исследовательском центре, у Спонсора или его представителей, будет храниться в строгой секретности в соответствии с регуляторными требованиями.

#### 10.2. Ответственность Исследователя

Исследователь должен вести клиническое исследование в соответствии с протоколом исследования, Руководствами по Надлежащей клинической практике Международной конференции по гармонизации (ICH GCP E6 (R2)) и Евразийского экономического союза (EAЭС), с принципами, заявленными в Хельсинкской декларации и в соответствии с действующими законами и нормативами.

Исследователь должен разрешить проведение мониторингов, аудитов и инспекций в исследовательском центре и в любое время предоставить прямой доступ ко всем материалам, имеющим отношение к исследованию Спонсору или его представителям, Независимому этическому комитету и регуляторным органам.

Исследователь должен хранить оригиналы всех подписанных информированных согласий, а также полный список участников исследования, включая полные имена, адреса и номера телефонов, чтобы их можно было позднее идентифицировать при необходимости. Эти документы не должны копироваться для передачи Спонсору или его представителям.

Исследователь обязан обеспечить целостность и полноту материалов исследования, в том числе первичной документации, копий индивидуальных регистрационных карт и Папки Исследователя в течение не менее 15 лет после завершения исследования или до момента, указанного Спонсором. Исследователь обязан убедиться, что первичная документация ведется качественно, разборчиво, заполняется своевременно, является подлинной, точной и полной.

В любом случае, перед утилизацией документации учреждению необходимо получить письменное разрешение компании Домпе.

# 10.3. Процедуры мониторинга

Главный Исследователь должен предоставить прямой доступ ко всей первичной документации, эИРК и Файлу исследователя представителям Спонсора, а также представителям регуляторных органов. Первичная документация включает оригиналы документов, данные и записи (например, больничные записи, истории болезни, заметки, дневники, опросники, документы учета препарата, данные, полученные с записи автоматических аппаратов, верифицированные и заверенные копии выписки из истории болезни, фотонегативы, фотопленки или записи на магнитных носителях, рентгеновские снимки и любые другие записи, имеющие отношение к пациенту и использующиеся в клиническом исследовании).

Мониторинг будет проводиться представителями компании ИФАРМА в соответствии с со стандартными операционными процедурами компании и Планом мониторинга, разработанным для данного исследования. Помимо обычных мониторинговых визитов, Спонсор может принять решение о проведении совместного мониторингового визита по соглашению с компанией ИФАРМА.

КОНФИДЕНЦИАЛЬНО Страница 69 из 76

# 10.4. Электронные регистрационные карты для записи данных

Исследователь должен перенести данные клинического исследования из первичной документации в эИРК в необходимом количестве. Руководство по заполнению эИРК должны быть изучены на митинге Исследователей и/или на инициирующем визите в центре. Если Главный Исследователь делегирует обязанности по заполнению эИРК другим работникам исследовательского центра, то их имена, занимаемые должности, инициалы и подписи должны быть внесены в Журнал распределения обязанностей и переданы Спонсору или его представителю. Все изменения, внесенные в эИРК, должны отслеживаться, что означает сохранение как исправленых данных, так и данных до исправления, с указанием причины исправления, даты исправления и данных о лице, которое внесло исправления. Заполненная эИРК должна быть заверена электронной подписью Главного Исследователя.

#### 10.5. Хранение записей

Первичная документация, а также электронные копии эИРК и Файлы Исследователя должны храниться в исследовательском центре или в специальном хранилище с ограниченным доступом в течение не менее 15 лет после окончания исследования или до сроков, указанных Спонсором. В случае попадания документов к другим лицам или в другие учреждения Спонсор должен быть уведомлен об этом. В любом случае, перед утилизацией документации учреждению необходимо получить письменное разрешение компании Домпе.

Материалы, относящиеся к исследованию, должны сохраняться Спонсором и его представителями в соответствии с регуляторными требованиями.

#### 10.6. Этические аспекты

#### 10.6.1. Независимый этический комитет

Перед началом клинического исследования все исследовательские центры должны получить письменное разрешение на проведение исследования от Независимых этических комитетов (НЭК) в соответствии с руководствами по Надлежащей клинической практике Международной конференции по гармонизации (ICH GCP E6 (R2)) и Евразийского экономического союза (ЕАЭС), принципами, заявленными в Хельсинкской декларации и в соответствии с действующими законами и нормативами Российской Федерации. В Независимый этический комитет должны быть представлены следующие документы: протокол исследования с поправками, информационный листок пациента и форма информированного согласия, письменные материалы, которые должны быть предоставлены пациентам, Брошюра Исследователя, информация по безопасности исследуемого препарата, информация по выплатам и компенсациям для участников исследования, резюме исследователей и другие документы по запросу.

Спонсору должен быть предоставлен список членов НЭК и заявление о соответствии принципам Надлежащей клинической практики (GCP) и регуляторным требованиям.

#### 10.6.2. Некоторые вопросы, касающиеся этики

Процедуры, описанные в протоколе клинического исследования, связанные сего применением, оценками и документированием результатов, разработаны для того чтобы гарантировать соответствие действий Спонсора и Исследователя руководствам по Надлежащей клинической практике Международной конференции по гармонизации (ІСН GCP E6 (R2)) и Евразийского экономического союза (ЕАЭС). Данное клиническое исследование также может проводиться в соответствии с действующими законами и нормативными требованиями. Это подразумевает возможность проведения аудита

КОНФИДЕНЦИАЛЬНО Страница 70 из 76

представителями Спонсора и/или регуляторных органов. Исследователь должен разрешить проведение мониторингов, аудитов и инспекций в исследовательском центре и в любое время предоставить прямой доступ ко всем материалам, имеющим отношение к исследованию Спонсору или его представителям, Независимому этическому комитету и регуляторным органам.

# 10.6.3. Информированное согласие

Перед началом клинического исследования Исследователь должен получить от Независимого этического комитета письменное одобрение Информационного листка пациента и Формы информированного согласия и любых иных письменных/печатных материалов, предоставляемых пациентам. Письменное одобрение от НЭК и одобренные документы должны храниться в Папке Исследователя.

При получении информированного согласия Исследователь должен действовать в соответствии с руководствами по Надлежащей клинической практике Международной конференции по гармонизации (ICH GCP E6 (R2)) и Евразийского экономического союза (ЕАЭС), принципами, заявленными в Хельсинкской декларации и в соответствии с действующими законами и нормативами Российской Федерации. Форма информированного согласия должна быть датирована и подписана лично пациентом перед началом любых процедур исследования.

Процесс получения информированного согласия должен быть подробно описан в первичной документации, в том числе с указанием согласия пациента на участие в этом клиническом исследовании и даты подписания формы информированного согласия.

# 10.7. Финансирование

Настоящее исследование проводится и полностью спонсируется компанией "Dompé farmaceutici s.p.a." (Италия). Все затраты, связанные с проведением исследования, включая государственные пошлины, страховки и оплату работы исследовательских центров, Исследователей и третьих лиц, участвующих в проведении исследования, а также поставки исследуемого препарата и других материалов исследования, покрываются компанией "Dompé farmaceutici s.p.a." в соответствии с тем как это описано в контракте между компанией ИФАРМА и компанией "Dompé farmaceutici s.p.a.".

Участие в этом исследовании не требует каких-либо финансовых затрат от педиатрических пациентов. Все процедуры исследования, включая визиты в исследовательский центр, лабораторные и инструментальные обследования, будут проводиться бесплатно. Участие в этом исследовании не подразумевает оплату для пациентов.

Жизнь и здоровье пациентов, принимающих участие в этом клиническом исследовании, будут застрахованы в соответствии с законодательством Российской Федерации (Статья 44 федерального закона "Об обращении лекарственных средств" № 61-ФЗ от 12 апреля 2010 года и другие действующие регуляторные требования). После подписания формы информированного согласия пациенты получат сертификат страхования здоровья для участников исследования.

# 10.8. Политика в отношении публикаций

Полные и частичные результаты данного исследования, выполненные в соответствии с настоящим протоколом, а также любая другая информация, представленная Спонсором в елях проведения исследования, запрещены к публикации или к передаче любым третьим лицам без согласия Спонсора исследования. Все Исследователи, принимающие участие в

КОНФИДЕНЦИАЛЬНО Страница 71 из 76

Исследуемый препарат ОКИТАСК $^{\otimes}$  Протокол исследования KSL0117 Финальная версия 1.0

Dompé farmaceutici s.p.a. 26 сентября 2017 года (в редакции от 25 января 2018 года)

проведении этого исследования, должны предоставить спонсору полные результаты тестов и все данные, полученные в ходе этого исследования.

КОНФИДЕНЦИАЛЬНО Страница 72 из 76

#### 11. ЛИТЕРАТУРНЫЕ ССЫЛКИ

- 1. Veys EM. 20 Years' Experience with Ketoprofen. Scand J Rheumatol 1991; Suppl. 90: 3-44.
- 2. Singla NK, Desjardins PJ, Chang PD. A comparison of the clinical and experimental characteristics of four acute surgical pain models: dental extraction, bunionectomy, joint replacement, and soft tissue surgery. Pain. 2014 Mar;155(3):441-56
- 3. Seymour R A, Kelly P J, Hawkesford J E. The efficacy of ketoprofen and paracetamol (acetaminophen) in postoperative pain after third molar surgery. Br J Clin Pharmacol 1996; 41: 581–585.
- 4. SAS 9.2 http://support.sas.com/documentation/92/
- 5. MeDRA. https://www.meddra.org/
- 6. Grichnik K P, FERRANTE F M. The Difference between Acute and Chronic Pain The E Mount Sinai Journal of Medicine 1991, 58:3 217-219
- 7. Kantor TG. A Review of Its Pharmacologic and Clinical Properties. Pharmacotherapy 1986; 6(3): 93-103.
- 8. Martindale: the Complete Drug Reference: Ketoprofen. Available at: <a href="http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference-Accessed 13 July 2015">http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference-Accessed 13 July 2015</a>.
- 9. KSL0112 (CRO-PK-11-262) Two-way crossover, randomised, single dose bioequivalence phase I study of ketoprofen lysine salt as orodispersible granules (40 mg administered without water) versus ketoprofen lysine salt as granules for oral solution (80 mg bipartite sachet, half sachet) after oral administration to healthy volunteers of both sexes. 30 April 2012.
- 10. Panerai A E, Lanata L, Ferrari M, Bagnasco M. A new ketoprofen lysine salt formulation: 40 mg orodispersible granules Trends in Medicine 2012 October, 12:159-167.
- 11. RBM 930475. Single dose toxicity study in mice treated by oral route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofen Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, July 7, 1994.
- 12. RBM 930473. Single dose toxicity study in rats treated by oral route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofene Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, June 23, 1994.
- 13. RBM 930476. Single dose toxicity study in mice treated by intraperitoneal route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofen Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, July 7, 1994
- 14. RBM 930474. Single dose toxicity study in rats treated by intraperitoneal route with Ketoprofen lysine salt, S-Ketoprofen Lysine salt, R-Ketoprofen Lysine salt and Ketoprofen. RBM, Colleretto Giacosa (TO), Italy, June 23, 1994.
- 15. RBM 930477 KLS, S-ketoprofen Lysine salt, R-ketoprofen Lysine salt and ketoprofen. 2-week toxicity studies in rats treated by oral route. RBM, Colleretto Giacosa (TO), Italy, July 21, 1994.
- 16. RBM 910102. 13-week repeated dose toxicity study in Sprague Dawley Crl:CD (SD) BR rats treated with the test article Ketoprofen lysine salt administered by oral route at the

КОНФИДЕНЦИАЛЬНО Страница 73 из 76

- doses of 0, 2.5, 7.5 and 15 mg/kg/day followed by a 6-week recovery period. RBM, Colleretto Giacosa (TO), Italy, March 2,1993
- 17. DOM/007/AKL Repeat dose dermal toxicity to rats. A 13-week study. Life Science Research Israel Ltd., Israel, Januray 7, 1991.
- 18. Cimini A, Brandolini L, Gentile R, Cristiano L, et al. Gastroprotective Effects of Lysine Salification of Ketoprefen in Ethanol-Injured Gastric Mucosa. J Cell Physiol. 2015 230: 813-820
- 19. DOM/008/AKL Repeat dose dermal toxicity to rabbits. A l3-week study. Life Science Research Israel Ltd., Israel, Januray 6, 1991.
- RBM 930478 KLS, S-ketoprofen Lysine salt, R-ketoprofen Lysine salt and ketoprofen. Dose Range finding study by oral route in dogs - RBM, Colleretto Giacosa (TO), Italy, July 20, 1994.
- 21. RBM 880004. 13-week repeated dose toxicity study in marmosets treated with the test article Ketoprofen lysine salt administered by oral route at the doses of 0, 2.5, 7.5 and 15 mg/kg/day followed by a 6-week recovery period. RBM, Colleretto Giacosa (TO), Italy, 14 April 1989.
- 22. RBM 880006. Ketoprofen lysine salt. Ames test. RBM, Colleretto Giacosa (TO), Italy, February 29, 1988.
- 23. RBM 890666. Ketoprofen lysine salt. Chromosome aberrations in human lymphocytes. RBM, Colleretto Giacosa (TO), Italy, May 26, 1990.
- 24. RBM 880007. Ketoprofen lysine salt. Gene conversion test in S. cerevisiae D4. RBM, Colleretto Giacosa (TO), Italy, March 30, 1988.
- 25. RBM 920773. Ketoprofen lysine salt. Unscheduled DNA synthesis in cultured HeLa cells. RBM, Colleretto Giacosa (TO), Italy, Febbruary 16, 1993.
- 26. RBM 880008. Ketoprofen lysine salt. Micronucleus test in rat bone marrow. RBM, Colleretto Giacosa (TO), Italy, April 18, 1988
- 27. RBM 880005. Ketoprofen lysine salt. Preliminary teratogenesis study by oral route in rabbits. RBM, Colleretto Giacosa (TO), Italy, December 21, 1989.
- 28. RBM 910272 4-week toxicity study in rabbis by vaginal route. RBM, Colleretto Giacosa (TO), Italy, November 14, 1991.
- 29. Sarzi-Puttini P, Atzeni F, Lanata L et al. Pain and ketoprofen: what is its role in clinical practice? Reumatismo, 2010; 62(3): 172-188.
- 30. Geisslinger G, Menzel S, Wissel K, K. Brune K. Pharmacokinetics of ketoprofen enantiomers after different doses of the racemate. Br J Clin Pharmacol 1995; 40: 73-75
- 31. Bannwarth B, Lapicque F, Netter P, Monot C, Tamisier JN, Thomas P, Royer RJ. The effect of food on the systemic availability of ketoprofen. Eur J Clin Pharmacol. 1988;33(6):643-5.
- 32. Martindale: the Complete Drug Reference: Ketoprofen. Available at: <a href="http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference-Accessed 13 July 2015">http://www.pharmpress.com/product/MC\_MART/martindale-the-complete-drug-reference-Accessed 13 July 2015</a>.
- 33. Netter P, Lapicque F, Bannwarth B, Tamisier JN, et al. Diffusion of Intramuscular Ketoprofen Into the Cerebrospinal Fluid. Eur J Clin Pharmacol. 1985; 29:319-21.

КОНФИДЕНЦИАЛЬНО Страница 74 из 76

- 34. Advenier C, Roux A, Gobert C et al. Pharmacokinetics of ketoprofen in the elderly. Br J Clin Pharmacol 1983; 16: 65-70.
- 35. Skeith KJ, Dasgupta M, Lange R, Jamali F. The influence of renal function on the pharmacokinetics of unchanged and acyl-glucuroconjugated ketoprofen enantiomers after 50 and 100 mg racemic ketoprofen. Br J Clin Pharmacol 1996; 42: 163–169.
- 36. Stafanger G, Larsen HW, Hansen H, Sorensen K. Pharmacokinetics of ketoprofen in patients with chronic renal failure. Scand J Rheumatology 1981; 10: 189-192.
- 37. Vallés J, Artigas J R, Bertolotti M, Crea3 A, Müller F, Paredes I, Capriati A Single and Repeated Dose Pharmacokinetics of Dexketoprofen Trometamol in Young and Elderly Subjects. Methods Find Exp Clin Pharmacol 2006, 28(Suppl. A): 13-19.
- 38. Upton, RA, Buskin, JN, Williams, RL, Holford, NHG, Riegelman, S. Negligible excretion of unchanged ketoprofen, naproxen and probenecid in urine, J Pharm Sci 1980 69: 1254-1257.
- 39. Dawood, M.Y. Nonsteroidal antiinflammatory drugs and reproduction. Am. J. Obstet. Gynecol., 1993, 169, 1255-1265.
- 40. Van der Weiden, R.M.; Helmerhorst, F.M.; Keirse, M.J. Influence of prostaglandins and platelet activating factor on implantation. Hum. Reprod., 1991, 6, 436-442
- 41. Van der Weiden, R.M.; Helmerhorst, F.M.; Keirse, M.J. Prostanoid excretion in incipient singleton and twin pregnancies. Am. J. Obstet. Gynecol., 1996, 174, 1614-1617.
- 42. Van der Weiden, R.M.; Wouters, J.M. Infertility may sometimes be associated with nonsteroidal anti-inflammatory drug consumption. Br. J. Rheumatol., 1997, 36, 605.
- 43. Siu, S.S.; Yeung, J.H.; Lau, T.K. An in-vivo study on placental transfer of naproxen in early human pregnancy. Hum. Reprod., 2002, 17, 1056-1059.
- 44. Antonucci R, Zaffanello M, Puxeddu E, Porcella A et al. Use of Non-steroidal Antiinflammatory Drugs in Pregnancy: Impact on the Fetus and Newborn. Curr Drug Metab. 2012; 13(4):474-90.
- 45. Ofori, B.; Oraichi, D.; Blais, L.; Rey, E.; Bérard, A. Risk of congenital anomalies in pregnant users of non-steroidal anti-inflammatory drugs: A nested case-control study. Birth Defects Res. B. Dev. Reprod. Toxicol., 2006, 77(4), 268-279.
- 46. Ericson A, Källén BA. Nonsteroidal anti-inflammatory drugs in early pregnancy. Reprod. Toxicol. 2001 Jul-Aug; 15(4):371-5 2001.
- 47. Dollery C, ed. Therapeutic Drugs. Second Edition. Churchill Livingstone. Edinburgh 1999.
- 48. Becker J C, Domschke W, Pohle T. Current approaches to prevent NSAID-induced gastropathy COX selectivity and beyond Br J Clin Pharmacol 58:6 587–600 587.

КОНФИДЕНЦИАЛЬНО Страница 75 из 76

# 12. ПРИЛОЖЕНИЕ

# 12.1. Визуально-аналоговая шкала "Интенсивность боли"

Пожалуйста, поставьте отметку на шкале ниже в соответствии с интенсивностью Вашей боли в настоящий момент.

Боли нет

Самая сильная боль, какую можно представить

# 12.2. Визуально-аналоговая шкала "Снижение интенсивности боли"

Пожалуйста, поставьте отметку на шкале ниже в соответствии со степенью снижения интенсивности Вашей боли в настоящий момент.

#### Снижения боли нет

**Максимальное снижение** боли

# 12.3. Общая оценка, проведенная самими пациентами (по 5-балльной шкале)

С учетом всех аспектов, связанных с Вашей болью, насколько хорошо Вы себя чувствуете?

| 1 = очень<br>хорошо | 2 = хорошо | 3 =<br>удовлетворительно | 4 = плохо | 5 = очень<br>плохо |
|---|---|---|---|---|

КОНФИДЕНЦИАЛЬНО Страница 76 из 76